# Replication of the EINSTEIN-DVT Anticoagulant Trial in Healthcare Claims Data

NCT04736420

September 14 2021

#### 1. RCT Details

This section provides a high-level overview of a **published** RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Oral Rivaroxaban for Symptomatic Venous Thromboembolism (EINSTEIN DVT)

### 1.2 Intended aim(s)

To compare the risk of symptomatic, recurrent venous thromboembolism (VTE) in patients with acute, symptomatic deep vein thrombosis (DVT) for rivaroxaban versus standard therapy of warfarin.

### 1.3 Primary endpoint for replication

The primary outcome of the study was symptomatic, recurrent VTE

### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

Assuming a noninferiority margin of 2.0, it was determined that about 3,000 patients would be needed to achieve 90% power to conclude noninferiority of rivaroxaban over standard therapy at two-sided alpha of 0.05.

### 1.5 Secondary endpoint for replication (assay sensitivity) and RCT finding

Major bleeding; RR = 0.65 (95% CI 0.33-1.30)

### 1.6 Trial estimate

RR = 0.68 (95% CI 0.44-1.04) comparing rivaroxaban vs standard therapy (Agnelli et al., 2010)

### 2. Person responsible for implementation of replication in Aetion

Dureshahwar Jawaid, MPH implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

### 3. Data Source(s)

Optum, MarketScan, Medicare

### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Figure 1.

Design Diagram – EINSTEIN-DVT TRIAL REPLICATION



### 5. Cohort Identification

### 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing rivaroxaban to warfarin users. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of rivaroxaban or warfarin (index date). We will restrict the analyses to patients with a diagnosis of proximal DVT without symptomatic PE.

### 5.2 Important steps for cohort formation

New use of rivaroxaban, exposure, and warfarin, comparator, is defined as no use of either therapy in 180 days prior to index date.

### 5.2.1 Eligible cohort entry dates

Market availability of rivaroxaban in the U.S. prevention of venous thromboembolism after orthopedic surgery started on July 30, 2008

- For Medicare: July 30, 2008– December 31, 2017 (end of available data)
- For Marketscan: July 30, 2008 December 31, 2018 (end of available data)
- For Optum: July 30, 2008 March 31, 2020 (end of available data)
- 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date.

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

### 5.3 Flowchart of the study cohort assembly

| | Optum | | Truven | | Medicare | |
|---|---|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 77,673,639 | | 200,203,908 | | 6,886,908 |

| Did not meet cohort entry criteria | -76,678,873 | 994,766 | -199,008,369 | 1,195,539 | -1,964,276 | 4,922,632 |
|---|---|---|---|---|---|---|
| Excluded due to insufficient enrollment | -118,721 | 876,045 | -99,207 | 1,096,332 | -232,358 | 4,690,274 |
| Excluded due to prior use of referent | -516,528 | 359,517 | -684,176 | 412,156 | -3,197,338 | 1,492,936 |
| Excluded due to prior use of exposure and because patient qualified in >1 exposure category | -221,490 | 138,027 | -216,501 | 195,655 | -834,065 | 658,871 |
| Excluded based on Age (<65 - Medicare only) | - | - | - | - | -72456 | 586,415 |
| Excluded based on Age (missing) | 0 | 138,027 | 0 | 195,655 | -214 | 586,201 |
| Excluded based on Gender | 0 | 138,027 | 0 | 195,655 | 0 | 586,201 |
| Excluded based on Use of other NOACs (dabigatran, apixaban, edoxaban) | -5421 | 132,606 | -4267 | 191,388 | -21987 | 564,214 |
| Excluded based on Inclusion # 1 - DVT w/o Symptomatic PE and based on Exclusion # 1 - Age <=18 | -117,812 | 14,794 | -168,633 | 22,755 | -499,609 | 64,605 |
| Excluded based on Exclusion # 2 - Thrombobectomy, Caval Filter | -210 | 14,584 | -335 | 22,420 | -903 | 63,702 |
| Excluded based on Exclusion # 3 - other indications for VKA | -1721 | 12,863 | -2,053 | 20,367 | -9,815 | 53,887 |
| Excluded based on Exclusion # 6 - CKD stage 4/5/ESRD | -114 | 12,749 | -121 | 20,246 | -496 | 53,391 |
| Excluded based on Exclusion # 7 - Liver Disease and based on Exclusion # 8 - Bacterial Endocarditis | -497 | 12,252 | -767 | 19,479 | -1,320 | 52,071 |
| Excluded based on Exclusion # 9 - CCI | -184 | 12,068 | -155 | 19,324 | -348 | 51,723 |
| Excluded based on Exclusion # 10 - Active Bleeding/High Risk for Bleeding | -295 | 11,773 | -478 | 18,846 | -1,156 | 50,567 |
| Excluded based on Exclusion # 11 - Malignant Hypertension and based on Exclusion # 12 - Pregnancy | -39 | 11,734 | -116 | 18,730 | -120 | 50,447 |
| Excluded based on Exclusion # 14 - CYP3A4 Inhibitors | -12 | 11,722 | -28 | 18,702 | -72 | 50,375 |
| Excluded based on Exclusion # 15 - Symptomatic Pulmonary Embolism | -369 | 11,353 | -817 | 17,885 | -1008 | 49,367 |
| Final cohort | | 11353 | | 17885 | | 49367 |

Effectiveness research with Real World Data to support FDA's regulatory decision making

#### 6. Variables

#### 6.1 Exposure-related variables:

### Study drug:

The study exposure of interest is initiation of rivaroxaban. New initiation will be defined by no use of rivaroxaban or warfarin in the prior 6 months before treatment initiation (washout period).

#### **Comparator:**

New initiators of warfarin, defined by no use of rivaroxaban or warfarin in the prior 6 months.

#### 6.2 Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B).

### 6.3 Outcome variables and study follow-up:

### 6.3.1 Outcome variables

Primary Effectiveness outcomes of interest: (definitions provided in **Appendix A**):

• Primary Outcome: VTE

Safety outcomes of interest:

1. Major bleeding

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the primary analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of rivaroxaban and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (rivaroxaban and comparator) plus a defined grace period (i.e., 10 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from exposure to comparator or vice versa or augmentation/switching to any other NOAC (e.g. switching from rivaroxaban to apixaban would be a censoring event);
  - o A dosage change on the index treatment does not fulfill this criterion
  - o An added treatment that is not part of the exposure or comparator group does not fulfill this criterion

For the intention-to-treat (ITT) analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

#### 7. Initial Feasibility Analysis

#### Aetion report name:

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1482/results/64422/result/0">https://bwh-dope.aetion.com/projects/details/1482/results/64422/result/0</a>
MarketScan- <a href="https://bwh-dope.aetion.com/projects/details/1480/results/64423/result/0">https://bwh-dope.aetion.com/projects/details/1480/results/64423/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/projects/details/1479/results/64424/result/0">https://bwh-dope.aetion.com/projects/details/1480/results/64423/result/0</a>

Date conducted: 1/15/2021

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of study population
- Report median follow-up time by treatment group
- Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

### Aetion report name:

For rivaroxaban vs. warfarin

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1482/results/63169/result/0">https://bwh-dope.aetion.com/projects/details/1482/results/63169/result/0</a>
Mediare- <a href="https://bwh-dope.aetion.com/projects/details/1479/results/63200/result/0">https://bwh-dope.aetion.com/projects/details/1480/results/63169/result/0</a>
Mediare- <a href="https://bwh-dope.aetion.com/projects/details/1479/results/63200/result/0">https://bwh-dope.aetion.com/projects/details/1480/results/63168/result/0</a>

Date conducted: 12/22/2020 (Medicare 12/23/20)

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 2 covariates: age and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

- Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.
- Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 11/18/2020 |
|-------------------------|------------------|----------------|------------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 11/29/2020 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

### **Aetion report links:**

Optum: https://bwh-dope.aetion.com/projects/details/1482/results/63187/result/0

Marketscan: https://bwh-dope.aetion.com/projects/details/1480/results/63178/result/0

Medicare: https://bwh-dope.aetion.com/projects/details/1479/results/63202/result/0

Date conducted: 12/23/20

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy outcome | 326 (1.04%) | 175 (1.11%) | 151 (0.96%) |
| Death | 698 (2.22%) | 345 (2.20%) | 353 (2.25%) |
| Start of an additional exposure | 1,548 (4.93%) | 983 (6.26 %) | 565 (3.60%) |
| End of index exposure | 23,549 (74.98%) | 11,297 (71.94%) | 12,252 (78.02%) |
| Specified date reached | 1,374 (4.37%) | 711 (4.53%) | 663 (4.22%) |
| End of patient enrollment | 925 (2.95%) | 503 (3.20%) | 422 (2.69%) |
| Switch to other NOACs (for censoring) + nursing home admission | 2,988 (9.51%) | 1,690 (10.76%) | 1,298 (8.27%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | | |
|---|---|---|---|
| Patient Group Optum Marketscan Medicare | | | |
| Overall Patient Population | 59 [29-131] | 73 [38-146] | 73 [38-154] |
| Referent | 64 [28-138] | 78 [38-150] | 82 [38-165] |
| Exposure | 54 [29-126] | 67 [38-141] | 65 [38-139] |

• Report overall risk of the primary outcome.

| | Optum | Marketscan | Medicare | Pooled |
|-------------------------|-------|------------|----------|--------|
| Risk per 1,000 patients | 17.57 | 18.15 | 18.96 | 18.54 |

### **10. Final Power Assessment**

Date conducted: 12/23/20

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

### o Pooled

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | 25,970 | Number of patients matched | 25,970 |
| Reference | 12,985 | Reference | 12,985 |
| Exposed | 12,985 | Exposed | 12,985 |
| Risk per 1,000 patients | 18.54 | Risk per 1,000 patients | 18.54 |
| Desired HR from RCT | 0.68 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 2 |
| Number of events expected | 481.4838 | Number of events expected | 481.4838 |
| Power | 0.988435033 | Power | 0.999999992 |

# o Optum

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | 3,150 | Number of patients matched | 3,150 |
| Reference | 1,575 | Reference | 1,575 |
| Exposed | 1,575 | Exposed | 1,575 |
| Risk per 1,000 patients | 17.57 | Risk per 1,000 patients | 17.57 |
| Desired HR from RCT | 0.68 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 2 |
| Number of events expected | 55.3455 | Number of events expected | 55.3455 |
| Power | 0.299994744 | Power | 0.731829277 |

### Marketscan

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | 5,798 | Number of patients matched | 5,798 |
| Reference | 2,899 | Reference | 2,899 |
| Exposed | 2,899 | Exposed | 2,899 |
| Risk per 1,000 patients | 18.15 | Risk per 1,000 patients | 18.15 |
| Desired HR from RCT | 0.68 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 2 |
| Number of events expected | 105.2337 | Number of events expected | 105.2337 |
| Power | 0.507287833 | Power | 0.944678362 |

Effectiveness research with Real World Data to support FDA's regulatory decision making

#### Medicare

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | 17,022 | Number of patients matched | 17,022 |
| Reference | 8,511 | Reference | 8,511 |
| Exposed | 8,511 | Exposed | 8,511 |
| Risk per 1,000 patients | 18.96 | Risk per 1,000 patients | 18.96 |
| Desired HR from RCT | 0.68 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 2 |
| Number of events expected | 322.73712 | Number of events expected | 322.73712 |
| Power | 0.933738593 | Power | 0.999990058 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 12/24/2020 |
|-------------------------|--------------|----------------|------------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 01/18/2020 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

### 11. Study Confidence and Concerns

Deadline for voting on study confidence and listing concerns:

Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the

success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the individual respondent.

• After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

### 12. Register study protocol on clinicalTrials.gov

### Date conducted:

• Register the study on <u>clinicalTrials.gov</u> and upload this document.

### 13. Comparative Analyses

Aetion report name:

Date conducted:

- 13.1 For primary analysis:
- 13.2 <u>For sensitivity analyses:</u>

### 14. Requested Results

### 14.1 Table 1: Baseline characteristics before and after adjustment

| Variable | Before adjustment | | After adjustment | | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |

### 14.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

### 14.3 <u>Table 3: Censoring events</u>

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

# 14.4 <u>Table 4: Results from primary analyses;</u>

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; CI, Confidence Interval.

Effectiveness research with Real World Data to support FDA's regulatory decision making

### 14.5 Table 5: Results from secondary analyses;

### 15. References

Agnelli G, Berkowitz S, Bounameaux H, et al. Oral Rivaroxaban for Symptomatic Venous Thromboembolism. N Engl J Med. 2010; 363:2499-2510

Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

| # | EINSTEIN DVT trial definitions | Implementation in routine care | Please see the following Google Drive for further details or any missing infor <a href="https://drive.google.com/drive/folders/1WD618wnyw/jEaXzfl.Tcuk.VCcnb6b-gV?">https://drive.google.com/drive/folders/1WD618wnyw/jEaXzfl.Tcuk.VCcnb6b-gV?</a> | |
|---|---|---|---|---|
| | Trial details- Primary approval; Unintended S with label change | | Some codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be available in the above Google Drive Folder (link above). ICD-9 to ICD-10 code conversions were completed using a SAS macro that implements, forward/backward mapping based on the CMS ICD-9 to ICD-10 mapping; https://www.nber.ore/data/icd9-icd-10-cm-and-ocs-crosswalk-general-equivalence-mapping.html. | |
| | EXPOSUR | Evs. COMPARISON | References/Rationale | Color coding |
| | Rivaroxaban (15 mg twice daily for 3 wks followed by 20 mg once daily) vs Warfarin (or acenocoumarol) | Rivaroxaban vs. Warfarin | | Criteria |
| | PRIM | ARY OUTCOME Measured 1 day after drug initiation in any diagnosis position and in an inpatient care setting | | Adequate mapping in claims |
| | Recurrent thromboembolism defined as the composite of (Deep vein thrombosis) DVT or nonfatal or fatal pulmonary embolism (PE) | Recurrent VTE (composite of DVT or PE): See 'VTE' sheet for codes | Fang MC, Fan D, Sung SH, et al. Validity of Using Inpatient and Outpatient Administrative Codes to Identify<br>Acute Venous Thromboembolism: The CVRN VTE Study. Med Care. 2017;55(12):e137-e143. | Intermediate mapping in claims |
| | | | | Poor mapping or cannot be measured |
| - | INCLU | ISION CRITERIA Measured 14 days prior to and including the day of drug initiation in any diagnosis position and in an inpatient or ED | | in claims |
| | Confirmed acute symptomatic proximal DVT without symptomatic PE | DVT: \(\text{LCD-9 Dx:}\) 45.1.1x, 451.2x, 451.81, 451.9x, 453.1x, 453.2x, 453.8x, 453.9x, 453.40, 453.41, 453.42, 453.0 \(\text{LCD-10 Dx:}\) 180.1*, 180.2, 180.3, 180.9, 182.0, 182.1, 182.2*EXCEPT182.2%1, 182.4*, 182.6*, 182.890, 182.90, 182.A1*, 182.81*, 182.C1*, 1800XXA (and 126.90 or 126.99), 181718A (and 126.90 or 126.99), 182818A (and 126.90 or 126.99), 182818A (and 126.90 or 126.99) | We will apply PE as exclusion criteria. | Can't be measured in claims but not important for the analysis |
| 2 | Written informed consent | N/A | | |
| | | ISION CRITERIA Measured on day of drug initiation | | |
| 1 | Legal lower age limitations | Age 118 Measured 14 days prior to and including the day of drug initiation in any diagnosis position and in an inpatient or | | |
| 2 | Thrombobectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current episode of DVT or PE | outpatient care setting as defined below: Thrombectomy: ICD-9 Fx. 39.74 ICD-10 Px: 03CG3ZZ, 03CH3ZZ, 03CH3ZZ, 03CH4ZZ, 03CJ3ZZ, 03CJ4ZZ, 03CK3ZZ, 03CK4ZZ, 03CL3ZZ, 03CL4ZZ, 03CM3ZZ, 03CM3ZZ, 03CM3ZZ, 03CM4ZZ, 03CM3ZZ, 03CM3ZZ, 03CM4ZZ, 03CM3ZZ, | | |
| 3 | Other indications for VKA than DVT and/or PE More than 48 hours pre-randomization treatment with therapeutic dosages of anti-coagulant treatment or | Measured 180 days prior to drug initiation in any diagnosis position and inpatient or outpatient care setting as defined below: Atrial fibrillation: [CD-9 Dx: 427.3x Acute coronary syndrome: [CD-9 Dx: 411.xx [CD-10 Dx: 124.9 Heart failure: [CD-9 Dx: 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 Prosthetic heart valve: [CD-9 Dx: 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 Prosthetic heart valve: [CD-9 Dx: 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 Prosthetic heart valve: [CD-9 Dx: 428.x, 398.91, 402.01, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 Prosthetic heart valve: [CD-9 Dx: 428.x, 436.xx N/A | | |
| 4 | More than 48 hours pre-randomization treatment with therapeutic dosages of anti-coagulant treatment or more than a single dose of VKA prior to randomization | | | |

| | | N/A |
|---|---|---|
| | Participation in another pharmacotherapeutic study within 30 days | |
| 6 | Creatinine clearance <30 ml/min | Measured 180 days prior to and including the day of drug initiation in any diagnosis position and in an inpatient or outpatient care setting as defined below: CKD states 4/5/ESRD: ICD-9 Dx: S85.4x, S85.5x, S85.6x ICD-10 Dx: N18.4x, N18.5x, N18.6x |
| 7 | Significant liver disease (e.g. acute hepatitis, chronic active hepatitis, cirrhosis) or ALAT>3x ULN | Measured 180 days prior to and including the day of drug initiation in any diagnosis position and in an inpatient or outpatient care setting as defined below: Moderate/severe liver disease: 100-9 Dx; 100- |
| 8 | Bacterial endocarditis | Measured 180 days prior to and including the day of drug initiation in any diagnosis position and in an inpatient or outpatient care setting as defined below: Bacterial endocarditis: 109 0x: 110-10 0x: 133.x |
| 9 | Life expectancy <3 months | Measured over 365 days prior to drug initiation: CCI >= 10 |
| 10 | Active bleeding or high risk for bleeding contraindicating treatment with enoxaparin or VKA | Measured 180 days prior to and including the day of drug initiation in any diagnosis position and in an inpatient or outpatient care setting as defined below: Active bleeding or bleeding history—see 'Major Bleeding' sheet |
| 11 | Systolic blood pressure > 180 mgHg or diastolic blood pressure > 110 mgHg | Measured 180 days prior to and including the day of drug initiation in any diagnosis position and in an inpatient or outpatient care setting as defined below: Malignant Hypertension: 109-101. 401.0, 402.0, 402.01, 403.0, 403.00, 403.01, 404.0, 404.00, 404.01, 404.02, 404.03, 405.0, 405.01, 405.09 |
| 12 | Childbearing potential without proper contraceptive measures, pregnancy or breastfeeding | Measured 180 days prior to and including they day of drug initiation in any diagnosis position and in an inpatient or outpatient care setting as defined below: Pregnancy or lactation—see 'Pregnancy' sheet |
| 13 | Any other contraindication listed in the local labeling of enoxaparin, warfarin, or acenocoumarol | N/A |
| 14 | Concomitant use of strong CYP3A4 inhibitors (e.g. HIV protease inhibitors, systemic ketoconazole) or strong CYP3A4 inducers rifampin | Prescription claim for following CYP3A inhibitors or strong CYP3A inducers Measured 14 days prior to and also on the drug initiation date Inhibitors: Ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nefinavir, indinavir, atazanavir Inducers: Rifampin, rifampicin/rifampin, phenytoin, carbamazepine |
| 15 | Symptomatic pulmonary embolism | Measured 14 days prior to and including the day of drug initiation in any diagnosis position and in an inpatient care setting as defined below: Pulmonary embolism: ICD 9 Dx: 415.1x ICD-10 Dx: 126.* EXCEPT 126.90 |

| Trial Catergory | Secondary initiation |
|---|---|
| RCT Category | 5a- Successful NI with label change |
| Trial Name (with web links) | <u>EINSTEIN DVT</u> |
| Study Batch | NOACs |
| <u>NCT</u> | <u>NCT00440193</u> |
| Therapeutic Area | Cardiology/Vascular Diseases |
| Brand Name | Xarelto |
| <b>Generic Name</b> | Rivaroxaban |
| <u>Sponsor</u> | Bayer |
| <u>Year</u> | 2010 |
| Measurable endpoint | Percentage of Participants With Symptomatic Recurrent Venous Thromboembolism [VTE] (i.e. the Composite of |
| | Recurrent Deep Vein Thrombosis [DVT] or Fatal or Non-fatal Pulmonary Embolism [PE]) Until the Intended End of Study |
| | Treatment |
| <u>Exposure</u> | Rivaroxaban |
| <u>Comparator</u> | Enoxaparin/VKA |
| Trial finding | HR = 0.68 (95% CI 0.44–1.04) |
| No. of Patients | 3,449 |
| Non-inferiority margin | HR = 2.0 |
| Finding for potential Assay Sens. Outcome | HR 0.72, 95% CI 0.53-0.99 |
| from trial- | HR 0.72, 95% CI 0.53-0.99 |
| Assay Sens. Finding | Percentage of Participants With the Composite Variable Comprising Recurrent DVT, Non-fatal PE and All Cause Mortality |
| | Until the Intended End of Study Treatment |
| <u>Power</u> | 0.90. Assuming equal efficacy, a total of 88 events was calculated to give a power of 90% to prove that rivaroxaban is at |
| | least as effective as the comparator, considering a non-inferiority upper CI margin for the hazard ratio of 2.0 (two-sided |
| | lpha=0.05). A mean incidence for the primary efficacy outcome of 3% was expected and at least 1465 participants per |
| | group were determined to be necessary. This number was to be adjusted based on the observed overall incidence of |
| | symptomatic recurrent VTE. |

| Title | |
|---|---|
| Venous Thromboembolism (VTE) | |
| ICD-9 Dx inpatient primary position | |
| PE | |
| 415.1 | PULMONARY EMBOLISM AND INFARCTION |
| 415.11 | IATROGENIC PULMONARY EMBOLISM AND INFARCTION |
| 415.19 | OTHER PULMONARY EMBOLISM AND INFARCTION |
| DVT | |
| 451.1 | PHLEBITIS AND THROMBOPHLEBITIS OF DEEP VEINS OF LOWER EXTREMITIES |
| 451.11 | PHLEBITIS AND THROMBOPHLEBITIS OF FEMORAL VEIN (DEEP) (SUPERFICIAL) |
| 451.19 | PHLEBITIS AND THROMBOPHLEBITIS OF OTHER |
| 451.2 | PHLEBITIS AND THROMBOPHLEBITIS OF LOWER EXTREMITIES UNSPECIFIED |
| 451.81 | PHLEBITIS AND THROMBOPHLEBITIS OF ILIAC VEIN |
| 451.9 | PHLEBITIS AND THROMBOPHLEBITIS OF UNSPECIFIED SITE |
| 453 | BUDD-CHIARI SYNDROME |
| 453.1 | THROMBOPHLEBITIS MIGRANS |
| 453.2 | EMBOLISM AND THROMBOSIS OF INFERIOR VENA CAVA |
| 453.4 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF DEEP VESSELS OF LOWER EXTREMITY |
| 453.4 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF UNSPECIFIED DEEP VESSELS OF LOWER EXTREMITY |
| 453.41 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF DEEP VESSELS OF PROXIMAL LOWER EXTREMITY |
| 453.42 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF DEEP VESSELS OF DISTAL LOWER EXTREMITY |
| 453.5 | CHRONIC VENOUS EMBOLISM AND THROMBOSIS OF DEEP VESSELS OF LOWER EXTREMITY |
| 453.5 | CHRONIC VENOUS EMBOLISM AND THROMBOSIS OF UNSPECIFIED DEEP VESSELS OF LOWER EXTREMITY |
| 453.51 | CHRONIC VENOUS EMBOLISM AND THROMBOSIS OF DEEP VESSELS OF PROXIMAL LOWER EXTREMITY |
| 453.52 | CHRONIC VENOUS EMBOLISM AND THROMBOSIS OF DEEP VESSELS OF DISTAL LOWER EXTREMITY |
| 453.8 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF OTHER SPECIFIED VEINS |
| 453.82 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF DEEP VEINS OF UPPER EXTREMITY |
| 453.83 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF UPPER EXTREMITY UNSPECIFIED |
| 453.84 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF AXILLARY VEINS |
| 453.85 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF SUBCLAVIAN VEINS |
| 453.86 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF INTERNAL JUGULAR VEINS |
| 453.87 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF OTHER THORACIC VEINS |
| 453.89 | ACUTE VENOUS EMBOLISM AND THROMBOSIS OF OTHER SPECIFIED VEINS |

| 453.9 | EMBOLISM AND THROMBOSIS OF UNSPECIFIED SITE |
|---|---|
| ICD-10 Dx inpatient pri | imary nosition |
| PE | mially position |
| 126.0 | Pulmonary embolism with acute cor pulmonale |
| 126.01 | Septic pulmonary embolism with acute cor pulmonale |
| 126.02 | Saddle embolus of pulmonary artery with acute cor pulmonale |
| 126.09 | Other pulmonary embolism with acute cor pulmonale |
| 126.9 | Pulmonary embolism without acute cor pulmonale |
| 126.99 | Other pulmonary embolism without acute cor pulmonale |
| DVT | |
| 180.1 | Phlebitis and thrombophlebitis of femoral vein |
| 180.10 | Phlebitis and thrombophlebitis of unspecified femoral vein |
| 180.11 | Phlebitis and thrombophlebitis of right femoral vein |
| 180.12 | Phlebitis and thrombophlebitis of left femoral vein |
| 180.13 | Phlebitis and thrombophlebitis of femoral vein, bilateral |
| 180.2 | Phlebitis and thrombophlebitis of other and unspecified deep vessels of lower extremities |
| 180.20 | Phlebitis and thrombophlebitis of unspecified deep vessels of lower extremities |
| 180.201 | Phlebitis and thrombophlebitis of unspecified deep vessels of right lower extremity |
| 180.202 | Phlebitis and thrombophlebitis of unspecified deep vessels of left lower extremity |
| 180.203 | Phlebitis and thrombophlebitis of unspecified deep vessels of lower extremities, bilateral |
| 180.209 | Phlebitis and thrombophlebitis of unspecified deep vessels of unspecified lower extremity |
| 180.21 | Phlebitis and thrombophlebitis of iliac vein |
| 180.211 | Phlebitis and thrombophlebitis of right iliac vein |
| 180.212 | Phlebitis and thrombophlebitis of left iliac vein |
| 180.213 | Phlebitis and thrombophlebitis of iliac vein, bilateral |
| 180.219 | Phlebitis and thrombophlebitis of unspecified iliac vein |
| 180.22 | Phlebitis and thrombophlebitis of popliteal vein |
| 180.221 | Phlebitis and thrombophlebitis of right popliteal vein |
| 180.222 | Phlebitis and thrombophlebitis of left popliteal vein |
| 180.223 | Phlebitis and thrombophlebitis of popliteal vein, bilateral |
| 180.229 | Phlebitis and thrombophlebitis of unspecified popliteal vein |
| 180.23 | Phlebitis and thrombophlebitis of tibial vein |
| 180.231 | Phlebitis and thrombophlebitis of right tibial vein |

| 180.232 | Phlebitis and thrombophlebitis of left tibial vein |
|---|---|
| 180.233 | Phlebitis and thrombophlebitis of tibial vein, bilateral |
| 180.239 | Phlebitis and thrombophlebitis of unspecified tibial vein |
| 180.29 | Phlebitis and thrombophlebitis of other deep vessels of lower extremities |
| 180.291 | Phlebitis and thrombophlebitis of other deep vessels of right lower extremity |
| 180.292 | Phlebitis and thrombophlebitis of other deep vessels of left lower extremity |
| 180.293 | Phlebitis and thrombophlebitis of other deep vessels of lower extremity, bilateral |
| 180.299 | Phlebitis and thrombophlebitis of other deep vessels of unspecified lower extremity |
| 180.3 | Phlebitis and thrombophlebitis of lower extremities, unspecified |
| 180.9 | Phlebitis and thrombophlebitis of unspecified site |
| 182.0 | Exposure) Rivaroxaban+E+E6 |
| 182.1 | Thrombophlebitis migrans |
| 180.3 | Phlebitis and thrombophlebitis of lower extremities, unspecified |
| 182.4 | Acute embolism and thrombosis of deep veins of lower extremity |
| 182.40 | Acute embolism and thrombosis of unspecified deep veins of lower extremity |
| 182.401 | Acute embolism and thrombosis of unspecified deep veins of right lower extremity |
| 182.402 | Acute embolism and thrombosis of unspecified deep veins of left lower extremity |
| 182.403 | Acute embolism and thrombosis of unspecified deep veins of lower extremity, bilateral |
| 182.409 | Acute embolism and thrombosis of unspecified deep veins of unspecified lower extremity |
| 182.41 | Acute embolism and thrombosis of femoral vein |
| 182.411 | Acute embolism and thrombosis of right femoral vein |
| 182.412 | Acute embolism and thrombosis of left femoral vein |
| 182.413 | Acute embolism and thrombosis of femoral vein, bilateral |
| 182.419 | Acute embolism and thrombosis of unspecified femoral vein |
| 182.42 | Acute embolism and thrombosis of iliac vein |
| 182.421 | Acute embolism and thrombosis of right iliac vein |
| 182.422 | Acute embolism and thrombosis of left iliac vein |
| 182.423 | Acute embolism and thrombosis of iliac vein, bilateral |
| 182.429 | Acute embolism and thrombosis of unspecified iliac vein |
| 182.43 | Acute embolism and thrombosis of popliteal vein |
| 182.431 | Acute embolism and thrombosis of right popliteal vein |
| 182.432 | Acute embolism and thrombosis of left popliteal vein |
| 182.433 | Acute embolism and thrombosis of popliteal vein, bilateral |
| 182.439 | Acute embolism and thrombosis of unspecified popliteal vein |
| 182.44 | Acute embolism and thrombosis of tibial vein |

| 182.441 | Acute embolism and thrombosis of right tibial vein |
|---|---|
| 182.442 | Acute embolism and thrombosis of left tibial vein |
| 182.443 | Acute embolism and thrombosis of tibial vein, bilateral |
| 182.449 | Acute embolism and thrombosis of unspecified tibial vein |
| 182.49 | Acute embolism and thrombosis of other specified deep vein of lower extremity |
| 182.491 | Acute embolism and thrombosis of other specified deep vein of right lower extremity |
| 182.492 | Acute embolism and thrombosis of other specified deep vein of left lower extremity |
| 182.493 | Acute embolism and thrombosis of other specified deep vein of lower extremity, bilateral |
| 182.499 | Acute embolism and thrombosis of other specified deep vein of unspecified lower extremity |
| 182.4Y | Acute embolism and thrombosis of unspecified deep veins of proximal lower extremity |
| I82.4Y1 | Acute embolism and thrombosis of unspecified deep veins of right proximal lower extremity |
| 182.4Y2 | Acute embolism and thrombosis of unspecified deep veins of left proximal lower extremity |
| I82.4Y3 | Acute embolism and thrombosis of unspecified deep veins of proximal lower extremity, bilateral |
| 182.4Y9 | Acute embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremity |
| I82.4Z | Acute embolism and thrombosis of unspecified deep veins of distal lower extremity |
| 182.4Z1 | Acute embolism and thrombosis of unspecified deep veins of right distal lower extremity |
| 182.4Z2 | Acute embolism and thrombosis of unspecified deep veins of left distal lower extremity |
| 182.4Z3 | Acute embolism and thrombosis of unspecified deep veins of distal lower extremity, bilateral |
| 182.479 | Acute embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity |
| 182.5 | Chronic embolism and thrombosis of deep veins of lower extremity |
| 182.50 | Chronic embolism and thrombosis of unspecified deep veins of lower extremity |
| 182.501 | Chronic embolism and thrombosis of unspecified deep veins of right lower extremity |
| 182.502 | Chronic embolism and thrombosis of unspecified deep veins of left lower extremity |
| 182.503 | Chronic embolism and thrombosis of unspecified deep veins of lower extremity, bilateral |
| 182.509 | Chronic embolism and thrombosis of unspecified deep veins of unspecified lower extremity |
| 182.51 | Chronic embolism and thrombosis of femoral vein |
| 182.511 | Chronic embolism and thrombosis of right femoral vein |
| 182.512 | Chronic embolism and thrombosis of left femoral vein |
| 182.513 | Chronic embolism and thrombosis of femoral vein, bilateral |
| 182.519 | Chronic embolism and thrombosis of unspecified femoral vein |
| 182.52 | Chronic embolism and thrombosis of iliac vein |
| 182.521 | Chronic embolism and thrombosis of right iliac vein |
| 182.522 | Chronic embolism and thrombosis of left iliac vein |
| 182.523 | Chronic embolism and thrombosis of iliac vein, bilateral |
| 182.529 | Chronic embolism and thrombosis of unspecified iliac vein |

| 182.53 | Chronic embolism and thrombosis of popliteal vein |
|---|---|
| 182.531 | Chronic embolism and thrombosis of right popliteal vein |
| 182.532 | Chronic embolism and thrombosis of left popliteal vein |
| 182.533 | Chronic embolism and thrombosis of popliteal vein, bilateral |
| 182.539 | Chronic embolism and thrombosis of unspecified popliteal vein |
| 182.54 | Chronic embolism and thrombosis of tibial vein |
| 182.541 | Chronic embolism and thrombosis of right tibial vein |
| 182.542 | Chronic embolism and thrombosis of left tibial vein |
| 182.543 | Chronic embolism and thrombosis of tibial vein, bilateral |
| 182.549 | Chronic embolism and thrombosis of unspecified tibial vein |
| 182.59 | Chronic embolism and thrombosis of other specified deep vein of lower extremity |
| 182.591 | Chronic embolism and thrombosis of other specified deep vein of right lower extremity |
| 182.592 | Chronic embolism and thrombosis of other specified deep vein of left lower extremity |
| 182.593 | Chronic embolism and thrombosis of other specified deep vein of lower extremity, bilateral |
| 182.599 | Chronic embolism and thrombosis of other specified deep vein of unspecified lower extremity |
| 182.5Y | Chronic embolism and thrombosis of unspecified deep veins of proximal lower extremity |
| 182.5Y1 | Chronic embolism and thrombosis of unspecified deep veins of right proximal lower extremity |
| 182.5Y2 | Chronic embolism and thrombosis of unspecified deep veins of left proximal lower extremity |
| 182.5Y3 | Chronic embolism and thrombosis of unspecified deep veins of proximal lower extremity, bilateral |
| 182.5Y9 | Chronic embolism and thrombosis of unspecified deep veins of unspecified proximal lower extremity |
| I82.5Z | Chronic embolism and thrombosis of unspecified deep veins of distal lower extremity |
| 182.5Z1 | Chronic embolism and thrombosis of unspecified deep veins of right distal lower extremity |
| 182.5Z2 | Chronic embolism and thrombosis of unspecified deep veins of left distal lower extremity |
| 182.5Z3 | Chronic embolism and thrombosis of unspecified deep veins of distal lower extremity, bilateral |
| 182.529 | Chronic embolism and thrombosis of unspecified deep veins of unspecified distal lower extremity |
| 182.6 | Acute embolism and thrombosis of veins of upper extremity |
| 182.60 | Acute embolism and thrombosis of unspecified veins of upper extremity |
| 182.601 | Acute embolism and thrombosis of unspecified veins of right upper extremity |
| 182.602 | Acute embolism and thrombosis of unspecified veins of left upper extremity |
| 182.603 | Acute embolism and thrombosis of unspecified veins of upper extremity, bilateral |
| 182.609 | Acute embolism and thrombosis of unspecified veins of unspecified upper extremity |
| 182.62 | Acute embolism and thrombosis of deep veins of upper extremity |
| 182.621 | Acute embolism and thrombosis of deep veins of right upper extremity |
| 182.622 | Acute embolism and thrombosis of deep veins of left upper extremity |
| 182.623 | Acute embolism and thrombosis of deep veins of upper extremity, bilateral |

| 182.629 | Acute embolism and thrombosis of deep veins of unspecified upper extremity |
|---|---|
| 182.890 | Acute embolism and thrombosis of other specified veins |
| 182.90 | Acute embolism and thrombosis of unspecified vein |
| 182.A1 | Acute embolism and thrombosis of axillary vein |
| I82.A11 | Acute embolism and thrombosis of right axillary vein |
| I82.A12 | Acute embolism and thrombosis of left axillary vein |
| I82.A13 | Acute embolism and thrombosis of axillary vein, bilateral |
| I82.A19 | Acute embolism and thrombosis of unspecified axillary vein |
| 182.B1 | Acute embolism and thrombosis of subclavian vein |
| I82.B11 | Acute embolism and thrombosis of right subclavian vein |
| I82.B12 | Acute embolism and thrombosis of left subclavian vein |
| I82.B13 | Acute embolism and thrombosis of subclavian vein, bilateral |
| I82.B19 | Acute embolism and thrombosis of unspecified subclavian vein |
| 182.C1 | Acute embolism and thrombosis of internal jugular vein |
| 182.C11 | Acute embolism and thrombosis of right internal jugular vein |
| 182.C12 | Acute embolism and thrombosis of left internal jugular vein |
| 182.C13 | Acute embolism and thrombosis of internal jugular vein, bilateral |
| I82.C19 | Acute embolism and thrombosis of unspecified internal jugular vein |

| Title | |
|---|---|
| Major Bleeding | |
| , , | |
| ICD-9 Dx: 1 inpatient or 2 outpatient | |
| 562.02 | DIVERTICULOSIS OF SMALL INTESTINE WITH HEMORRHAGE |
| 562.03 | DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE |
| 562.12 | DIVERTICULOSIS OF COLON WITH HEMORRHAGE |
| 562.13 | DIVERTICULITIS OF COLON WITH HEMORRHAGE |
| 568.81 | HEMOPERITONEUM (NONTRAUMATIC |
| 569.3 | HEMORRHAGE OF RECTUM AND ANUS |
| 569.83 | PERFORATION OF INTESTINE |
| 569.85 | ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE OF INTESTINE |
| 569.86 | DIEULAFOY LESION (HEMORRHAGIC |
| 578 | HEMATEMESIS |
| 578.9 | HEMORRHAGE OF GASTROINTESTINAL TRACT UNSPECIFIED |
| 423 | HEMOPERICARDIUM |
| 432 | NONTRAUMATIC EXTRADURAL HEMORRHAGE |
| 432.1 | SUBDURAL HEMORRHAGE |
| 432.9 | UNSPECIFIED INTRACRANIAL HEMORRHAGE |
| 459 | HEMORRHAGE UNSPECIFIED |
| 531 | ACUTE GASTRIC ULCER WITH HEMORRHAGE |
| 531 | ACUTE GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 531.01 | ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 531.2 | ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION |
| 531.2 | ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 531.21 | ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 531.4 | CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE |
| 531.4 | CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 531.41 | CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 531.6 | CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION |
| 531.6 | CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 531.61 | CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 532 | ACUTE DUODENAL ULCER WITH HEMORRHAGE |
| 532 | ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 532.01 | ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 532.2 | ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 532.2 | ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 532.21 | ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 532.4 | CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE |
| 532.4 | CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 532.41 | CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |

| 532.6 | CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION |
|---|---|
| 532.6 | CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 532.61 | CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 533 | ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE |
| 533 | ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 533.01 | ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION |
| 533.2 | ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION |
| 533.2 | ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 533.21 | ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 533.4 | CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE |
| 533.4 | CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 533.41 | CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION |
| 533.6 | CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION |
| 533.6 | CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 533.61 | CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 534 | ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE |
| 534 | ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 534.01 | ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 534.2 | ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 534.2 | ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 534.21 | ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 534.4 | CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE |
| 534.4 | CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 534.41 | CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION |
| 534.6 | CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 534.6 | CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 534.61 | CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 578.1 | BLOOD IN STOOL |
| 719.1 | HEMARTHROSIS |
| 719.1 | HEMARTHROSIS SITE UNSPECIFIED |
| 719.11 | HERARTHROSIS INVOLVING SHOULDER REGION |
| 719.12 | HEMARTHORSIS INVOLVING UPPER ARM |
| 719.13 | HEMARTHROSIS INVOLVING FOREARM |
| 719.14 | HEMARTHROSIS INVOLVING HAND |
| 719.15 | HEMARTHROSIS INVOLVING PELVIC REGION AND THIGH |
| 719.16 | HEMARTHROSIS INVOLVING LOWER LEG |
| 719.17 | HEMARTHROSIS INVOLVING ANKLE AND FOOT |
| 719.18 | HEMARTHROSIS INVOLVING OTHER SPECIFIED SITES |
| 719.19 | HEMARTHROSIS INVOLVING MULTIPLE SITES |
| 430 | SUBARACHNOID HEMORRHAGE |
| 431 | INTRACEREBRAL HEMORRHAGE |

| HEMORRHAGE FROM THROAT | 784.7 | EPISTAXIS |
|---|---|---|
| S99.7 HEMATURIA | | |
| S99.71 SORS HEMATURIA UNSPECIFIED | | |
| S99.71 GROSS HEMATURIA | | |
| MICROSCOPIC HEMATURIA | | |
| HEMOPTYSIS UNSPECIFIED | | |
| PRESCRIPTION PRES | | |
| ACUTE IDIOPATHIC PULMONARY HEMORRHAGE IN INFANTS | | |
| ICD-10 Dx: 1 inpatient or 2 outpatient | | |
| ICD-10 Dx: 1 inpatient or 2 outpatient 13.1.2 | | |
| 13.1.2 Hemopericardium, not elsewhere classified | 760.33 | OTTENTIEND 11313 |
| 13.1.2 Hemopericardium, not elsewhere classified | ICD-10 Dx: 1 innatient or 2 outnatient | |
| Nontraumatic subarachnoid hemorrhage from unspecified carotid siphon and bifurcation | | Hamonericardium, not elsewhere classified |
| Nontraumatic subarachnoid hemorrhage from right carotid siphon and bifurcation | | ' ' |
| Nontraumatic subarachnoid hemorrhage from left carotid siphon and bifurcation | | |
| 160.10 Nontraumatic subarachnoid hemorrhage from unspecified middle cerebral artery | | |
| 160.11 Nontraumatic subarachnoid hemorrhage from right middle cerebral artery | | · |
| 160.12 Nontraumatic subarachnoid hemorrhage from left middle cerebral artery | | |
| 160.2 Nontraumatic subarachnoid hemorrhage from unspecified posterior communicating artery | | , , |
| Nontraumatic subarachnoid hemorrhage from unspecified posterior communicating artery | | - |
| Nontraumatic subarachnoid hemorrhage from right posterior communicating artery | | |
| Nontraumatic subarachnoid hemorrhage from left posterior communicating artery | | |
| Nontraumatic subarachnoid hemorrhage from basilar artery | | |
| Nontraumatic subarachnoid hemorrhage from unspecified vertebral artery | | |
| Nontraumatic subarachnoid hemorrhage from right vertebral artery | | |
| Nontraumatic subarachnoid hemorrhage from left vertebral artery | | |
| Nontraumatic subarachnoid hemorrhage from other intracranial arteries | | |
| Nontraumatic subarachnoid hemorrhage from unspecified intracranial artery 160.8 | | |
| Other nontraumatic subarachnoid hemorrhage | | |
| Nontraumatic subarachnoid hemorrhage, unspecified 161.0 | | |
| 161.0 Nontraumatic intracerebral hemorrhage in hemisphere, subcortical 161.1 Nontraumatic intracerebral hemorrhage in hemisphere, cortical 161.2 Nontraumatic intracerebral hemorrhage in hemisphere, unspecified 161.3 Nontraumatic intracerebral hemorrhage in brain stem 161.4 Nontraumatic intracerebral hemorrhage in cerebellum 161.5 Nontraumatic intracerebral hemorrhage, intraventricular 161.6 Nontraumatic intracerebral hemorrhage, multiple localized 161.8 Other nontraumatic intracerebral hemorrhage 161.9 Nontraumatic intracerebral hemorrhage, unspecified 161.0 Nontraumatic intracerebral hemorrhage 161.0 Nontraumatic intracereb | | Ţ. |
| I61.1Nontraumatic intracerebral hemorrhage in hemisphere, corticalI61.2Nontraumatic intracerebral hemorrhage in hemisphere, unspecifiedI61.3Nontraumatic intracerebral hemorrhage in brain stemI61.4Nontraumatic intracerebral hemorrhage in cerebellumI61.5Nontraumatic intracerebral hemorrhage, intraventricularI61.6Nontraumatic intracerebral hemorrhage, multiple localizedI61.8Other nontraumatic intracerebral hemorrhageI61.9Nontraumatic intracerebral hemorrhage, unspecified | | |
| Nontraumatic intracerebral hemorrhage in hemisphere, unspecified Nontraumatic intracerebral hemorrhage in brain stem Nontraumatic intracerebral hemorrhage in cerebellum Nontraumatic intracerebral hemorrhage, intraventricular Nontraumatic intracerebral hemorrhage, multiple localized Nontraumatic intracerebral hemorrhage Nontraumatic intracerebral hemorrhage Nontraumatic intracerebral hemorrhage Nontraumatic intracerebral hemorrhage | | |
| Nontraumatic intracerebral hemorrhage in brain stem 161.4 Nontraumatic intracerebral hemorrhage in cerebellum 161.5 Nontraumatic intracerebral hemorrhage, intraventricular 161.6 Nontraumatic intracerebral hemorrhage, multiple localized 161.8 Other nontraumatic intracerebral hemorrhage 161.9 Nontraumatic intracerebral hemorrhage, unspecified 161.9 Nontraumatic intracerebral hemorrhage 161.9 Nontrauma | | |
| I61.4 Nontraumatic intracerebral hemorrhage in cerebellum I61.5 Nontraumatic intracerebral hemorrhage, intraventricular I61.6 Nontraumatic intracerebral hemorrhage, multiple localized I61.8 Other nontraumatic intracerebral hemorrhage I61.9 Nontraumatic intracerebral hemorrhage, unspecified | | |
| 161.5 Nontraumatic intracerebral hemorrhage, intraventricular Nontraumatic intracerebral hemorrhage, multiple localized 161.8 Other nontraumatic intracerebral hemorrhage Nontraumatic intracerebr | 161.4 | |
| I61.6 Nontraumatic intracerebral hemorrhage, multiple localized I61.8 Other nontraumatic intracerebral hemorrhage I61.9 Nontraumatic intracerebral hemorrhage, unspecified | | · |
| I61.8 Other nontraumatic intracerebral hemorrhage I61.9 Nontraumatic intracerebral hemorrhage, unspecified | 161.6 | |
| Nontraumatic intracerebral hemorrhage, unspecified | 161.8 | |
| | 161.9 | · |
| Ib2.UU Nontraumatic subdural hemorrhage, unspecified | 162.00 | Nontraumatic subdural hemorrhage, unspecified |

| 162.01 | Nontraumatic acute subdural hemorrhage |
|---|---|
| 162.02 | Nontraumatic subacute subdural hemorrhage |
| 162.03 | Nontraumatic chronic subdural hemorrhage |
| 162.1 | Nontraumatic extradural hemorrhage |
| 162.9 | Nontraumatic intracranial hemorrhage, unspecified |
| K25.0 | Acute gastric ulcer with hemorrhage |
| K25.2 | Acute gastric ulcer with both hemorrhage and perforation |
| K25.4 | Chronic or unspecified gastric ulcer with hemorrhage |
| K25.6 | Chronic or unspecified gastric ulcer with both hemorrhage and perforation |
| K26.0 | Acute duodenal ulcer with hemorrhage |
| K26.2 | Acute duodenal ulcer with both hemorrhage and perforation |
| K26.4 | Chronic or unspecified duodenal ulcer with hemorrhage |
| K26.6 | Chronic or unspecified duodenal ulcer with both hemorrhage and perforation |
| K27.0 | Acute peptic ulcer, site unspecified, with hemorrhage |
| K27.2 | Acute peptic ulcer, site unspecified, with both hemorrhage and perforation |
| K27.4 | Chronic or unspecified peptic ulcer, site unspecified, with hemorrhage |
| K27.6 | Chronic or unspecified peptic ulcer, site unspecified, with both hemorrhage and perforation |
| K28.0 | Acute gastrojejunal ulcer with hemorrhage |
| K28.2 | Acute gastrojejunal ulcer with both hemorrhage and perforation |
| K28.4 | Chronic or unspecified gastrojejunal ulcer with hemorrhage |
| K28.6 | Chronic or unspecified gastrojejunal ulcer with both hemorrhage and perforation |
| K55.21 | Angiodysplasia of colon with hemorrhage |
| K56.60 | Unspecified intestinal obstruction |
| K57.01 | Diverticulitis of small intestine with perforation and abscess with bleeding |
| K57.11 | Diverticulosis of small intestine without perforation or abscess with bleeding |
| K57.13 | Diverticulitis of small intestine without perforation or abscess with bleeding |
| K57.21 | Diverticulitis of large intestine with perforation and abscess with bleeding |
| K57.31 | Diverticulosis of large intestine without perforation or abscess with bleeding |
| K57.33 | Diverticulitis of large intestine without perforation or abscess with bleeding |
| K57.41 | Diverticulitis of both small and large intestine with perforation and abscess with bleeding |
| K57.51 | Diverticulosis of both small and large intestine without perforation or abscess with bleeding |
| K57.53 | Diverticulitis of both small and large intestine without perforation or abscess with bleeding |
| K57.81 | Diverticulitis of intestine, part unspecified, with perforation and abscess with bleeding |
| K57.91 | Diverticulosis of intestine, part unspecified, without perforation or abscess with bleeding |
| K57.93 | Diverticulitis of intestine, part unspecified, without perforation or abscess with bleeding |
| K62.5 | Hemorrhage of anus and rectum |
| K63.1 | Perforation of intestine (nontraumatic |
| K63.81 | Dieulafoy lesion of intestine |
| K66.1 | Hemoperitoneum |
| K92.0 | Hematemesis |
| K92.1 | Melena |

| K92.2 | Gastrointestinal hemorrhage, unspecified |
|---------|-----------------------------------------------------|
| M25.00 | Hemarthrosis, unspecified joint |
| M25.011 | Hemarthrosis, right shoulder |
| M25.012 | Hemarthrosis, left shoulder |
| M25.019 | Hemarthrosis, unspecified shoulder |
| M25.021 | Hemarthrosis, right elbow |
| M25.022 | Hemarthrosis, left elbow |
| M25.029 | Hemarthrosis, unspecified elbow |
| M25.031 | Hemarthrosis, right wrist |
| M25.032 | Hemarthrosis, left wrist |
| M25.039 | Hemarthrosis, unspecified wrist |
| M25.041 | Hemarthrosis, right hand |
| M25.042 | Hemarthrosis, left hand |
| M25.049 | Hemarthrosis, unspecified hand |
| M25.051 | Hemarthrosis, right hip |
| M25.052 | Hemarthrosis, left hip |
| M25.059 | Hemarthrosis, unspecified hip |
| M25.061 | Hemarthrosis, right knee |
| M25.062 | Hemarthrosis, left knee |
| M25.069 | Hemarthrosis, unspecified knee |
| M25.071 | Hemarthrosis, right ankle |
| M25.072 | Hemarthrosis, left ankle |
| M25.073 | Hemarthrosis, unspecified ankle |
| M25.074 | Hemarthrosis, right foot |
| M25.075 | Hemarthrosis, left foot |
| M25.076 | Hemarthrosis, unspecified foot |
| M25.08 | Hemarthrosis, other specified site |
| R58 | Hemorrhage, not elsewhere classified |
| R04 | Hemorrhage from respiratory passages |
| R04.0 | Epistaxis |
| R04.1 | Hemorrhage from throat |
| R04.2 | Hemoptysis |
| R04.8 | Hemorrhage from other sites in respiratory passages |
| R04.81 | Acute idiopathic pulmonary hemorrhage in infants |
| R04.89 | Hemorrhage from other sites in respiratory passages |
| R04.9 | Hemorrhage from respiratory passages, unspecified |
| R31 | Hematuria |
| R31.0 | Gross hematuria |
| R31.1 | Benign essential microscopic hematuria |
| R31.2 | Other microscopic hematuria |
| R31.21 | Asymptomatic microscopic hematuria |

| R31.29 | Other microscopic hematuria |
|---|---|
| R31.9 | Hematuria, unspecified |
| ICD-9 Px | |
| 44.43 | ENDOSCOPIC CONTROL OF GASTRIC OF DUODENAL BLEEDING |
| ICD-10 Px | |
| OW3P8ZZ | Control Bleeding in Gastrointestinal Tract, Via Natural or Artificial Opening Endoscopic |
| HCPCS | |
| | Esophagogastroduodenoscopy, flexible, transoral; with control of bleeding, any method / Upper gastrointestinal endoscopy |
| 43255 | including esophagus, stomach, and either the duodenum and/or jejunum as appropriate; with control of bleeding, any method |

# **Pregnancy** Dx codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY **Procedure codes** 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY 72.39 OTHER HIGH FORCEPS OPERATION

- 72.4 FORCEPS ROTATION OF FETAL HEAD
- 72.5 BREECH EXTRACTION
- 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.52 OTHER PARTIAL BREECH EXTRACTION
- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR
- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION
- 74.1 LOW CERVICAL CESAREAN SECTION
- 74.2 EXTRAPERITONEAL CESAREAN SECTION

- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS



| Column | | | | | | Unmatched | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Part | | Optun | | | MarketSca | n | | Medicare | | | | | |
| Martin M | Variable | Reference-warfarin Conv | | St Diff Refe | aranca-warfarin Conv. avah | an (15 or 20 mg) Conv | St Diff Bof | aranca-warfarin Conv. 1 | 5 or 20 mg/Conv | St Diff P. | afaranca-warfarin Conv | | St. Diff |
| Mathematical Math | | | | Jt. Dill. Reid | | | St. Dill. Rei | | | 3t. Dill. 10 | | | Jt. Dill. |
| March Marc | • | ,,-13 | 3,540 | | 13,5 | 3,500 | | 32,013 | 10,740 | | 54,005 | 24,550 | |
| March Marc | mean (sd) | 64.55 (15.26) | 64.30 (15.26) | 0.02 | 56.88 (15.95) | 54.05 (15.64) | 0.18 | 77.01 (8.04) | 75.83 (7.74) | 0.15 | 70.09 (11.70) | 70.52 (10.81) | -0.04 |
| 1.00 | Age categories without zero category | | | | | | | | | | | | |
| 1.00 | | , , | , | | | | | | , | | , , | , | 0.08 |
| | | , , | | | | | | | , | | -,, | , , , , | 0.09 |
| The Control of Contr | | | | | | | | | | | | | -0.15 |
| | | 2,275 (30.7%) | 1,067 (27.1%) | 0.08 | 2,082 (14.9%) | 399 (10.2%) | 0.14 | 18,298 (56.1%) | 8,383 (50.1%) | 0.12 | 22,655 (41.9%) | 9,849 (40.0%) | 0.04 |
| The Control | | 2 260 (45 29/) | 1 004 (45 00/) | 0.01 | 6 030 (40 00/) | 1 000 (40 60/) | 0.01 | 11 769 (26 19/) | 6 572 (20 20/) | 0.06 | 21 066 (40 79/) | 10 375 (41 99/) | -0.02 |
| | | | | | | | | | | | | | 0.02 |
| | | 4,032 (34.7%) | 2,130 (34.2%) | 0.01 | 7,135 (31.170) | 2,010 (31.4%) | -0.01 | 20,831 (03.5%) | 10,173 (00.8%) | 0.00 | 32,042 (35.370) | 14,321 (30.270) | 0.02 |
| | | | | | | | | 27.361 (83.9%) | 14.167 (84.6%) | | 27.361 (83.9%) | 14.167 (84.6%) | 0.00 |
| | Black; n (%) | | | | | | | | 1,731 (10.3%) | | | 1,731 (10.3%) | 0.00 |
| | Asian; n (%) | | | | | | | 255 (0.8%) | 138 (0.8%) | | 255 (0.8%) | 138 (0.8%) | 0.00 |
| | Hispanic; n (%) | | | | | | | 699 (2.1%) | 351 (2.1%) | | 699 (2.1%) | 351 (2.1%) | 0.00 |
| Property | | | | | | | | | | | | | 0.00 |
| Manuscape for caregory based of pumps Manu | Other/Unknown; n (%) | | | | | | | 477 (1.5%) | 310 (1.9%) | | 477 (1.5%) | 310 (1.9%) | 0.00 |
| Manuscape for caregory based of pumps Manu | Missing: n (%) | | | | | | | | | | | | |
| missing missin | | | | | | | | | | | | | |
| | | - | | #VALUE! | 2,574 (18.4%) | | 0.03 | | 3,229 (19.3%) | 0.00 | #VALUE! | #VALUE! | #VALUE |
| Mathematic Mat | Northeast; n (%) | | | | | | | | | | | | -0.07 |
| Change C | South; n (%) | | , , , , , , | -0.05 | | | -0.15 | -, , | -,, | 0.13 | , , | , . , , | 0.06 |
| Conting | | | | | | | | | | | | | -0.01 |
| Inform | | N/A | N/A | #VALUE! | 179 (1.3%) | 40 (1.0%) | 0.03 | N/A | N/A | #VALUE! | 179 (1.3%) | 40 (1.0%) | 0.03 |
| March Marc | | 4 075 (4 4 50/) | 537 (43 40) | 0.00 | 4 507 (44 50/) | 275 (2.50() | 0.05 | 5 002 (24 40) | 2.452 (40.00() | 0.05 | 0.574.47.00() | 4.055 (4.5.50() | 0.04 |
| Action A | | | () | | -, (, | | | | 0,200 (20.0) | | -,, | ., (==:-,-, | 0.04 |
| Contact Cont | | | | | | | | | | | | | #VALUE |
| Select angroup (R) 127 (2.7%) 74 (1.2%) 0.02 146 (1.2%) 131 (1.0%) 0.02 0.08 | | , | | | , | , | | - ( / | , | | | | 0.01 |
| Communication and name formout formo | | | | | | | | | | | | | -0.01 |
| Chee missencification Control Corporation Septimina Septimina Control Corporation Control Corporat | | , , | ,, | | | | | | | | | | |
| Product Prod | ischemic heart disease; n (%) | | 448 (11.4%) | 0.05 | | 304 (7.8%) | | | 2,807 (16.8%) | | | | 0.05 |
| MALPH MAL | | 76 (1.0%) | 38 (1.0%) | 0.00 | 132 (0.9%) | 19 (0.5%) | 0.05 | 473 (1.5%) | 161 (1.0%) | 0.05 | 681 (1.3%) | 218 (0.9%) | 0.04 |
| History CLAS GO PT TAX (PLS) 300 (AS) 131 (BS) 0.01 23 (BS) 0.01 23 (BS) 0.00 | | | | | | | | | | | | | |
| A year ( | | | | | | | | | | | | | #VALUE! |
| Infertion (Inferton) Color ( | | , | | | | - ( , | | ,- , - , | | | | | 0.02<br>#DIV/0! |
| Infection (p (s) | , , . , | 0 (0.0%) | 0 (0.0%) | #DIV/U! | 0 (0.0%) | 0 (0.0%) | #DIV/U! | 0 (0.0%) | 0 (0.0%) | #510/0! | 0 (0.0%) | 000 (0.0%) | #DIV/U |
| Memorthagic stroken (%) | | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 000 (0.0%) | #DIV/0 |
| Chem cerebrowascular disasser, (%) 151, (159) 0,00% 0 | | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 0 (0.0%) | #DIV/0 |
| Cerebrasoulur procedure, N\$ 0,00% | TIA; n (%) | 74 (1.0%) | 29 (0.7%) | 0.03 | 110 (0.8%) | 31 (0.8%) | 0.00 | 400 (1.2%) | 174 (1.0%) | 0.02 | 584 (1.1%) | 234 (1.0%) | 0.01 |
| Next Table Next Table Next | Other cerebrovascular disease; n (%) | 135 (1.8%) | 41 (1.0%) | 0.07 | | 31 (0.8%) | 0.06 | 748 (2.3%) | 309 (1.8%) | 0.04 | 1078 (2.0%) | 381 (1.5%) | 0.04 |
| Perpland Vascular Disonse (PVD) or PVD Surgery V2 Perpland Vascula | | | | #DIV/0! | | | | | | | | | #VALUE |
| | | ** (0.1%) | 0 (0.0%) | 0.04 | ** (0.1%) | ** (0.1%) | 0.00 | 13 (0.0%) | ** (0.0%) | #DIV/0! | #VALUE! | #VALUE! | #VALUE! |
| Arial Brillation, n (S) 0,0 (M) | | | | | | | | | | | | // | |
| Other cardiac depthylthmia; n (%) | | | | | | | | | | | | | 0.04<br>#DIV/01 |
| Cardiac conduction disorder's n (%) 307 (4.1%) 174 (4.4%) 0.01 231 (2.8%) 0.15 (2.9%) 0.01 1,207 (5.5%) 932 (5.6%) 0.00 2.505 (4.6%) 122 (15.0%) 0.00 | | | | | - () | | | | - () | | | | 0.04 |
| Defect (Pr) | | | | | | | | | | | | | -0.02 |
| Courrence of Diabetic Neuropathy V2 Copy; n (%) | | | | | | | | , , | , | | | | 0.02 |
| Cocurrence of diabetic nephropathy V3 with ICD10 Copy; n (%) 235 (3.2%) 139 (3.5%) 139 (3.5%) 0.02 210 (1.5%) 5.2 (1.3%) 0.05 8.46 (2.6%) 3.89 (2.3%) 0.01 1,258 (2.3%) 460 (1.9%) 1,90 (1.9%) 1,9 | Diabetes-related complications | , -, -, | , | | , ., . , | | | ., ., ., | , , | | .,, | -, ( , | |
| Copy, n/S 235 (3.2%) 139 (3.5%) -0.02 -210 (1.5%) -52 (1.3%) -0.02 -813 (2.5%) -382 (2.3%) -0.01 -1.258 (2.3%) -573 (2.3%) -1.258 (2 | | 430 (5.8%) | 242 (6.1%) | -0.01 | 438 (3.1%) | 121 (3.1%) | 0.00 | 1,714 (5.3%) | 819 (4.9%) | 0.02 | 2582 (4.8%) | 1182 (4.8%) | 0.00 |
| Hypoglycemia v2; n(%) 125 (1.7%) 34 (0.9%) 0.07 202 (1.4%) 37 (0.9%) 0.05 84 6 (2.6%) 389 (2.3%) 0.02 1173 (2.2%) 460 (1.9%) Hypoglycemia, n (%) 432 (5.8%) 266 (6.8%) 0.04 536 (3.8%) 179 (4.6%) 0.04 2,248 (6.9%) 1,306 (7.8%) 0.03 3216 (6.0%) 171 (7.1%) Diabetic ketoacidosis; n(%) 43 (0.6%) 15 (0.4%) 0.03 76 (0.5%) 23 (0.6%) -0.01 99 (3.8%) 47 (0.3%) 0.00 212 (0.4%) 85 (0.3%) Hypertension: 1 inpatient or 2 outpatient claims 1 (1.5%) 1,912 (48.9%) 0.05 26,154 (80.2%) 12,823 (76.6%) 0.09 38,119 (70.6%) 17,160 (69.8%) Hyperipidemia v2; n (%) 3,522 (47.5%) 1,740 (44.2%) 0.07 4,709 (33.7%) 1,254 (32.1%) 0.03 17,566 (53.9%) 8,658 (51.7%) 0.04 25,797 (47.8%) 11,652 (47.4%) Edeman, n(%) 3,232 (31.4%) 1,209 (30.7%) 0.02 3,008 (21.5%) 981 (25.1%) 0.03 8,514 (20.2%) 4,346 (25.9%) 0.00 13,2 | | | | | | | | | | | | | |
| Hyperglycemia; n (%) | | | | | | | | | (=) | | | | 0.00 |
| Diabetic ketoacidosis; n (%) 43 (0.6%) 15 (0.4%) 0.03 76 (0.5%) 23 (0.6%) 0.01 93 (0.3%) 47 (0.3%) 0.00 212 (0.4%) 85 (0.3%) Hypertension: 1 inpatient or 2 outpatient claims within 365 days; n (%) 4,752 (64.1%) 2,425 (61.5%) 0.05 7,213 (51.6%) 1,912 (48.9%) 0.05 26,154 (80.2%) 12,823 (76.6%) 0.09 38,119 (70.6%) 17,160 (69.8%) Hyperlipidemia v2; n (%) 3,522 (47.5%) 1,740 (44.2%) 0.07 4,709 (33.7%) 1.254 (32.1%) 0.03 17,566 (53.9%) 8,658 (51.7%) 0.04 25,797 (47.8%) 11,652 (47.4%) 14,666 (61.1%) 1,752 (23.6%) 1,752 (2 | | | | | | | | | | | | | 0.02 |
| Hypertension: 1 inpatient or 2 outpatient claims Hypertension: 1 inpatient or 2 outpatient Hypertension: 1 inpatient or 2 outpatient Hypertension: 1 inpatient or 2 outpatient Hypertension: 1 inpatient or 2 outpatient Hypertension: 1 inpatient or 2 outpatient Hypertension: 1 inpatient Hypertension: 1 inpa | | | | | | | | | | | | | -0.04 |
| within 365 days; n (%) 4,752 (64.1%) 2,425 (61.5%) 0.05 7,213 (51.6%) 1,912 (48.9%) 0.05 26,154 (80.2%) 12,823 (76.6%) 0.09 38,119 (70.6%) 17,160 (69.8%) 17,40 (44.2%) 17,40 (44.2%) 0.07 4,709 (33.7%) 1,254 (32.1%) 0.03 17,566 (53.9%) 8,658 (51.7%) 0.04 25,797 (47.8%) 11,652 (47.4%) 1,652 (47.4% | | 43 (0.6%) | 15 (0.4%) | 0.03 | 76 (0.5%) | 23 (0.6%) | -0.01 | 93 (0.3%) | 47 (0.3%) | 0.00 | 212 (0.4%) | 85 (0.3%) | 0.02 |
| Hyperlipidemia v2; n (%) 3,522 (47.5%) 1,740 (44.2%) 0.07 4,709 (33.7%) 1,254 (32.1%) 0.03 17,566 (53.9%) 8,658 (51.7%) 0.04 25,797 (47.8%) 11,652 (47.4%) 626ma; n (%) 2,328 (31.4%) 1,209 (30.7%) 0.02 3,008 (21.5%) 981 (25.1%) 0.03 8,823 (27.0%) 3,546 (21.2%) 0.10 13852 (25.6%) 6536 (26.6%) 0.02 (3.0%) 0.03 8,823 (27.0%) 3,546 (21.2%) 0.14 12,825 (23.7%) 0.14 12,825 (23.7%) 0.14 12,825 (23. | | 4,752 (64.1%) | 2.425 (61 5%) | 0.05 | 7.213 (51.6%) | 1.917 (48 9%) | 0.05 | 26.154 (80 2%) | 12.823 (76.6%) | 0.09 | 38.119 (70 6%) | 17.160 (69 8%) | 0.02 |
| Edeman, 1(%) 2,228 (31.4%) 1,209 (30.7%) 0.02 3,008 (21.5%) 981 (25.1%) -0.09 8,516 (26.1%) 4,346 (25.9%) 0.00 13852 (25.6%) 6536 (26.6%) Renal Dysfunction (non-diabetic) v2; n (%) 1,752 (23.6%) 762 (19.3%) 0.10 2,250 (16.1%) 585 (15.0%) 0.03 8,823 (27.0%) 3,546 (21.2%) 0.14 12,825 (23.7%) 4,893 (19.9%) Occurrence of acute renal disease v2; n (%) 785 (10.0%) 321 (8.1%) 0.09 1,104 (7.9%) 319 (8.2%) -0.01 3,945 (12.1%) 1,484 (8.9%) 0.10 5834 (10.3%) 2124 (8.6%) Occurrence of chronic trenal insufficiency; n (%) 1,035 (14.0%) 403 (10.2%) 0.12 990 (7.1%) 188 (4.8%) 0.10 5,734 (17.6%) 1,950 (11.6%) 0.17 7,759 (14.4%) 2,541 (10.3%) CKD Stage 3-4; n (%) 597 (8.1%) 245 (6.2%) 0.07 515 (3.7%) 82 (2.1%) 0.10 3,238 (9.9%) 1,103 (6.6%) 0.12 4,350 (8.1%) 1,490 (8.9%) CKD Stage 3-4; n (%) 597 (8.1%) 245 (6.2%) 0.10 508 (3.6%) | | | | | | | | | , , | | | | 0.02 |
| Renal Dysfunction (non-diabetic) v2; n (%) 1,752 (23.6%) 762 (19.3%) 0.10 2,250 (16.1%) 585 (15.0%) 0.03 8,823 (27.0%) 3,546 (21.2%) 0.14 12,825 (23.7%) 4,893 (19.9%) 0.00 courrence of acute renal disease v2; n (%) 785 (10.6%) 321 (8.1%) 0.19 990 (7.1%) 188 (4.8%) 0.10 5,734 (17.6%) 1,950 (11.6%) 0.17 7,759 (14.4%) 2,541 (10.3%) 0.10 5,734 (17.6%) 1,950 (11.6%) 0.17 7,759 (14.4%) 2,541 (10.3%) 0.10 5,734 (17.6%) 1,950 (11.6%) 0.17 7,759 (14.4%) 2,541 (10.3%) 0.10 5,734 (17.6%) 1,950 (11.6%) 0.17 7,759 (14.4%) 2,541 (10.3%) 0.10 5,734 (17.6%) 1,950 (11.6%) 0.17 7,759 (14.4%) 2,541 (10.3%) 0.10 0.10 0.10 0.10 0.10 0.10 0.10 0.1 | | | | | | | | | | | | | -0.02 |
| Occurrence of chronic renal insufficiency; n (%) 1,035 (14.0%) 403 (10.2%) 0.12 990 (7.1%) 188 (8.8%) 0.10 5,734 (17.6%) 1,950 (11.6%) 0.17 7,759 (14.4%) 2,541 (10.3%) CKD Stage 3-4; n (%) 1,002 (13.5%) 387 (9.8%) 0.12 941 (6.7%) 164 (4.2%) 0.11 5,447 (16.7%) 1,859 (11.1%) 0.16 7,390 (13.7%) 2,410 (9.8%) CKD Stage 3-4; n (%) 597 (8.1%) 245 (6.2%) 0.07 515 (3.7%) 82 (2.1%) 0.10 3,238 (9.9%) 1,103 (6.6%) 0.12 4,350 (8.1%) 1,440 (6.7%) Occurrence of hypertensive nephropathy; n (%) 637 (8.6%) 240 (6.1%) 0.10 508 (3.6%) 80 (2.0%) 0.10 4,290 (13.2%) 1,327 (7.9%) 0.17 5,435 (0.1%) 1,647 (6.7%) Occurrence of miscellaneous renal insufficiency v2; n (%) 677 (9.1%) 300 (7.6%) 0.05 945 (6.8%) 248 (6.3%) 0.02 2,885 (8.8%) 1,275 (7.6%) 0.0 4,507 (8.3%) 1,823 (7.4%) User Grows and the contraction of the c | | | | 0.10 | 2,250 (16.1%) | | 0.03 | | 3,546 (21.2%) | 0.14 | 12,825 (23.7%) | 4,893 (19.9%) | 0.09 |
| Chronic kidney disease v2; n (%) 1,002 (13.5%) 387 (9.8%) 0.12 941 (6.7%) 164 (4.2%) 0.11 5,447 (16.7%) 1,859 (11.1%) 0.16 7,390 (13.7%) 2,410 (9.8%) CKD Stage 3-4; n (%) 597 (8.1%) 245 (6.2%) 0.07 515 (3.7%) 82 (2.1%) 0.10 3,238 (9.9%) 1,103 (6.6%) 0.12 4,350 (8.1%) 1,430 (5.8%) Cocurrence of hypertensive perhopathy; n (%) 637 (8.6%) 240 (6.1%) 0.10 508 (3.6%) 80 (2.0%) 0.10 4,290 (13.2%) 1,327 (7.9%) 0.17 5,335 (10.1%) 1,647 (6.7%) Cocurrence of miscellaneous renal insufficiency v2; n (%) 677 (9.1%) 300 (7.6%) 0.05 945 (6.8%) 248 (6.3%) 0.02 2,885 (8.8%) 1,275 (7.6%) 0.04 4,507 (8.3%) 1,823 (7.4%) Cher Covariates Liver disease, n (%) 0 (0.0%) **0,00% #DIV/0! 0 (0.0%) **DIV/0! 0 (0.0%) #DIV/0! 0 (0.0%) #DIV/0! 0 (0.0%) #VALUE! | | | | 0.09 | | | -0.01 | | | | | | 0.07 |
| CKD Stage 3-4; n (%) 597 (8.1%) 245 (6.2%) 0.07 515 (3.7%) 8.2 (2.1%) 0.10 3,238 (9.9%) 1,103 (6.6%) 0.12 4,350 (8.1%) 1,430 (5.8%) 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. | | | | | | | | | | | | | 0.12 |
| Occurrence of hypertensive nephropathy; n (%) 637 (8.6%) 240 (6.1%) 0.10 508 (3.6%) 80 (2.0%) 0.10 4,290 (13.2%) 1,327 (7.9%) 0.17 5,435 (10.1%) 1,647 (6.7%) Occurrence of miscellaneous renal insufficiency v2; n<br>(%) 677 (9.1%) 300 (7.6%) 0.05 945 (6.8%) 248 (6.3%) 0.02 2,885 (8.8%) 1,275 (7.6%) 0.04 4,507 (8.3%) 1,823 (7.4%) Other Covariates Liver disease; n (%) 0 (0.0%) **(0.0%) #DIV/0! 0 (0.0%) | | | | | | | | | | | | | 0.12 |
| Occurrence of miscellaneous renal insufficiency v2; n (%) 677 (9.1%) 300 (7.6%) 0.05 945 (6.8%) 248 (6.3%) 0.02 2,885 (8.8%) 1,275 (7.6%) 0.04 4,507 (8.3%) 1,823 (7.4%) Other Covariates Liver disease; n (%) 0 (0.0%) **(0.0%) #DIV/0! 0 (0.0%) #DIV/0! 0 (0.0%) #DIV/0! 0 (0.0%) #DIV/0! 0 (0.0%) #VALUE! | | (- , | | | | | | -, ( , | , , | | , , | | 0.09 |
| (%) 677 (9.1%) 300 (7.6%) 0.05 945 (6.8%) 248 (6.3%) 0.02 2,885 (8.8%) 1,275 (7.6%) 0.04 4,507 (8.3%) 1,823 (7.4%) Other Covariates Liver disease; n (%) 0 (0.0%) **(0.0%) #DIV/0! 0 (0.0%) #DI | | | 240 (6.1%) | 0.10 | 508 (3.6%) | 80 (2.0%) | 0.10 | 4,290 (13.2%) | 1,327 (7.9%) | 0.17 | 5,435 (10.1%) | 1,647 (6.7%) | 0.12 |
| Other Covariates Liver disease; n (%) 0 (0.0%) ** (0.0%) #DIV/0! 0 (0.0%) #DIV/0! 0 (0.0%) #DIV/0! 0 (0.0%) #VALUE! | | | 200 (7.5%) | 0.05 | 0.45 (5.004) | 248 (5.22() | 0.03 | 3 005 (0.004) | 1 275 (7 664) | 0.01 | 4 507 (0 201) | 1 022 /7 40/ | 0.03 |
| Liver disease; n (%) 0 (0.0%) **(0.0%) #DIV/O! 0 (0.0%) #VALUE! | 17 | 6//(9.1%) | 300 (7.6%) | 0.05 | 945 (6.8%) | 248 (b.5%) | 0.02 | 2,885 (8.8%) | 1,2/3 (/.6%) | 0.04 | 4,507 (8.3%) | 1,823 (7.4%) | 0.03 |
| | | 0 (0 0%) | ** (n n%) | #DIV/OI | 0 (0 0%) | 0 (0 0%) | #DIV/OI | 0 (0 0%) | 0 (0 0%) | #DIV/01 | 0 (0 0%) | #\/Δ F | #VALUE |
| Osteoarthritis: n (%) 2,271 (30,6%) 1,234 (31,3%) -0.02 3,146 (22.5%) 870 (71.0%) 0.04 11.878 (36.3%) 5.866 (35.0%) 0.03 17245 (31.9%) 7920 (32.2%) | Osteoarthritis; n (%) | 2,271 (30.6%) | 1,234 (31.3%) | -0.02 | 3,146 (22.5%) | 820 (21.0%) | 0.04 | 11,828 (36.3%) | 5,866 (35.0%) | 0.03 | 17245 (31.9%) | 7920 (32.2%) | -0.01 |

| Other arthritis, arthropathies and musculoskeletal | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| pain: n (%) | 6.356 (85.7%) | 3,246 (82.4%) | 0.09 | 10,836 (77.5%) | 3,049 (78.0%) | -0.01 | 24,897 (76.3%) | 12,838 (76.7%) | -0.01 | 42089 (77.9%) | 19133 (77.8%) | 0.00 |
| Dorsopathies; n (%) | 2,513 (33.9%) | 1,389 (35.3%) | -0.03 | 4,111 (29.4%) | 1,236 (31.6%) | -0.05 | 10,374 (31.8%) | 5.330 (31.8%) | 0.00 | 16998 (31.5%) | 7955 (32.3%) | -0.02 |
| Fractures; n (%) | 869 (11.7%) | 404 (10.3%) | 0.04 | 1,433 (10.3%) | 423 (10.8%) | -0.02 | 4,020 (12.3%) | 2,047 (12.2%) | 0.00 | 6322 (11.7%) | 2874 (11.7%) | 0.00 |
| Falls v2; n (%) | 692 (9.3%) | 396 (10.1%) | -0.03 | 370 (2.6%) | 139 (3.6%) | -0.02 | 1,680 (5.2%) | 735 (4.4%) | 0.04 | 2742 (5.1%) | 1270 (5.2%) | 0.00 |
| Osteoporosis: n (%) | 728 (9.8%) | 343 (8.7%) | 0.04 | 704 (5.0%) | 155 (4.0%) | 0.05 | 5.102 (15.6%) | 2,328 (13.9%) | 0.05 | 6534 (12.1%) | 2826 (11.5%) | 0.02 |
| Depression: n (%) | 1,346 (18.2%) | 655 (16.6%) | 0.04 | 1,914 (13.7%) | 561 (14.4%) | -0.02 | 5,417 (16.6%) | 2,468 (14.7%) | 0.05 | 8677 (16.1%) | 3684 (15.0%) | 0.02 |
| Anxiety; n (%) | 1,083 (14.6%) | 689 (17.5%) | -0.08 | 1,527 (10.9%) | 569 (14.6%) | -0.11 | 4,262 (13.1%) | 2,240 (13.4%) | -0.01 | 6872 (12.7%) | 3498 (14.2%) | -0.04 |
| Sleep_Disorder; n (%) | 777 (10.5%) | 252 (6.4%) | 0.15 | 1,462 (10.5%) | 352 (9.0%) | 0.05 | 2,779 (8.5%) | 938 (5.6%) | 0.11 | 5018 (9.3%) | 1542 (6.3%) | 0.11 |
| Dementia; n (%) | 706 (9.5%) | 355 (9.0%) | 0.02 | 574 (4.1%) | 167 (4.3%) | -0.01 | 5,539 (17.0%) | 2.441 (14.6%) | 0.11 | 6819 (12.6%) | 2963 (12.0%) | 0.02 |
| | | | | | | | | , , , , , , | | | | 0.02 |
| Delirium; n (%) | 281 (3.8%) | 120 (3.0%) | 0.04<br>0.04 | 387 (2.8%)<br>238 (1.7%) | 113 (2.9%) | -0.01<br>0.02 | 1,560 (4.8%)<br>1,203 (3.7%) | 754 (4.5%)<br>553 (3.3%) | 0.01<br>0.02 | 2228 (4.1%)<br>1656 (3.1%) | 987 (4.0%)<br>702 (2.9%) | 0.01 |
| Psychosis; n (%) | 215 (2.9%) | 91 (2.3%)<br>943 (23.9%) | -0.09 | | 58 (1.5%) | -0.15 | | 2.677 (16.0%) | 0.02 | | | -0.04 |
| Obesity; n (%) | 1,498 (20.2%) | ( / | -0.09 | 2,456 (17.6%) | 930 (23.8%) | | 5,202 (15.9%) | , , , , , , , | -0.05 | 9156 (17.0%) | 4550 (18.5%) | -0.04 |
| Overweight; n (%) | 244 (3.3%) | 249 (6.3%) | | 205 (1.5%) | 132 (3.4%) | -0.12 | 1,125 (3.4%) | 739 (4.4%) | | 1574 (2.9%) | 1120 (4.6%) | |
| Smoking; n (%) | 1,951 (26.3%) | 1,206 (30.6%) | -0.10 | 2,266 (16.2%) | 697 (17.8%) | -0.04 | 8,893 (27.3%) | 5,096 (30.4%) | -0.07 | 13110 (24.3%) | 6999 (28.5%) | -0.10 |
| Alcohol abuse or dependence; n (%) | 210 (2.8%) | 111 (2.8%) | 0.00 | 281 (2.0%) | 99 (2.5%) | -0.03 | 243 (0.7%) | 190 (1.1%) | -0.04 | 734 (1.4%) | 400 (1.6%) | -0.02 |
| Drug abuse or dependence; n (%) | 210 (2.8%) | 166 (4.2%) | -0.08 | 289 (2.1%) | 124 (3.2%) | -0.07 | 251 (0.8%) | 201 (1.2%) | -0.04 | 750 (1.4%) | 491 (2.0%) | -0.05 |
| COPD; n (%) | 1,066 (14.4%) | 502 (12.7%) | 0.05 | 1,214 (8.7%) | 299 (7.7%) | 0.04 | 5,389 (16.5%) | 2,517 (15.0%) | 0.04 | 7669 (14.2%) | 3318 (13.5%) | 0.02 |
| Asthma; n (%) | 710 (9.6%) | 418 (10.6%) | -0.03 | 1,139 (8.1%) | 344 (8.8%) | -0.03 | 2,725 (8.4%) | 1,431 (8.5%) | 0.00 | 4574 (8.5%) | 2193 (8.9%) | -0.01 |
| Obstructive sleep apnea; n (%) | 555 (7.5%) | 363 (9.2%) | -0.06 | 1,037 (7.4%) | 347 (8.9%) | -0.05 | 1,809 (5.5%) | 955 (5.7%) | -0.01 | 3401 (6.3%) | 1665 (6.8%) | -0.02 |
| Pneumonia; n (%) | 574 (7.7%) | 267 (6.8%) | 0.03 | 1,026 (7.3%) | 303 (7.8%) | -0.02 | 2,850 (8.7%) | 1,307 (7.8%) | 0.03 | 4450 (8.2%) | 1877 (7.6%) | 0.02 |
| Other Medications | | | | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 1,874 (25.3%) | 878 (22.3%) | 0.07 | 2,969 (21.2%) | 706 (18.1%) | 0.08 | 9,840 (30.2%) | 4,570 (27.3%) | 0.06 | 14683 (27.2%) | 6154 (25.0%) | 0.05 |
| Use of ARBs; n (%) | 899 (12.1%) | 585 (14.8%) | -0.08 | 1,741 (12.5%) | 472 (12.1%) | 0.01 | 5,634 (17.3%) | 3,141 (18.8%) | -0.04 | 8274 (15.3%) | 4198 (17.1%) | -0.05 |
| Use of Loop Diuretics - United; n (%) | 824 (11.1%) | 366 (9.3%) | 0.06 | 1,262 (9.0%) | 284 (7.3%) | 0.06 | 5,787 (17.7%) | 2,453 (14.6%) | 0.08 | 7873 (14.6%) | 3103 (12.6%) | 0.06 |
| Use of other diuretics- United; n (%) | 100 (1.3%) | 68 (1.7%) | -0.03 | 181 (1.3%) | 56 (1.4%) | -0.01 | 710 (2.2%) | 308 (1.8%) | 0.03 | 991 (1.8%) | 432 (1.8%) | 0.00 |
| Use of nitrates-United; n (%) | 171 (2.3%) | 88 (2.2%) | 0.01 | 327 (2.3%) | 62 (1.6%) | 0.05 | 1,485 (4.6%) | 622 (3.7%) | 0.05 | 1983 (3.7%) | 772 (3.1%) | 0.03 |
| Use of other hypertension drugs; n (%) | 336 (4.5%) | 147 (3.7%) | 0.04 | 577 (4.1%) | 123 (3.1%) | 0.05 | 2,141 (6.6%) | 909 (5.4%) | 0.05 | 3054 (5.7%) | 1179 (4.8%) | 0.04 |
| Use of Anti-arrhythmics; n (%) | 19 (0.3%) | ** (0.2%) | 0.02 | 59 (0.4%) | ** (0.3%) | 0.02 | 160 (0.5%) | 70 (0.4%) | 0.01 | 238 (0.4%) | #VALUE! | #VALUE! |
| Use of COPD/asthma meds- United; n (%) | 1,097 (14.8%) | 625 (15.9%) | -0.03 | 2,035 (14.6%) | 606 (15.5%) | -0.03 | 5,862 (18.0%) | 3,203 (19.1%) | -0.03 | 8994 (16.7%) | 4434 (18.0%) | -0.03 |
| Use of statins; n (%) | 2,353 (31.7%) | 1,257 (31.9%) | 0.00 | 3,676 (26.3%) | 877 (22.4%) | 0.09 | 13,267 (40.7%) | 6,840 (40.8%) | 0.00 | 19296 (35.7%) | 8974 (36.5%) | -0.02 |
| Use of other lipid-lowering drugs; n (%) | 391 (5.3%) | 177 (4.5%) | 0.04 | 851 (6.1%) | 167 (4.3%) | 0.08 | 2,075 (6.4%) | 1,096 (6.5%) | 0.00 | 3317 (6.1%) | 1440 (5.9%) | 0.01 |
| Use of antiplatelet agents; n (%) | 414 (5.6%) | 204 (5.2%) | 0.02 | 881 (6.3%) | 222 (5.7%) | 0.03 | 2,761 (8.5%) | 1,341 (8.0%) | 0.02 | 4056 (7.5%) | 1767 (7.2%) | 0.01 |
| Use of heparin and other low-molecular weight | | | | | | | | | | | | |
| heparins; n (%) | 3,868 (52.2%) | 211 (5.4%) | 1.21 | 25 (0.2%) | ** (0.1%) | 0.03 | 16,176 (49.6%) | 909 (5.4%) | 1.14 | 20069 (37.2%) | #VALUE! | #VALUE! |
| Use of NSAIDs; n (%) | 1,503 (20.3%) | 908 (23.0%) | -0.07 | 3,060 (21.9%) | 932 (23.8%) | -0.05 | 5,871 (18.0%) | 3,345 (20.0%) | -0.05 | 10434 (19.3%) | 5185 (21.1%) | -0.04 |
| Use of oral corticosteroids; n (%) | 1,930 (26.0%) | 1,065 (27.0%) | -0.02 | 3,566 (25.5%) | 1,121 (28.7%) | -0.07 | 9,326 (28.6%) | 4,915 (29.3%) | -0.02 | 14822 (27.4%) | 7101 (28.9%) | -0.03 |
| Use of bisphosphonate (United); n (%) | 283 (3.8%) | 123 (3.1%) | 0.04 | 321 (2.3%) | 57 (1.5%) | 0.06 | 1,786 (5.5%) | 824 (4.9%) | 0.03 | 2390 (4.4%) | 1004 (4.1%) | 0.01 |
| Use of opioids- United; n (%) | 4,042 (54.5%) | 1,932 (49.0%) | 0.11 | 8,355 (59.8%) | 2,318 (59.3%) | 0.01 | 15,563 (47.7%) | 7,860 (46.9%) | 0.02 | 27960 (51.8%) | 12110 (49.2%) | 0.05 |
| Use of antidepressants; n (%) | 1,919 (25.9%) | 1,055 (26.8%) | -0.02 | 3,269 (23.4%) | 937 (24.0%) | -0.01 | 9,282 (28.5%) | 4,711 (28.1%) | 0.01 | 14470 (26.8%) | 6703 (27.3%) | -0.01 |
| Use of antipsychotics; n (%) | 351 (4.7%) | 194 (4.9%) | -0.01 | 507 (3.6%) | 154 (3.9%) | -0.02 | 2,139 (6.6%) | 1,110 (6.6%) | 0.00 | 2997 (5.5%) | 1458 (5.9%) | -0.02 |
| Labs | | | | | | | | | | 21,390 | 7,848 | |
| Lab values- HbA1c (%) v3; n (%) | 651 (8.8%) | 506 (12.8%) | -0.13 | 130 (0.9%) | 46 (1.2%) | -0.03 | N/A | N/A | #VALUE! | 781 (3.7%) | 552 (7.0%) | -0.15 |
| Lab values- HbA1c (%) (within 3 months) v3; n (%) | 390 (5.3%) | 315 (8.0%) | -0.11 | 88 (0.6%) | 27 (0.7%) | -0.01 | N/A | N/A | #VALUE! | 478 (2.2%) | 342 (4.4%) | -0.12 |
| Lab values- HbA1c (%) (within 6 months) v3; n (%) | 651 (8.8%) | 506 (12.8%) | -0.13 | 130 (0.9%) | 46 (1.2%) | -0.03 | N/A | N/A | #VALUE! | 781 (3.7%) | 552 (7.0%) | -0.15 |
| Lab values- BNP; n (%) | 29 (0.4%) | 23 (0.6%) | -0.03 | ** (0.0%) | ** (0.1%) | -0.04 | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values- BNP (within 3 months); n (%) | 24 (0.3%) | 18 (0.5%) | -0.03 | ** (0.0%) | ** (0.1%) | -0.04 | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values- BNP (within 6 months); n (%) | 29 (0.4%) | 23 (0.6%) | -0.03 | ** (0.0%) | ** (0.1%) | -0.04 | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values- BUN (mg/dl); n (%) | 1,719 (23.2%) | 1.143 (29.0%) | -0.13 | 155 (1.1%) | 78 (2.0%) | -0.07 | N/A | N/A | #VALUE! | 1,874 (8.8%) | 1,221 (15.6%) | -0.21 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 1,189 (16.0%) | 815 (20.7%) | -0.12 | 106 (0.8%) | 56 (1.4%) | -0.06 | N/A | N/A | #VALUE! | 1,295 (6.1%) | 871 (11.1%) | -0.18 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 1,719 (23.2%) | 1.143 (29.0%) | -0.13 | 155 (1.1%) | 78 (2.0%) | -0.07 | N/A | N/A | #VALUE! | 1,874 (8.8%) | 1,221 (15.6%) | -0.21 |
| Lab values- Creatinine (mg/dl) v2: n (%) | 1,753 (23.6%) | 1,179 (29.9%) | -0.14 | 165 (1.2%) | 83 (2.1%) | -0.07 | N/A | N/A | #VALUE! | 1,918 (9.0%) | 1,262 (16.1%) | -0.22 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2; | -, () | -, (, | | () | () | | | .4 | | _,=== (====-, | -, (, | |
| n (%) | 1,211 (16.3%) | 846 (21.5%) | -0.13 | 114 (0.8%) | 60 (1.5%) | -0.07 | N/A | N/A | #VALUE! | 1,325 (6.2%) | 906 (11.5%) | -0.19 |
| Lab values- Creatinine (mg/dl) (within 6 months) v2; | • • | | | | . , | | • | • | | • • | | |
| n (%) | 1,753 (23.6%) | 1,179 (29.9%) | -0.14 | 165 (1.2%) | 83 (2.1%) | -0.07 | N/A | N/A | #VALUE! | 1,918 (9.0%) | 1,262 (16.1%) | -0.22 |
| Lab values- HDL level (mg/dl); n (%) | 962 (13.0%) | 693 (17.6%) | -0.13 | 96 (0.7%) | 46 (1.2%) | -0.05 | N/A | N/A | #VALUE! | 1,058 (4.9%) | 739 (9.4%) | -0.18 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 542 (7.3%) | 396 (10.1%) | -0.10 | 55 (0.4%) | 25 (0.6%) | -0.03 | N/A | N/A | #VALUE! | 597 (2.8%) | 421 (5.4%) | -0.13 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 962 (13.0%) | 693 (17.6%) | -0.13 | 96 (0.7%) | 46 (1.2%) | -0.05 | N/A | N/A | #VALUE! | 1,058 (4.9%) | 739 (9.4%) | -0.18 |
| Lab values- LDL level (mg/dl) v2; n (%) | 966 (13.0%) | 700 (17.8%) | -0.13 | 111 (0.8%) | 46 (1.2%) | -0.04 | N/A | N/A | #VALUE! | 1,077 (5.0%) | 746 (9.5%) | -0.17 |
| Lab values- LDL level (mg/dl) (within 3 months) v2; n | | | | | | | | | | | | |
| (%) | 547 (7.4%) | 399 (10.1%) | -0.10 | 66 (0.5%) | 24 (0.6%) | -0.01 | N/A | N/A | #VALUE! | 613 (2.9%) | 423 (5.4%) | -0.13 |
| Lab values-LDL level (mg/dl) (within 6 months) v2; n | | | | | | | | | | | | |
| (%) | 966 (13.0%) | 700 (17.8%) | -0.13 | 111 (0.8%) | 46 (1.2%) | -0.04 | N/A | N/A | #VALUE! | 1,077 (5.0%) | 746 (9.5%) | -0.17 |
| Lab values- NT-proBNP; n (%) | ** (0.1%) | ** (0.2%) | -0.03 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values- NT-proBNP (within 3 months); n (%) | ** (0.0%) | ** (0.2%) | -0.06 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | - |
| Lab values- NT-proBNP (within 6 months); n (%) | ** (0.1%) | ** (0.2%) | -0.03 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | - |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 972 (13.1%) | 702 (17.8%) | -0.13 | 99 (0.7%) | 46 (1.2%) | -0.05 | N/A | N/A | #VALUE! | 1,071 (5.0%) | 748 (9.5%) | -0.17 |
| Lab values-Total cholesterol (mg/dl) (within 3 | | | | | | | | | | | | |
| months) v2; n (%) | 549 (7.4%) | 401 (10.2%) | -0.10 | 55 (0.4%) | 25 (0.6%) | -0.03 | N/A | N/A | #VALUE! | 604 (2.8%) | 426 (5.4%) | -0.13 |
| Lab values-Total cholesterol (mg/dl) (within 6 | | | | | | | | | | | | |
| months) v2; n (%) | 972 (13.1%) | 702 (17.8%) | -0.13 | 99 (0.7%) | 46 (1.2%) | -0.05 | N/A | N/A | #VALUE! | 1,071 (5.0%) | 748 (9.5%) | -0.17 |
| Lab values-Triglyceride level (mg/dl); n (%) | 964 (13.0%) | 696 (17.7%) | -0.13 | 100 (0.7%) | 46 (1.2%) | -0.05 | N/A | N/A | #VALUE! | 1,064 (5.0%) | 742 (9.5%) | -0.17 |
| Lab values-Triglyceride level (mg/dl) (within 3 | | | | | | | | | | | | |
| months); n (%) | 544 (7.3%) | 397 (10.1%) | -0.10 | 57 (0.4%) | 24 (0.6%) | -0.03 | N/A | N/A | #VALUE! | 601 (2.8%) | 421 (5.4%) | -0.13 |

| Laborations Tainle consider level (mon/dl) (containing | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Lab values-Triglyceride level (mg/dl) (within 6 months); n (%) | 964 (13.0%) | 696 (17.7%) | -0.13 | 100 (0.7%) | 46 (1.2%) | -0.05 | N/A | N/A | #VALUE! | 1,064 (5.0%) | 742 (9.5%) | -0.17 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | 304 (13.070) | 030 (17.770) | 0.15 | 100 (0.770) | 40 (2.270) | 0.05 | .,,,, | .,,,, | ###E0E. | 2,004 (3.070) | 742 (3.370) | 0.17 |
| included) v4 | 650 | 505 | | 112 | 45 | | N/A | N/A | | 762 | 550 | |
| mean (sd) | 6.79 (1.57) | 6.72 (1.73) | 0.04 | 7.26 (1.63) | 7.18 (1.48) | 0.05 | N/A | N/A | #VALUE! | 6.86 (1.58) | 6.76 (1.71) | 0.06 |
| Missing; n (%) | 6,763 (91.2%) | 3,435 (87.2%) | 0.13 | 13,865 (99.2%) | 3,863 (98.8%) | 0.04 | N/A | N/A | #VALUE! | 20,628 (96.4%) | 7,298 (93.0%) | 0.15 |
| Lab result number- BNP mean v2 | 29 | 23 | | 4 | 5 | | N/A | N/A | | 33 | 28 | |
| mean (sd) | 74.87 (72.49) | 96.03 (235.14) | -0.12 | 19.25 (8.96) | 161.20 (119.25) | -1.68 | N/A | N/A | #VALUE! | 68.13 (70.09) | 107.67 (225.68) | -0.24 |
| Missing; n (%) | 7,384 (99.6%) | 3,917 (99.4%) | 0.03 | 13,973 (100.0%) | 3,903 (99.9%) | 0.04 | N/A | N/A | #VALUE! | 21,357 (99.8%) | 7,820 (99.6%) | 0.04 |
| Lab result number- BUN (mg/dl) mean v2 | 1,719<br>18.02 (7.51) | 1,143<br>17.09 (6.74) | 0.13 | 1.436.31 (17.669.46) | 78<br>17.18 (6.52) | 0.11 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 1,874<br>135.33 (5069.29) | 1,221 | 0.03 |
| mean (sd)Missing; n (%) | 18.02 (7.51)<br>5,694 (76.8%) | 2,797 (71.0%) | 0.13 | 1,436.31 (17,669.46) | 3,830 (98.0%) | 0.11 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 19,516 (91.2%) | 17.10 (6.73)<br>6,627 (84.4%) | 0.03 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 | 3,034 (70.6%) | 2,757 (71.0%) | 0.13 | 13,022 (30.370) | 3,030 (50.0%) | 0.07 | N/A | N/A | #VALUE: | 15,310 (51.276) | 0,027 (84.476) | 0.21 |
| to 15 included) v3 | 1.741 | 1.168 | | 160 | 81 | | N/A | N/A | | 1,901 | 1.249 | |
| mean (sd) | 1.00 (0.34) | 0.96 (0.29) | 0.13 | 0.98 (0.31) | 0.97 (0.29) | 0.03 | N/A | N/A | #VALUE! | 1.00 (0.34) | 0.96 (0.29) | 0.13 |
| Missing; n (%) | 5,672 (76.5%) | 2,772 (70.4%) | 0.14 | 13,817 (98.9%) | 3,827 (97.9%) | 0.08 | N/A | N/A | #VALUE! | 19,489 (91.1%) | 6,599 (84.1%) | 0.21 |
| Lab result number- HDL level (mg/dl) mean (only | | | | | | | | | | | | |
| =<5000 included) v2 | 962 | 693 | | 95 | 46 | | N/A | N/A | | 1,057 | 739 | |
| mean (sd) | 53.64 (17.08) | 53.25 (17.87) | 0.02 | 46.65 (12.95) | 48.63 (14.03) | -0.15 | N/A | N/A | #VALUE! | 53.01 (16.76) | 52.96 (17.67) | 0.00 |
| Missing; n (%) | 6,451 (87.0%) | 3,247 (82.4%) | 0.13 | 13,882 (99.3%) | 3,862 (98.8%) | 0.05 | N/A | N/A | #VALUE! | 20,333 (95.1%) | 7,109 (90.6%) | 0.18 |
| Lab result number- LDL level (mg/dl) mean (only<br>=<5000 included) v2 | 942 | 692 | | 97 | 44 | | N/A | N/A | | 1,039 | 736 | |
| =<5000 included) v2<br>mean (sd) | 102.51 (34.84) | 101.93 (36.29) | 0.02 | 96.33 (37.96) | 92.61 (31.60) | 0.11 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 101.93 (35.16) | 101.37 (36.06) | 0.02 |
| Missing; n (%) | 6,471 (87.3%) | 3,248 (82.4%) | 0.02 | 13,880 (99.3%) | 3,864 (98.9%) | 0.04 | N/A | N/A | #VALUE! | 20.351 (95.1%) | 7,112 (90.6%) | 0.02 |
| Lab result number-Total cholesterol (mg/dl) mean | 0,471 (07.570) | 3,240 (02.470) | 0.14 | 13,000 (33.370) | 3,004 (30.370) | 0.04 | 14/5 | 11/1 | #VALUE: | 20,331 (33.170) | 7,112 (50.070) | 0.10 |
| (only =<5000 included) v2 | 971 | 702 | | 98 | 46 | | N/A | N/A | | 1,069 | 748 | |
| mean (sd) | 184.17 (40.78) | 183.48 (41.96) | 0.02 | 176.51 (45.32) | 181.96 (42.96) | -0.12 | N/A | N/A | #VALUE! | 183.47 (41.23) | 183.39 (42.05) | 0.00 |
| Missing; n (%) | 6,442 (86.9%) | 3,238 (82.2%) | 0.13 | 13,879 (99.3%) | 3,862 (98.8%) | 0.05 | N/A | N/A | #VALUE! | 20,321 (95.0%) | 7,100 (90.5%) | 0.17 |
| Lab result number-Triglyceride level (mg/dl) mean | | | | | | | | | | | | |
| (only =<5000 included) v2 | 964 | 696 | | 99 | 46 | | N/A | N/A | | 1,063 | 742 | |
| mean (sd) | 136.73 (77.90) | 140.13 (102.33) | -0.04 | 159.89 (94.35) | 179.18 (110.20) | -0.19 | N/A | N/A | #VALUE! | 138.89 (79.60) | 142.55 (102.90) | -0.04 |
| Missing; n (%) | 6,449 (87.0%) | 3,244 (82.3%) | 0.13 | 13,878 (99.3%) | 3,862 (98.8%) | 0.05 | N/A | N/A | #VALUE! | 20,327 (95.0%) | 7,106 (90.5%) | 0.17 |
| Lab result number- Hemoglobin mean (only >0 | 4.202 | 952 | | 405 | | | | **** | | 4 400 | 4.000 | |
| included)<br>mean (sd) | 1,393<br>13.28 (1.90) | 13.37 (1.86) | -0.05 | 106<br>1.408.80 (14.373.80) | 71<br>12.85 (2.78) | 0.14 | N/A<br>N/A | N/A<br>N/A | #VALUE! | 1,499<br>111.96 (3808.03) | 1,023<br>13.33 (1.94) | 0.04 |
| Missing; n (%) | 6,020 (81.2%) | 2,988 (75.8%) | 0.03 | 13,871 (99.2%) | 3,837 (98.2%) | 0.09 | N/A | N/A | #VALUE! | 19,891 (93.0%) | 6,825 (87.0%) | 0.20 |
| Lab result number- Serum sodium mean (only > 90 | 0,020 (01.270) | 2,500 (75.070) | 0.13 | 13,071 (33.270) | 3,037 (30.270) | 0.05 | 14/5 | 11/1 | #VALUE: | 13,031 (33.070) | 0,023 (07.070) | 0.20 |
| and < 190 included) | 1,691 | 1,116 | | 143 | 77 | | N/A | N/A | | 1,834 | 1,193 | |
| mean (sd) | 139.91 (2.74) | 140.29 (2.71) | -0.14 | 139.13 (2.43) | 139.00 (3.00) | 0.05 | N/A | N/A | #VALUE! | 139.85 (2.72) | 140.21 (2.73) | -0.13 |
| Missing; n (%) | 5,722 (77.2%) | 2,824 (71.7%) | 0.13 | 13,834 (99.0%) | 3,831 (98.0%) | 0.08 | N/A | N/A | #VALUE! | 19,556 (91.4%) | 6,655 (84.8%) | 0.20 |
| Lab result number- Albumin mean (only >0 and <=10 | | | | | | | | | | | | |
| included) | 1,536 | 1,006 | | 116 | 66 | | N/A | N/A | | 1,652 | 1,072 | |
| mean (sd) | 4.08 (0.39) | 4.12 (0.40) | -0.10 | 3.95 (0.78) | 3.98 (0.64) | -0.04 | N/A | N/A | #VALUE! | 4.07 (0.43) | 4.11 (0.42) | -0.09 |
| Missing; n (%) | 5,877 (79.3%) | 2,934 (74.5%) | 0.11 | 13,861 (99.2%) | 3,842 (98.3%) | 0.08 | N/A | N/A | #VALUE! | 19,738 (92.3%) | 6,776 (86.3%) | 0.20 |
| Lab result number- Glucose (fasting or random) mean<br>(only 10-1000 included) | 1,667 | 1,111 | | 131 | 78 | | N/A | N/A | | 1,798 | 1,189 | |
| mean (sd) | 111.25 (46.51) | 113.95 (43.40) | -0.06 | 136.41 (56.48) | 147.32 (75.50) | -0.16 | N/A | N/A | #VALUE! | 113.08 (47.32) | 116.14 (46.18) | -0.07 |
| Missing; n (%) | 5,746 (77.5%) | 2,829 (71.8%) | 0.13 | 13,846 (99.1%) | 3,830 (98.0%) | 0.09 | N/A | N/A | #VALUE! | 19,592 (91.6%) | 6,659 (84.8%) | 0.21 |
| Lab result number- Potassium mean (only 1-7 | ., ., ., | , | | .,, | .,, | | • | | | .,, | ., | - |
| included) | 1,721 | 1,153 | | 155 | 75 | | N/A | N/A | | 1,876 | 1,228 | |
| mean (sd) | 4.31 (0.43) | 4.35 (0.44) | -0.09 | 4.23 (0.41) | 4.33 (0.40) | -0.25 | N/A | N/A | #VALUE! | 4.30 (0.43) | 4.35 (0.44) | -0.11 |
| Missing; n (%) | 5,692 (76.8%) | 2,787 (70.7%) | 0.14 | 13,822 (98.9%) | 3,833 (98.1%) | 0.07 | N/A | N/A | #VALUE! | 19,514 (91.2%) | 6,620 (84.4%) | 0.21 |
| Comorbidity Scores | | | | | | | | | | | | |
| Combined comorbidity score, 365 days Copy | | / / | | | | | | | | / | | |
| mean (sd) | 1.91 (2.34) | 2.06 (2.35) | -0.06 | 1.39 (2.10) | 1.58 (2.23) | -0.09 | 2.20 (2.56) | 2.04 (2.57) | 0.06 | 1.95 (2.42) | 1.97 (2.48) | -0.01<br>0.07 |
| Non-Frailty; n (%)<br>Frailty Score (mean): Empirical Version 365 days, v2 | 3,500 (47.2%) | 1,973 (50.1%) | -0.06 | 5,638 (40.3%) | 1,646 (42.1%) | -0.04 | 854 (2.6%) | 263 (1.6%) | 0.07 | 9,992 (18.5%) | 3,882 (15.8%) | 0.07 |
| mean (sd) | 0.19 (0.07) | 0.18 (0.07) | 0.14 | 0.17 (0.06) | 0.17 (0.06) | 0.00 | 0.11 (0.08) | 0.09 (0.08) | 0.25 | 0.14 (0.07) | 0.12 (0.08) | 0.27 |
| Healthcare Utilization | 0.13 (0.07) | 0.10 (0.07) | 0.14 | 0.17 (0.00) | 0.17 (0.00) | 0.00 | 0.11 (0.00) | 0.05 (0.08) | 0.23 | 0.14 (0.07) | 0.12 (0.00) | 0.27 |
| Any hospitalization; n (%) | 5,944 (80.2%) | 2,390 (60.7%) | 0.44 | 13,968 (99.9%) | 3,908 (100.0%) | -0.04 | 24,871 (76.2%) | 9,527 (56.9%) | 0.42 | 44,783 (82.9%) | 15,825 (64.3%) | 0.43 |
| Any hospitalization within prior 30 days; n (%) | 5,565 (75.1%) | 2,178 (55.3%) | 0.42 | 13,769 (98.5%) | 3,866 (98.9%) | -0.04 | 23,580 (72.3%) | 8,440 (50.4%) | 0.46 | 42914 (79.5%) | 14484 (58.9%) | 0.46 |
| Any hospitalization during prior 31-180 days; n (%) | 1,176 (15.9%) | 491 (12.5%) | 0.10 | 1,855 (13.3%) | 517 (13.2%) | 0.00 | 5,754 (17.6%) | 2,725 (16.3%) | 0.03 | 8785 (16.3%) | 3733 (15.2%) | 0.03 |
| Internal medicine/family medicine visits; n (%) | 6,578 (88.7%) | 3,420 (86.8%) | 0.06 | 10,624 (76.0%) | 3,112 (79.6%) | -0.09 | 30,337 (93.0%) | 15,307 (91.4%) | 0.06 | 47539 (88.0%) | 21839 (88.8%) | -0.02 |
| Internal medicine/family medicine visits (30 days | | | | | | | | | | | | |
| prior) v2; n (%) | 5,853 (79.0%) | 2,941 (74.6%) | 0.10 | 7,601 (54.4%) | 2,169 (55.5%) | -0.02 | 27,977 (85.8%) | 13,422 (80.1%) | 0.15 | 41431 (76.7%) | 18532 (75.3%) | 0.03 |
| Internal medicine/family medicine visits (31 to 180 | E 044 (C0 001) | 2 (27 (66 70/) | 0.03 | 0.752/62.69() | 2 400 (62 0%) | 0.03 | 22 700 (72 00/) | 12 120 (72 50) | 0.01 | 27504/50 52/1 | 47365 (70.30) | 0.04 |
| days prior) v2; n (%) | 5,044 (68.0%)<br>3,053 (41.2%) | 2,627 (66.7%)<br>1,683 (42.7%) | 0.03<br>-0.03 | 8,752 (62.6%)<br>3,042 (21.8%) | 2,499 (63.9%)<br>883 (22.6%) | -0.03<br>-0.02 | 23,788 (72.9%)<br>15,604 (47.8%) | 12,139 (72.5%)<br>7,724 (46.1%) | 0.01<br>0.03 | 37584 (69.6%)<br>21699 (40.2%) | 17265 (70.2%)<br>10290 (41.8%) | -0.01<br>-0.03 |
| Cardiologist visit; n (%) Number of Cardiologist visits (30 days prior); n (%) | 2,224 (30.0%) | 1,248 (31.7%) | -0.03 | 1,698 (12.1%) | 502 (12.8%) | -0.02 | 11,149 (34.2%) | 5,410 (32.3%) | 0.03 | 15071 (27.9%) | 7160 (29.1%) | -0.03 |
| Number of Cardiologist visits (30 days prior); it (%) Number of Cardiologist visits (31 to 180 days prior); | 2,224 (30.0%) | 1,240 (31.770) | -0.04 | 1,050 (12.1%) | 302 (12.0%) | -0.02 | 11,145 (34.2%) | 3,410 (32.3/6) | 0.04 | 130/1(2/.3%) | /100 (25.1%) | -0.03 |
| n (%) | 1,404 (18.9%) | 730 (18.5%) | 0.01 | 1,797 (12.9%) | 489 (12.5%) | 0.01 | 8,231 (25.2%) | 4,091 (24.4%) | 0.02 | 11432 (21.2%) | 5310 (21.6%) | -0.01 |
| Electrocardiogram v2; n (%) | 4,088 (55.1%) | 2,158 (54.8%) | 0.01 | 5,377 (38.5%) | 1,410 (36.1%) | 0.05 | 19,760 (60.6%) | 10,095 (60.3%) | 0.01 | 29225 (54.1%) | 13663 (55.5%) | -0.03 |
| Use of glucose test strips; n (%) | 126 (1.7%) | 54 (1.4%) | 0.02 | 168 (1.2%) | 40 (1.0%) | 0.02 | 535 (1.6%) | 273 (1.6%) | 0.00 | 829 (1.5%) | 367 (1.5%) | 0.00 |
| Dialysis; n (%) | 12 (0.2%) | 0 (0.0%) | 0.06 | 34 (0.2%) | ** (0.2%) | 0.00 | 50 (0.2%) | ** (0.0%) | 0.06 | 96 (0.2%) | #VALUE! | #VALUE! |
| number of different/distinct medication | | | | | | | | | | | | |
| prescriptions | | | | | | | | | | | | |
| mean (sd) | 9.27 (5.24) | 8.77 (5.41) | 0.09 | 9.24 (5.40) | 8.81 (5.72) | 0.08 | 10.13 (5.09) | 9.52 (5.21) | 0.12 | 9.78 (5.19) | 9.29 (5.33) | 0.00 |
| Number of Hospitalizations | 1.04(0.77) | 0.70 (0.00) | 0.33 | 1 20 (0 65) | 1 30 (0 65) | -0.02 | 1.07.(0.00) | 0.80 (0.04) | 0.30 | 1 12 (0.02) | 0.88/0.35 | 0.00 |
| mean (sd) | 1.04 (0.77) | 0.78 (0.80) | 0.33 | 1.29 (0.66) | 1.30 (0.66) | -0.02 | 1.07 (0.89) | 0.80 (0.91) | 0.30 | 1.12 (0.82) | 0.88 (0.86) | 0.00 |

| Norther of heavital days | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number of hospital days<br>mean (sd) | 5.40 (6.24) | 3.51 (5.41) | 0.32 | 7.63 (8.24) | 6.53 (7.92) | 0.14 | 6.13 (7.52) | 3.90 (6.63) | 0.31 | 6.42 (7.55) | 4.26 (6.68) | 0.00 |
| Number of Emergency Department (ED) visits v3 | 3.40 (0.24) | 3.31(3.41) | 0.52 | 7.05 (0.24) | 0.55 (7.52) | 0.14 | 0.13 (7.32) | 3.50 (0.05) | 0.51 | 0.42 (7.55) | 4.20 (0.00) | 0.00 |
| mean (sd) | 1.85 (2.17) | 2.24 (2.08) | -0.18 | 1.92 (4.54) | 2.74 (6.70) | -0.14 | 2.04 (2.04) | 2.42 (2.17) | -0.18 | 1.98 (2.91) | 2.44 (3.32) | 0.00 |
| Number of Office visits | | | | | | | | | | | | |
| mean (sd) | 5.48 (4.83) | 5.64 (4.79) | -0.03 | 5.53 (5.19) | 5.62 (5.12) | -0.02 | 12.84 (14.53) | 13.84 (15.97) | -0.07 | 9.94 (11.73) | 11.22 (13.47) | 0.00 |
| Number of internal medicine/family medicine visits | | | | | | | | | | | | |
| mean (sd) | 10.84 (15.87) | 9.07 (12.25) | 0.12 | 6.06 (11.94) | 5.97 (10.44) | 0.01 | 11.66 (12.16) | 10.09 (12.41) | 0.13 | 10.10 (12.68) | 9.27 (12.09) | 0.00 |
| Number of Cardiologist visits | | | | / | / ) | | | | | | | |
| mean (sd) | 1.39 (3.30) | 1.36 (3.07) | 0.01 | 0.61 (2.29) | 0.62 (2.33) | 0.00 | 1.79 (3.80) | 1.63 (3.45) | 0.04 | 1.43 (3.40) | 1.43 (3.24) | 0.00 |
| Number electrocardiograms received v2<br>mean (sd) | 1.16 (1.68) | 1.22 (1.70) | -0.04 | 0.65 (1.11) | 0.65 (1.16) | 0.00 | 1.32 (1.64) | 1.36 (1.67) | -0.02 | 1.12 (1.53) | 1.22 (1.60) | 0.00 |
| Number of HbA1c tests ordered | 1.10 (1.00) | 1.22 (1.70) | -0.04 | 0.03 (1.11) | 0.03 (1.10) | 0.00 | 1.32 (1.04) | 1.50 (1.07) | -0.02 | 1.12 (1.55) | 1.22 (1.00) | 0.00 |
| mean (sd) | 0.31 (0.64) | 0.36 (0.68) | -0.08 | 0.20 (0.53) | 0.22 (0.54) | -0.04 | 0.37 (0.70) | 0.39 (0.71) | -0.03 | 0.32 (0.65) | 0.36 (0.68) | 0.00 |
| Number of glucose tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.27 (2.73) | 0.37 (4.22) | -0.03 | 0.16 (0.98) | 0.16 (0.96) | 0.00 | 0.18 (0.72) | 0.18 (0.72) | 0.00 | 0.19 (1.26) | 0.21 (1.83) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.49 (0.77) | 0.48 (0.78) | 0.01 | 0.34 (0.75) | 0.36 (0.85) | -0.02 | 0.52 (0.72) | 0.54 (0.73) | -0.03 | 0.47 (0.73) | 0.50 (0.76) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | | | | | | | | | | | | |
| digit level Copy<br>mean (sd) | 6.61 (10.06) | 10.92 (12.43) | -0.38 | 5.13 (9.89) | 8.02 (11.79) | -0.27 | 9.35 (12.17) | 11.79 (13.06) | -0.19 | 7.88 (11.34) | 11.05 (12.77) | 0.00 |
| For PS | 0.01 (10.00) | 10.52 (12.43) | -0.36 | 3.13 (3.03) | 8.02 (11.79) | -0.27 | 5.55 (12.17) | 11.79 (13.00) | -0.15 | 7.00 (11.34) | 11.03 (12.77) | 0.00 |
| Hemorrhagic stroke+Other cerebrovascular | | | | | | | | | | | | |
| disease+Cerebrovascular procedure (for PS); n (%) | 135 (1.8%) | 41 (1.0%) | 0.07 | 199 (1.4%) | 31 (0.8%) | 0.06 | 748 (2.3%) | 309 (1.8%) | 0.04 | 1082 (2.0%) | 381 (1.5%) | 0.04 |
| immobilization; n (%) | 766 (10.3%) | 378 (9.6%) | #DIV/0! | 1,385 (9.9%) | 417 (10.7%) | #DIV/0! | 2,774 (8.5%) | 1,488 (8.9%) | #DIV/0! | 1,385 (9.9%) | 417 (10.7%) | -0.03 |
| Occurrence of creatinine tests ordered (for PS); n (%) | 592 (8.0%) | 317 (8.0%) | 0.00 | 926 (6.6%) | 247 (6.3%) | 0.01 | 3,559 (10.9%) | 1,774 (10.6%) | 0.01 | 5077 (9.4%) | 2338 (9.5%) | 0.00 |
| Occurrence of BUN tests ordered (for PS); n (%) | 350 (4.7%) | 160 (4.1%) | 0.03 | 597 (4.3%) | 140 (3.6%) | 0.04 | 2,099 (6.4%) | 998 (6.0%) | 0.02 | 3046 (5.6%) | 1298 (5.3%) | 0.01 |
| Occurrence of chronic renal insufficiency w/o CKD | 593 (8.0%) | 179 (4.5%) | 0.14 | 599 (4.3%) | 109 (2.8%) | 0.08 | 3,259 (10.0%) | 967 (5.8%) | 0.16 | 4451 (8.2%) | 1255 (5.1%) | 0.12 |
| (for PS) v2; n (%)<br>Chronic kidney disease Stage 1-2 (for PS); n (%) | 154 (2.1%) | 66 (1.7%) | 0.14 | 124 (0.9%) | 29 (0.7%) | 0.08 | 566 (1.7%) | 262 (1.6%) | 0.10 | 844 (1.6%) | 357 (1.5%) | 0.12 |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 597 (8.1%) | 245 (6.2%) | 0.07 | 515 (3.7%) | 82 (2.1%) | 0.10 | 3,238 (9.9%) | 1,103 (6.6%) | 0.12 | 4350 (8.1%) | 1430 (5.8%) | 0.09 |
| Acute kidney injury; n (%) | 818 (11.0%) | 329 (8.4%) | #DIV/0! | 1,167 (8.3%) | 331 (8.5%) | #DIV/0! | 4,121 (12.6%) | 1,533 (9.2%) | #DIV/0! | 1,167 (8.3%) | 331 (8.5%) | -0.01 |
| Bladder stones+Kidney stones (for PS); n (%) | 243 (3.3%) | 140 (3.6%) | -0.02 | 397 (2.8%) | 120 (3.1%) | -0.02 | 1,013 (3.1%) | 500 (3.0%) | 0.01 | 1653 (3.1%) | 760 (3.1%) | 0.00 |
| Alcohol abuse or dependence+Drug abuse or | | | | | | | | | | | | |
| dependence (for PS); n (%) | 394 (5.3%) | 260 (6.6%) | -0.05 | 528 (3.8%) | 206 (5.3%) | -0.07 | 471 (1.4%) | 376 (2.2%) | -0.06 | 1393 (2.6%) | 842 (3.4%) | -0.05 |
| Other atherosclerosis+Cardiac conduction | 4 205 (40 70/) | 720 (40 70) | 0.00 | 2 457 (47 70/) | 504 (47 50/) | | 5 740 (20 50) | 2 222 (40 20() | | 40573 (40.50() | 45.44.(40.00() | 0.03 |
| disorders+Other CVD (for PS) v2 Copy; n (%) | 1,386 (18.7%) | 738 (18.7%) | 0.00 | 2,467 (17.7%) | 684 (17.5%) | 0.01 | 6,719 (20.6%) | 3,222 (19.2%) | 0.04 | 10572 (19.6%) | 4644 (18.9%) | 0.02 |
| Previous cardiac procedure (CABG or PTCA or Stent) +<br>History of CABG or PTCA (for PS) v3; n (%) | 312 (4.2%) | 154 (3.9%) | 0.02 | 303 (2.2%) | 69 (1.8%) | 0.03 | 2,603 (8.0%) | 1,073 (6.4%) | 0.06 | 3218 (6.0%) | 1296 (5.3%) | 0.03 |
| Diabetes with complication; n (%) | 812 (11.0%) | 438 (11.1%) | #DIV/0! | 1,013 (7.2%) | 311 (8.0%) | #DIV/0! | 3,661 (11.2%) | 1,716 (10.2%) | #DIV/0! | 1,013 (7.2%) | 311 (8.0%) | -0.03 |
| Delirium + Psychosis (for PS); n (%) | 433 (5.8%) | 186 (4.7%) | 0.05 | 551 (3.9%) | 154 (3.9%) | 0.00 | 2,441 (7.5%) | 1,151 (6.9%) | 0.02 | 3425 (6.3%) | 1491 (6.1%) | 0.01 |
| Any use of Meglitinides (for PS); n (%) | 13 (0.2%) | ** (0.3%) | -0.02 | 30 (0.2%) | ** (0.1%) | 0.03 | 108 (0.3%) | 48 (0.3%) | 0.00 | 151 (0.3%) | #VALUE! | #VALUE! |
| Any use of AGIs (for PS); n (%) | ** (0.1%) | ** (0.1%) | 0.00 | ** (0.0%) | ** (0.1%) | -0.04 | 32 (0.1%) | ** (0.0%) | 0.04 | #VALUE! | #VALUE! | #VALUE! |
| CKD stage 3-6 + dialysis (for PS); n (%) | 609 (8.2%) | 247 (6.3%) | 0.07 | 546 (3.9%) | 89 (2.3%) | 0.09 | 3,272 (10.0%) | 1,110 (6.6%) | 0.12 | 4427 (8.2%) | 1446 (5.9%) | 0.09 |
| Use of thiazide- United; n (%) | 671 (9.1%) | 365 (9.3%) | -0.01 | 1,101 (7.9%) | 246 (6.3%) | 0.06 | 3,945 (12.1%) | 1,768 (10.6%) | 0.05 | 5717 (10.6%) | 2379 (9.7%) | 0.03 |
| Use of beta blockers; n (%) | 1,762 (23.8%) | 811 (20.6%) | 0.08 | 3,041 (21.8%) | 707 (18.1%) | 0.09 | 11,260 (34.5%) | 5,254 (31.4%) | 0.07 | 16063 (29.7%) | 6772 (27.5%) | 0.05 |
| Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) | 1,415 (19.1%)<br>1,120 (15.1%) | 722 (18.3%)<br>574 (14.6%) | 0.02<br>0.01 | 2,267 (16.2%)<br>1,771 (12.7%) | 545 (13.9%)<br>458 (11.7%) | 0.06<br>0.03 | 8,772 (26.9%)<br>5,547 (17.0%) | 4,060 (24.2%)<br>2,680 (16.0%) | 0.06<br>0.03 | 12454 (23.1%)<br>8438 (15.6%) | 5327 (21.7%)<br>3712 (15.1%) | 0.03<br>0.01 |
| DM Medications - Insulin Copy; n (%) | 441 (5.9%) | 217 (5.5%) | 0.01 | 779 (5.6%) | 196 (5.0%) | 0.03 | 1,692 (5.2%) | 734 (4.4%) | 0.03 | 2912 (5.4%) | 1147 (4.7%) | 0.01 |
| Use of Low Intensity Statins; n (%) | 1,617 (21.8%) | 763 (19.4%) | 0.02 | 2,357 (16.9%) | 521 (13.3%) | 0.10 | 9,199 (28.2%) | 4,445 (26.5%) | 0.04 | 13173 (24.4%) | 5729 (23.3%) | 0.03 |
| Use of High Intensity Statins; n (%) | 769 (10.4%) | 503 (12.8%) | -0.08 | 1,328 (9.5%) | 365 (9.3%) | 0.01 | 4,205 (12.9%) | 2,477 (14.8%) | -0.06 | 6302 (11.7%) | 3345 (13.6%) | -0.06 |
| Malignant hypertension; n (%) | 771 (10.4%) | 206 (5.2%) | 0.19 | 6,113 (43.7%) | 1,154 (29.5%) | 0.30 | 13,959 (42.8%) | 4,636 (27.7%) | 0.32 | 20843 (38.6%) | 5996 (24.4%) | 0.31 |
| Cardiovascular stress test; n (%) | 29 (0.4%) | ** (0.2%) | 0.04 | 51 (0.4%) | 15 (0.4%) | 0.00 | 174 (0.5%) | 81 (0.5%) | 0.00 | 254 (0.5%) | #VALUE! | #VALUE! |
| Echocardiogram; n (%) | 1,217 (16.4%) | 712 (18.1%) | -0.05 | 2,591 (18.5%) | 783 (20.0%) | -0.04 | 6,200 (19.0%) | 3,177 (19.0%) | 0.00 | 10008 (18.5%) | 4672 (19.0%) | -0.01 |
| Number of BNP tests | | | | | | | | | | | | |
| mean (sd) | 0.06 (0.28) | 0.11 (0.38) | -0.15 | 0.03 (0.20) | 0.05 (0.25) | -0.09 | 0.09 (0.33) | 0.12 (0.37) | -0.09 | 0.07 (0.29) | 0.11 (0.36) | -0.12 |
| Number of Cardiac biomarkers tests (tropnin, CK-MBs, M | roglobin CDK) | | | | | | | | | | | |
| mean (sd) | 0.32 (1.21) | 0.40 (1.19) | -0.07 | 0.22 (0.95) | 0.28 (1.06) | -0.06 | 0.22 (0.55) | 0.27 (0.62) | -0.09 | 0.23 (0.79) | 0.29 (0.82) | 0.00 |
| | | *****(====) | | | () | | 0.22 (0.00) | () | | | 0.20 (0.02) | |
| Number of Ambulatory Blood pressure monitoring tests | | | | | | | | | | | | |
| mean (sd) | 0.00 (0.04) | 0.00 (0.00) | 0.00 | 0.00 (0.04) | 0.00 (0.04) | 0.00 | 0.00 (0.03) | 0.00 (0.04) | 0.00 | 0.00 (0.03) | 0.00 (0.04) | 0.00 |
| N. C. L. C. | | | | | | | | | | | | |
| N of days on antihypertensive medications during baselin<br>mean (sd) | e 78.67 (79.06) | 79.51 (80.27) | -0.01 | 67.34 (78.33) | 58.24 (75.77) | 0.12 | 0<br>107.82 (76.83) | 0<br>104.35 (78.11) | 0.04 | 93.34 (77.53) | 93.04 (78.09) | 0.00 |
| N of days in database anytime prior | 78.07 (79.00) | 79.51 (80.27) | -0.01 | 07.34 (78.33) | 38.24 (/3.//) | 0.12 | 107.82 (76.83) | 104.35 (78.11) | 0.04 | 93.34 (77.53) | 93.04 (78.09) | 0.00 |
| mean (sd) | 1,629.27 (1,170.61) | 1,681.72 (1,331.40) | -0.04 | 1,747.51 (1,223.63) | 2,037.38 (1,445.60) | -0.22 | 619.84 (384.70) | 645.09 (368.82) | -0.07 | 1050.22 (815.43) | 1032.36 (841.75) | 0.00 |
| () | ,,, ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | ., (1,001.40) | 0.0- | , (2,225.05) | ., (2,3.00) | 0.22 | | (300.02) | 0.07 | | | 0.00 |
| Mean Copay for per prescription cost (charges in U.S. \$) ( | 180-1 day prior) | | | | | | 0 | 0 | | | | |
| mean (sd) | 24.96 (37.89) | 23.57 (44.39) | 0.03 | 17.03 (20.99) | 14.53 (58.71) | 0.06 | 108.59 (118.97) | 107.60 (113.33) | 0.01 | 73.42 (94.13) | 79.35 (98.03) | 0.00 |
| Missing; n (%) | 471 (6.4%) | 263 (6.7%) | -0.01 | 1,064 (7.6%) | 305 (7.8%) | -0.01 | 1,114 (3.4%) | 643 (3.8%) | -0.02 | 2649 (4.9%) | 1211 (4.9%) | 0.00 |
| Colonoscopy; n (%) | 293 (4.0%) | 150 (3.8%) | 0.01 | 631 (4.5%) | 158 (4.0%) | 0.02 | 1,423 (4.4%) | 690 (4.1%) | 0.01 | 2347 (4.3%) | 998 (4.1%) | 0.01 |
| Fecal occult blood (FOB) test; n (%) | 275 (3.7%)<br>1.060 (14.3%) | 117 (3.0%)<br>612 (15.5%) | 0.04<br>-0.03 | 517 (3.7%)<br>1,272 (9.1%) | 97 (2.5%)<br>355 (9.1%) | 0.07<br>0.00 | 879 (2.7%)<br>9.282 (28.5%) | 487 (2.9%)<br>4,854 (29.0%) | -0.01<br>-0.01 | 1671 (3.1%)<br>11614 (21.5%) | 701 (2.9%)<br>5821 (23.7%) | 0.01<br>-0.05 |
| Flu vaccine; n (%)<br>Mammogram; n (%) | 1,060 (14.3%)<br>745 (10.0%) | 612 (15.5%)<br>421 (10.7%) | -0.03<br>-0.02 | 1,272 (9.1%)<br>1,269 (9.1%) | 355 (9.1%)<br>351 (9.0%) | 0.00 | 9,282 (28.5%)<br>3,468 (10.6%) | 4,854 (29.0%)<br>1,907 (11.4%) | -0.01<br>-0.03 | 11614 (21.5%)<br>5482 (10.2%) | 5821 (23.7%)<br>2679 (10.9%) | -0.05<br>-0.02 |
| Pap smear; n (%) | 353 (4.8%) | 421 (10.7%)<br>171 (4.3%) | 0.02 | 991 (7.1%) | 291 (7.4%) | -0.01 | 841 (2.6%) | 453 (2.7%) | -0.03 | 2185 (4.0%) | 915 (3.7%) | 0.02 |
| Prieumonia vaccine; n (%) | 693 (9.3%) | 688 (17.5%) | -0.24 | 499 (3.6%) | 264 (6.8%) | -0.01 | 4,756 (14.6%) | 3,881 (23.2%) | -0.01 | 5948 (11.0%) | 4833 (19.6%) | -0.24 |
| | (5/0) | (/0) | | (2.070) | == : (=:0/0) | | ., (=/0) | , (/-) | | (0/0) | () | |

| Marches Marc | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| March Marc | PSA test or Prostate exam for DRE; n (%) | | | -0.03 | 1,136 (8.1%) | 325 (8.3%) | -0.01 | 3,297 (10.1%) | 1,947 (11.6%) | -0.05 | | 2705 (11.0%) | |
| Martin M | | | | | | | | | ( ) | | | (,- | |
| March Marc | Use of CNS stimulants; n (%) | 52 (0.7%) | 26 (0.7%) | 0.00 | 188 (1.3%) | 72 (1.8%) | -0.04 | 95 (0.3%) | 68 (0.4%) | -0.02 | 335 (0.6%) | 166 (0.7%) | -0.01 |
| March Marc | Use of estrogens, progestins, androgens; n (%) | 469 (6.3%) | 238 (6.0%) | 0.01 | 1,441 (10.3%) | 456 (11.7%) | -0.04 | 1,116 (3.4%) | 615 (3.7%) | -0.02 | 3026 (5.6%) | 1309 (5.3%) | 0.01 |
| March Marc | Use of Angiogenesis inhibitors; n (%) | ** (0.0%) | ** (0.1%) | -0.04 | ** (0.1%) | ** (0.2%) | -0.03 | 29 (0.1%) | 16 (0.1%) | 0.00 | #VALUE! | #VALUE! | #VALUE! |
| March Marc | | 35 (0.5%) | ** (0.3%) | 0.03 | 132 (0.9%) | 14 (0.4%) | 0.06 | 41 (0.1%) | 16 (0.1%) | 0.00 | 208 (0.4%) | #VALUE! | #VALUE! |
| March Control Contro | | | | 0.15 | 240 (1.7%) | | 0.13 | 387 (1.2%) | 24 (0.1%) | 0.14 | 747 (1.4%) | #VALUE! | #VALUE! |
| Control proposed Control pro | | , | | | | , | | | | | , , | | |
| Control Cont | | 0 (0.0%) | 0 (0.0%) | #DIV/01 | 0 (0.0%) | 0 (0.0%) | #DIV/01 | 0 (0.0%) | 0 (0.0%) | #DIV/01 | 0 (0.0%) | 0 (0.0%) | #DIV/01 |
| Part | | | | | | | | | | | | | |
| Part | | | | | | | | | | | | | |
| Part | | (0.0%) | (0.170) | -0.04 | (0.170) | (0.170) | 0.00 | 24 (0.176) | 22 (0.1%) | 0.00 | #VALUE: | #VALUE: | #VALUE: |
| Part | | 0.05 (0.37) | 0.11 (0.36) | 0.16 | 0.05 (0.35) | 0.07 (0.30) | 0.04 | 0.00 (0.30) | 0.11 (0.24) | 0.00 | 0.07 (0.30) | 0.10/0.24\ | 0.00 |
| Part | | 0.00 (0.27) | 0.11(0.30) | -0.10 | 0.00 (0.20) | 0.07 (0.25) | -0.04 | 0.08 (0.30) | 0.11(0.54) | -0.05 | 0.07 (0.29) | 0.10 (0.54) | 0.00 |
| Part | | | | | () | / | | | | | | | |
| Person P | | 0.14 (0.66) | 0.18 (0.85) | -0.05 | 0.12 (0.62) | 0.17(0.72) | -0.07 | 0.15 (0.72) | 0.17(0.67) | -0.03 | 0.14 (0.69) | 0.17(0.71) | 0.00 |
| Part | | | | | | | | | | | | | |
| Part | | 1.04 (2.19) | 0.96 (1.60) | 0.04 | 0.72 (1.79) | 0.70 (1.51) | 0.01 | 0.62 (1.10) | 0.61 (0.89) | 0.01 | 0.70 (1.49) | 0.68 (1.15) | 0.00 |
| Marie Mari | | | | | | | | | | | | | |
| Part | | 0.00 (0.02) | 0.00 (0.00) | 0.00 | 0.00 (0.03) | 0.00 (0.03) | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 |
| March Marc | HAS-BLED Score (ICD-9 and ICD-10), 180 days | | | | | | | | | | | | |
| March Marc | mean (sd) | 2.86 (1.05) | 2.80 (1.04) | 0.06 | 2.41 (1.01) | 2.32 (0.98) | 0.09 | 3.46 (0.81) | 3.40 (0.82) | 0.07 | 3.11 (0.90) | 3.13 (0.89) | 0.00 |
| Part | N of Generic name drugs | | | | | | | | | | | | |
| March Marc | mean (sd) | 18.04 (16.90) | 16.55 (17.28) | 0.09 | 14.06 (11.77) | 13.04 (12.54) | 0.08 | 19.33 (15.03) | 17.38 (15.17) | 0.13 | 17.79 (14.54) | 16.56 (15.15) | 0.00 |
| Part | | | | | | | | | | | | | |
| Control Cont | | 3.33 (5.27) | 3.81 (4.55) | -0.10 | 3.46 (4.75) | 3.79 (3.90) | -0.08 | 3.58 (5.38) | 4.07 (4.63) | -0.10 | 3.51 (5.21) | 3.98 (4.51) | 0.00 |
| | | | | | | | | | ( , | | , | - , , | |
| Part Principal 19.10 19. | | | | | | | | | | | | | |
| Fin December December Decem | | | | | | | | | | | | | |
| Composition effects (as of part) Composition ef | | | | , | | | | , | - ( - , | , | | | |
| State Content of the Content of Content | | | | | | | | , , | , , | | | | |
| 18.5 m/s 1.3 | | 252 (3.4%) | 86 (2.2%) | #DIV/0! | 501 (3.6%) | 130 (3.3%) | #DIV/0! | 632 (1.9%) | 214 (1.3%) | #DIV/0! | 501 (3.6%) | 130 (3.3%) | 0.02 |
| International refrequentional part international pa | | | | | | | | | | | | | |
| Paper Pape | 183 days; n (%) | 1,806 (24.4%) | 910 (23.1%) | 0.03 | 2,635 (18.9%) | 692 (17.7%) | 0.03 | 9,089 (27.9%) | 4,176 (24.9%) | 0.07 | 13530 (25.1%) | 5778 (23.5%) | 0.04 |
| Property | Intracranial or retroperitoneal hemorrhage: 1 | | | | | | | | | | | | |
| Page Dept | inpatient or 2 outpatient claims within 183 days; n | | | | | | | | | | | | |
| Major Sergir, 1963 9.56 7.86 9.50 9.00/10 1.309 6.46 1.309 6.46 1.309 6.40 | (%) | ** (0.1%) | ** (0.1%) | 0.00 | 12 (0.1%) | 0 (0.0%) | 0.04 | 42 (0.1%) | 12 (0.1%) | 0.00 | #VALUE! | #VALUE! | #VALUE! |
| | Peptic Ulcer Disease; n (%) | 1,859 (25.1%) | 979 (24.8%) | 0.01 | 2,501 (17.9%) | 762 (19.5%) | -0.04 | 9,584 (29.4%) | 4,607 (27.5%) | 0.04 | 13944 (25.8%) | 6348 (25.8%) | 0.00 |
| Dept | Major Surgery ; n (%) | 566 (7.6%) | 355 (9.0%) | #DIV/0! | 1,309 (9.4%) | 327 (8.4%) | #DIV/0! | 2,682 (8.2%) | 1,655 (9.9%) | #DIV/0! | 1,309 (9.4%) | 327 (8.4%) | 0.04 |
| Lower Lowe | | 0 (0.0%) | 0 (0.0%) | #DIV/0! | | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Profession 19 19 19 19 19 19 19 1 | | | | #DIV/0! | | | #DIV/0! | | | #DIV/0! | | | #DIV/0! |
| Chem | | 30 (0.4%) | 13 (0.3%) | 0.02 | 85 (0.6%) | 42 (1.1%) | -0.05 | ** (0.0%) | ** (0.0%) | #DIV/01 | #VALUE! | | #VALUE! |
| Processor Pis 92 12 24 97 17 18 58 18 18 18 18 18 18 | | | | | | | | (,-) | | | | | |
| Part | Other bleeds: n (%) | 430 (5.8%) | 200 (5.1%) | 0.03 | 796 (5.7%) | 218 (5.6%) | 0.00 | 1 841 (5 6%) | 769 (4 6%) | | 3067 (5.7%) | 1187 (4.8%) | |
| Application (Ps) Application (Ps) Application (Ps) *** (0.15) **** (0.15) | | | | | | | | | | | | | |
| Application Contemp | Prior cancer; n (%) | 922 (12.4%) | 707 (17.9%) | -0.15 | 1,383 (9.9%) | 519 (13.3%) | -0.11 | 4,862 (14.9%) | 3,362 (20.1%) | -0.14 | 7167 (13.3%) | 4588 (18.7%) | -0.15 |
| Policy P | Prior cancer; n (%)<br>Antibiotics; n (%) | 922 (12.4%)<br>3,535 (47.7%) 1,9 | 707 (17.9%)<br>930 (49.0%) | -0.15<br>#DIV/0! | 1,383 (9.9%)<br>7,040 (50.4%) | 519 (13.3%)<br>2,046 (52.4%) | -0.11<br>#DIV/0! | 4,862 (14.9%)<br>17,449 (53.5%) | 3,362 (20.1%)<br>9,034 (53.9%) | -0.14<br>#DIV/0! | 7167 (13.3%)<br>7,040 (50.4%) | 4588 (18.7%)<br>2,046 (52.4%) | -0.15<br>-0.04 |
| Post | Prior cancer; n (%)<br>Antibiotics; n (%)<br>Aspirin; n (%) | 922 (12.4%)<br>3,535 (47.7%) 1,9<br>44 (0.6%) | 707 (17.9%)<br>930 (49.0%)<br>31 (0.8%) | -0.15<br>#DIV/0!<br>-0.02 | 1,383 (9.9%)<br>7,040 (50.4%)<br>160 (1.1%) | 519 (13.3%)<br>2,046 (52.4%)<br>63 (1.6%) | -0.11<br>#DIV/0!<br>-0.04 | 4,862 (14.9%)<br>17,449 (53.5%)<br>146 (0.4%) | 3,362 (20.1%)<br>9,034 (53.9%)<br>67 (0.4%) | -0.14<br>#DIV/0!<br>0.00 | 7167 (13.3%)<br>7,040 (50.4%)<br>350 (0.6%) | 4588 (18.7%)<br>2,046 (52.4%)<br>161 (0.7%) | -0.15<br>-0.04<br>-0.01 |
| Chine patriagnote; Ne (N) (10) (13) | Prior cancer; n (%)<br>Antibiotics; n (%)<br>Aspirin; n (%)<br>Aspirin/dipyridamole; n (%) | 922 (12.4%)<br>3,535 (47.7%) 1,5<br>44 (0.6%)<br>** (0.1%) | 707 (17.9%)<br>930 (49.0%)<br>31 (0.8%)<br>** (0.1%) | -0.15<br>#DIV/0!<br>-0.02<br>0.00 | 1,383 (9.9%)<br>7,040 (50.4%)<br>160 (1.1%)<br>22 (0.2%) | 519 (13.3%)<br>2,046 (52.4%)<br>63 (1.6%)<br>** (0.1%) | -0.11<br>#DIV/0!<br>-0.04<br>0.03 | 4,862 (14.9%)<br>17,449 (53.5%)<br>146 (0.4%)<br>113 (0.3%) | 3,362 (20.1%)<br>9,034 (53.9%)<br>67 (0.4%)<br>45 (0.3%) | -0.14<br>#DIV/0!<br>0.00<br>0.00 | 7167 (13.3%)<br>7,040 (50.4%)<br>350 (0.6%)<br>#VALUE! | 4588 (18.7%)<br>2,046 (52.4%)<br>161 (0.7%)<br>#VALUE! | -0.15<br>-0.04<br>-0.01<br>#VALUE! |
| Number of flipid tests ordered | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) | 922 (12.4%)<br>3,535 (47.7%) 1,9<br>44 (0.6%)<br>** (0.1%)<br>21 (0.3%) | 707 (17.9%)<br>930 (49.0%)<br>31 (0.8%)<br>** (0.1%)<br>** (0.3%) | -0.15<br>#DIV/0!<br>-0.02<br>0.00<br>0.00 | 1,383 (9.9%)<br>7,040 (50.4%)<br>160 (1.1%)<br>22 (0.2%)<br>67 (0.5%) | 519 (13.3%)<br>2,046 (52.4%)<br>63 (1.6%)<br>** (0.1%)<br>** (0.3%) | -0.11<br>#DIV/0!<br>-0.04<br>0.03<br>0.03 | 4,862 (14.9%)<br>17,449 (53.5%)<br>146 (0.4%)<br>113 (0.3%)<br>181 (0.6%) | 3,362 (20.1%)<br>9,034 (53.9%)<br>67 (0.4%)<br>45 (0.3%)<br>100 (0.6%) | -0.14<br>#DIV/0!<br>0.00<br>0.00<br>0.00 | 7167 (13.3%)<br>7,040 (50.4%)<br>350 (0.6%)<br>#VALUE!<br>269 (0.5%) | 4588 (18.7%)<br>2,046 (52.4%)<br>161 (0.7%)<br>#VALUE!<br>#VALUE! | -0.15<br>-0.04<br>-0.01<br>#VALUE!<br>#VALUE! |
| | Prior cancer; n (%) Antibiotics, n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) | 922 (12.4%) 3,535 (47.7%) 1,9 44 (0.6%) ** (0.1%) 21 (0.3%) 1,375 (18.5%) | 707 (17.9%) 930 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) | -0.15<br>#DIV/0!<br>-0.02<br>0.00<br>0.00<br>0.04 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.3%) 720 (18.4%) | -0.11<br>#DIV/0!<br>-0.04<br>0.03<br>0.03<br>0.03 | 4,862 (14.9%)<br>17,449 (53.5%)<br>146 (0.4%)<br>113 (0.3%)<br>181 (0.6%)<br>7,501 (23.0%) | 3,362 (20.1%)<br>9,034 (53.9%)<br>67 (0.4%)<br>45 (0.3%)<br>100 (0.6%)<br>3,737 (22.3%) | -0.14<br>#DIV/0!<br>0.00<br>0.00<br>0.00<br>0.02 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUE! 269 (0.5%) 11632 (21.5%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #VALUE! #VALUE! 5124 (20.8%) | -0.15<br>-0.04<br>-0.01<br>#VALUE!<br>#VALUE!<br>0.02 |
| Proton pump inhibitor; n (%) 1,695 (2.9 %) 892 (2.5 %) 0.01 3,099 (2.2 %) 8.5 (2.1 %) 0.03 10,056 (3.8 %) 4,868 (29.1 %) 0.04 14850 (77.5 %) 5.55 (5.5 %) 1.00 (0.0 %) 0.04 27 (0.0 %) 0.04 14850 (77.5 %) 0.00 2 265 (5.5 %) 133 (2.5 %) 0.00 2 245 (5.5 %) 1.00 (0.0 %) 0.06 0.06 0.06 0.06 0.06 0.06 0.06 0.0 | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) | 922 (12.4%) 3,535 (47.7%) 1,9 44 (0.6%) ** (0.1%) 21 (0.3%) 1,375 (18.5%) | 707 (17.9%) 930 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) | -0.15<br>#DIV/0!<br>-0.02<br>0.00<br>0.00<br>0.04 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.3%) 720 (18.4%) | -0.11<br>#DIV/0!<br>-0.04<br>0.03<br>0.03<br>0.03 | 4,862 (14.9%)<br>17,449 (53.5%)<br>146 (0.4%)<br>113 (0.3%)<br>181 (0.6%)<br>7,501 (23.0%) | 3,362 (20.1%)<br>9,034 (53.9%)<br>67 (0.4%)<br>45 (0.3%)<br>100 (0.6%)<br>3,737 (22.3%) | -0.14<br>#DIV/0!<br>0.00<br>0.00<br>0.00<br>0.02 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUE! 269 (0.5%) 11632 (21.5%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #VALUE! #VALUE! 5124 (20.8%) | -0.15<br>-0.04<br>-0.01<br>#VALUE!<br>#VALUE!<br>0.02 |
| 12 12 12 13 14 15 15 15 15 15 15 15 | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) | 922 (12.4%) 3,535 (47.7%) 1,1 44 (0.5%) ** (0.1%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) | 707 (17.9%) 930 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) | -0.15<br>#DIV/0!<br>-0.02<br>0.00<br>0.00<br>0.04<br>-0.02 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.3%) 720 (18.4%) 78 (2.0%) | -0.11<br>#DIV/0!<br>-0.04<br>0.03<br>0.03<br>0.03<br>-0.04 | 4,862 (14.9%)<br>17,449 (53.5%)<br>146 (0.4%)<br>113 (0.3%)<br>181 (0.6%)<br>7,501 (23.0%)<br>554 (1.7%) | 3,362 (20.1%)<br>9,034 (53.9%)<br>67 (0.4%)<br>45 (0.3%)<br>100 (0.6%)<br>3,737 (22.3%)<br>258 (1.5%) | -0.14<br>#DIV/0!<br>0.00<br>0.00<br>0.00<br>0.02<br>0.02 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #VALUE! #VALUE! 5124 (20.8%) 394 (1.6%) | -0.15<br>-0.04<br>-0.01<br>#VALUE!<br>#VALUE!<br>0.02<br>0.00 |
| Victor V | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests ordered | 922 (12.4%) 3,535 (47.7%) 1,1 44 (0.5%) ** (0.1%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) | 707 (17.9%) 930 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) | -0.15<br>#DIV/0!<br>-0.02<br>0.00<br>0.00<br>0.04<br>-0.02 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.3%) 720 (18.4%) 78 (2.0%) | -0.11<br>#DIV/0!<br>-0.04<br>0.03<br>0.03<br>0.03<br>-0.04 | 4,862 (14.9%)<br>17,449 (53.5%)<br>146 (0.4%)<br>113 (0.3%)<br>181 (0.6%)<br>7,501 (23.0%)<br>554 (1.7%) | 3,362 (20.1%)<br>9,034 (53.9%)<br>67 (0.4%)<br>45 (0.3%)<br>100 (0.6%)<br>3,737 (22.3%)<br>258 (1.5%) | -0.14<br>#DIV/0!<br>0.00<br>0.00<br>0.00<br>0.02<br>0.02 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #VALUE! #VALUE! 5124 (20.8%) 394 (1.6%) | -0.15<br>-0.04<br>-0.01<br>#VALUE!<br>#VALUE!<br>0.02<br>0.00 |
| Victor V | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) | 922 (12.4%) 1, 3,535 (47.7%) 44 (0.6%) ** (0.1%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) | 707 (17.9%) 930 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) | -0.15<br>#DIV/0!<br>-0.02<br>0.00<br>0.00<br>0.04<br>-0.02 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.3%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) | -0.11<br>#DIV/0!<br>-0.04<br>0.03<br>0.03<br>-0.04 | 4,862 (14.9%)<br>17,449 (53.5%)<br>146 (0.4%)<br>113 (0.3%)<br>181 (0.6%)<br>7,501 (23.0%)<br>554 (1.7%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) | -0.14<br>#DIV/0!<br>0.00<br>0.00<br>0.00<br>0.02<br>0.02 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #VALUE! #VALUE! 5124 (20.8%) 394 (1.6%) 0.52 (0.81) | -0.15<br>-0.04<br>-0.01<br>#VALUE!<br>#VALUE!<br>0.02<br>0.00 |
| Number of IFNR (prothrombin) tests ordered | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) ** (0.1%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) | 707 (17.9%)<br>930 (49.0%)<br>31 (0.8%)<br>** (0.1%)<br>** (0.3%)<br>667 (16.9%)<br>58 (1.5%)<br>0.48 (0.78)<br>892 (22.6%) | -0.15<br>#DIV/0!<br>-0.02<br>0.00<br>0.00<br>0.04<br>-0.02 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.3%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) | -0.11<br>#DIV/0!<br>-0.04<br>0.03<br>0.03<br>-0.04<br>-0.02 | 4,862 (14.9%)<br>17,449 (53.5%)<br>146 (0.4%)<br>113 (0.3%)<br>181 (0.6%)<br>7,501 (23.0%)<br>554 (1.7%)<br>0.54 (0.79)<br>10,056 (30.8%) | 3,362 (20.1%)<br>9,034 (53.9%)<br>67 (0.4%)<br>45 (0.3%)<br>100 (0.6%)<br>3,737 (22.3%)<br>258 (1.5%)<br>0.56 (0.80)<br>4,868 (29.1%) | -0.14<br>#DIV/0!<br>0.00<br>0.00<br>0.00<br>0.02<br>0.02 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #VALUE! #VALUE! 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) | -0.15<br>-0.04<br>-0.01<br>#VALUE!<br>#VALUE!<br>0.02<br>0.00 |
| men (d) | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.5%) 40 (0.5%) 21 (0.3%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) | 707 (17.9%) 930 (49.0%) 31 (0.8%) **(0.1%) **(0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) | -0.15<br>#DIV/0!<br>-0.02<br>0.00<br>0.00<br>-0.04<br>-0.02<br>0.01 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.3%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) | -0.11<br>#DIV/0!<br>-0.04<br>0.03<br>0.03<br>-0.04<br>-0.02<br>0.03<br>-0.05 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 7,501 (23.0%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.6%) | 3,362 (20.1%)<br>9,034 (53.9%)<br>67 (0.4%)<br>45 (0.3%)<br>100 (0.6%)<br>3,737 (22.3%)<br>258 (1.5%)<br>0.56 (0.80)<br>4,868 (29.1%)<br>1,010 (6.0%) | -0.14<br>#DIV/0!<br>0.00<br>0.00<br>0.00<br>0.02<br>0.02<br>-0.03<br>0.04<br>0.02 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #VALUE! #VALUE! 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) | -0.15<br>-0.04<br>-0.01<br>#VALUE!<br>#VALUE!<br>0.02<br>0.00<br>0.00<br>0.02<br>0.00 |
| Treating prescriber - Cardiologist; n (%) | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.5%) 40 (0.5%) 21 (0.3%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) | 707 (17.9%) 930 (49.0%) 31 (0.8%) **(0.1%) **(0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) | -0.15<br>#DIV/0!<br>-0.02<br>0.00<br>0.00<br>-0.04<br>-0.02<br>0.01 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.3%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) | -0.11<br>#DIV/0!<br>-0.04<br>0.03<br>0.03<br>-0.04<br>-0.02<br>0.03<br>-0.05 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 7,501 (23.0%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.6%) | 3,362 (20.1%)<br>9,034 (53.9%)<br>67 (0.4%)<br>45 (0.3%)<br>100 (0.6%)<br>3,737 (22.3%)<br>258 (1.5%)<br>0.56 (0.80)<br>4,868 (29.1%)<br>1,010 (6.0%) | -0.14<br>#DIV/0!<br>0.00<br>0.00<br>0.00<br>0.02<br>0.02<br>-0.03<br>0.04<br>0.02 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #VALUE! #VALUE! 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) | -0.15<br>-0.04<br>-0.01<br>#VALUE!<br>#VALUE!<br>0.02<br>0.00<br>0.00<br>0.02<br>0.00 |
| Treating prescriber - Primary Care Physician; n (%) | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin/dipyridamole; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests ordered | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) ** (0.1%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) ** (0.1%) | 707 (17.9%) 31 (0.9%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (1.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) | -0.15<br>#DIV/0!<br>-0.02<br>-0.00<br>-0.00<br>-0.04<br>-0.02<br>-0.01<br>-0.01<br>-0.01 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.3%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) | -0.11<br>#DIV/01<br>-0.04<br>-0.03<br>-0.03<br>-0.04<br>-0.02<br>-0.02<br>0.03<br>-0.05<br>-0.05 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 7,501 (2.3.0%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.6%) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) | -0.14 #DIV/0! 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/0! | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) #VALUE! | 4588 (18.7%) 2,046 (52.4%) 151 (0.7%) #VALUE! #VALUE! 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUE! | -0.15 -0.04 -0.01 #VALUE! #VALUE! 0.02 0.00 0.00 0.02 0.00 #VALUE! |
| Treating prescriber; n (%) 7,407 (99.9%) 3,938 (99.9%) 295 (7.5%) 295 (7. | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin k therapy; n (%) Number of lNR (prothrombin) tests orderedmean (sd) | 922 (12.4%) 3,535 (47.7%) 44 (0.5%) 40 (0.5%) 21 (0.3%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 4 (0.1%) 0.73 (1.63) | 707 (17.9%) 33 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) | -0.15 #DIV/0! -0.02 -0.00 -0.00 -0.04 -0.02 -0.01 -0.01 -0.04 -0.15 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) | -0.11<br>#DIV/01<br>-0.04<br>-0.03<br>-0.03<br>-0.04<br>-0.02<br>-0.03<br>-0.05<br>-0.06 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 7,501 (23.0%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.6%) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUEI 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) #VALUEI | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #VALUEI 17A-VLUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI | -0.15 -0.04 -0.01 #VALUE! #VALUE! 0.02 0.00 0.00 0.02 0.00 #VALUE! |
| Alpha blockers; n (%) 527 (7.1%) 295 (7.5%) -0.02 872 (6.2%) 204 (5.2%) 0.04 3,226 (9.9%) 1,744 (10.4%) 0.02 4625 (8.6%) 2243 (9.1%) -0.02 CHAZDS2 VASC score, 180 days, V | Prior cancer; n (%) Antibiotics, n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 1,(1.5%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 10 (1.3%) 0.73 (1.63) 2,275 (30.7%) | 707 (17.9%) 930 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) | -0.15<br>#DIV/OI<br>-0.02<br>0.00<br>0.00<br>0.04<br>-0.02<br>0.01<br>0.01<br>-0.01<br>-0.04<br>0.15 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) | -0.11<br>#DIV/0!<br>-0.04<br>0.03<br>0.03<br>-0.04<br>-0.02<br>0.03<br>-0.05<br>0.06 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 7,501 (23.0%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.6%) **(0.0%) 0.58 (1.01) 11,149 (34.2%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUEI 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) #VALUEI 0.59 (1.17) 17762 (32.9%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #NALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (32.8%) | -0.15 -0.04 -0.01 #VALUE! #VALUE! 0.02 0.00 0.02 0.00 #VALUE! |
| CHA2DS2 VASc score, 180 days, V mean (sd) 3.72 (1.81) 2.57 (1.68) 0.66 3.50 (1.56) 2.64 (1.73) 0.52 4.65 (1.70) 3.61 (1.83) 0.59 4.22 (1.68) 3.29 (1.79) 0.01 Use of Prasugrel, n (%) 13 (0.2%) ** (0.1%) 0.03 27 (0.2%) ** (0.3%) 0.02 ** (0.3%) 0.02 ** (0.0%) ** (0.1%) ** (0.0%) ** (0.1%) ** (0.0%) ** (0. | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of link (prothrombin) tests orderedmean (sd) Treating prescriber - Primary Care Physician; n (%) | 3,535 (47.7%) 44 (0.6%) 44 (0.6%) 1,1,1 (0.1%) 1,1 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 41 (0.1%) 0.73 (1.63) 2,275 (0.7%) 6,535 (88.2%) | 707 (17.9%) 330 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) | -0.15 #DIV/01 -0.02 -0.00 -0.00 -0.04 -0.02 -0.01 -0.01 -0.04 -0.15 -0.04 -0.15 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.5%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) | 519 (13.3 %) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.3%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) | -0.11<br>#DIV/0!<br>-0.04<br>-0.03<br>-0.03<br>-0.04<br>-0.02<br>-0.03<br>-0.05<br>-0.06<br>-0.06<br>-0.09<br>-0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.5%) 7,501 (23.0%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.6%) **(0.0%) 0.58 (10.1) 11,149 (34.2%) 13,113 (40.2%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) *** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) | -0.14 #DIV/01 0.00 0.00 0.00 0.02 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) #VALUE! 0.59 (1.17) 17762 (32.9%) 254319 (47.1%) | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUE! 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUE! 0.54 (0.82) 8064 (22.8%) 11218 (45.5%) | -0.15 -0.04 -0.01 #VALUE! #VALUE! 0.02 0.00 0.02 0.00 #VALUE! |
| men (sc) 3.72 (1.81) 2.57 (1.68) 0.66 3.50 (1.56) 2.64 (1.73) 0.52 4.65 (1.70) 3.61 (1.83) 0.59 4.22 (1.68) 3.29 (1.79) 0.01 Use of Prasugref; n (%) 13 (0.2%) *** (0.1%) 0.03 27 (0.2%) *** (0.3%) -0.02 **** (0.0%) **** | Prior cancer; n (%) Antibiotics, n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of liNR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Primary Care Physician; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 44 (0.6%) 42 (1.0%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 42 (0.1%) 0.73 (1.63) 2,275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) | 707 (17.9%) 31 (0.9%) 31 (0.8%) ** (0.1%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) | -0.15 #DIV/01 -0.02 -0.00 -0.00 -0.00 -0.04 -0.02 -0.01 -0.01 -0.04 -0.04 -0.09 -0.04 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) | -0.11<br>#DIV/0!<br>-0.04<br>0.03<br>0.03<br>-0.04<br>-0.02<br>0.03<br>-0.05<br>0.06<br>-0.09<br>-0.09 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 7,501 (23.0%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.6%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 32,361 (99.2%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 16,705 (99.7%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/0! | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUEI 269 (0.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) #VALUEI 0.59 (1.17) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (32.8%) 11218 (45.6%) 24375 (99.1%) | -0.15 -0.04 -0.01 #WALUE! 0.02 0.00 0.00 0.02 0.00 #VALUE! 0.00 0.00 -0.00 0.00 0.00 0.00 0.00 0. |
| Use of Prasugrel; n (%) | Prior cancer; n (%) Antibiotics, n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 44 (0.6%) 42 (1.0%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 42 (0.1%) 0.73 (1.63) 2,275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) | 707 (17.9%) 31 (0.9%) 31 (0.8%) ** (0.1%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) | -0.15 #DIV/01 -0.02 -0.00 -0.00 -0.00 -0.04 -0.02 -0.01 -0.01 -0.04 -0.04 -0.09 -0.04 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) | -0.11<br>#DIV/0!<br>-0.04<br>0.03<br>0.03<br>-0.04<br>-0.02<br>0.03<br>-0.05<br>0.06<br>-0.09<br>-0.09 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 7,501 (23.0%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.6%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 32,361 (99.2%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 16,705 (99.7%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/0! | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUEI 269 (0.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) #VALUEI 0.59 (1.17) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (32.8%) 11218 (45.6%) 24375 (99.1%) | -0.15 -0.04 -0.01 #WALUE! 0.02 0.00 0.00 0.02 0.00 #VALUE! 0.00 0.00 -0.00 0.00 0.00 0.00 0.00 0. |
| Use of Loop Diurettics-other diurettics-other hypertension drugs; n (%) 1,136 (15.3%) 532 (13.5%) 0.05 1,808 (12.9%) 427 (10.9%) 0.06 7,645 (23.4%) 3,294 (19.7%) 0.09 10589 (19.6%) 4253 (17.3%) 0.06 Commercial (19.5%) Model (24.4%) Model (2 | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of link (prothrombin) tests orderedmean (sd) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DSZ VASC score, 180 days, V | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 1,1,1 (0.1%) 1,21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 10.73 (1.63) 2,275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) | 707 (17.9%) 330 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) | -0.15 #DIV/01 -0.02 -0.00 -0.00 -0.04 -0.02 -0.01 -0.01 -0.04 -0.15 -0.04 -0.19 -0.00 -0.02 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) | 519 (13.3 %) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.3%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (34.4%) 3,732 (95.5%) 204 (5.2%) | -0.11 #DIV/0! -0.04 0.03 0.03 0.03 -0.04 -0.02 0.03 -0.05 0.06 0.06 -0.09 -0.04 -0.01 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.5%) 7,501 (23.0%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.6%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 32,361 (99.2%) 3,226 (9.9%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 16,705 (99.7%) 1,744 (10.4%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUEI 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) #VALUEI 0.59 (1.17) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (27.8%) 12128 (45.6%) 24375 (99.1%) | -0.15 -0.04 -0.01 #WALUE! #VALUE! #0.02 0.00 0.02 0.00 #VALUE! 0.00 0.00 -0.00 -0.00 -0.00 -0.00 -0.00 -0.00 |
| hypertension drugs; n(%) 1,136 (15.3%) 532 (13.5%) 532 (13.5%) 532 (13.5%) 0.05 1,808 (12.9%) 427 (10.9%) 0.06 7,645 (23.4%) 3,294 (19.7%) 0.09 10589 (19.6%) 4253 (17.3%) 0.06 Commercial vs Medicare Advantage. Business Type Code - CORRECT ONE - OPTION | Prior cancer; n (%) Antibiotics, n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) Off inhibitors; n (%) Off inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of liNR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 44 (0.6%) 42 (0.1%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 42 (0.1%) 0.73 (1.63) 2,275 (30.7%) 6,535 (38.2%) 7,407 (99.2%) 527 (7.1%) | 707 (17.9%) 31 (0.8%) ** (0.1%) ** (0.1%) *667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1.282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) | -0.15 #DIV/01 -0.02 -0.00 -0.00 -0.04 -0.02 -0.01 -0.01 -0.04 -0.15 -0.04 -0.19 -0.00 -0.02 -0.02 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) | -0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.05 -0.06 -0.09 -0.04 -0.01 -0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 7,501 (22.0%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.6%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 16,705 (99.7%) 1,744 (10.4%) 3.61 (1.83) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/0! 0.02 0.04 0.05 -0.07 -0.02 | 7167 (33.3%) 7,040 (50.4%) 350 (0.6%) #VALUEL 269 (0.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) 2966 (5.5%) #VALUEL 0.59 (1.17) 17762 (32.9%) 2419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) 1359 (5.5%) 1478 (20.82) 8064 (22.8%) 1218 (45.6%) 24375 (99.1%) 2243 (9.1%) | -0.15 -0.04 -0.01 #WALUE! 0.02 0.00 0.00 0.02 0.00 #WALUE! 0.00 0.00 0.00 -0.00 0.00 0.00 0.00 0. |
| Commercial vs Medicare Advantage Business Type Code - CORRECT ONE - OPTIVM 2,640 (35.6%) 1277 (32.4%) 0.07 3,998 (28.6%) 835 (21.4%) 0.17 - | Prior cancer; n (%) Antibiotics, n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) Use of Prasugrel; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 44 (0.6%) 42 (0.1%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 42 (0.1%) 0.73 (1.63) 2,275 (30.7%) 6,535 (38.2%) 7,407 (99.2%) 527 (7.1%) | 707 (17.9%) 31 (0.8%) ** (0.1%) ** (0.1%) *667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1.282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) | -0.15 #DIV/01 -0.02 -0.00 -0.00 -0.04 -0.02 -0.01 -0.01 -0.04 -0.15 -0.04 -0.19 -0.00 -0.02 -0.02 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) | -0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.05 -0.06 -0.09 -0.04 -0.01 -0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 7,501 (22.0%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.6%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 16,705 (99.7%) 1,744 (10.4%) 3.61 (1.83) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/0! 0.02 0.04 0.05 -0.07 -0.02 | 7167 (33.3%) 7,040 (50.4%) 350 (0.6%) #VALUEL 269 (0.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) 2966 (5.5%) #VALUEL 0.59 (1.17) 17762 (32.9%) 2419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) 1359 (5.5%) 1478 (20.82) 8064 (22.8%) 1218 (45.6%) 24375 (99.1%) 2243 (9.1%) | -0.15 -0.04 -0.01 #WALUE! 0.02 0.00 0.00 0.02 0.00 #WALUE! 0.00 0.00 0.00 -0.00 0.00 0.00 0.00 0. |
| Code - CORRECTIONE - OPTUM Commercial; n(%) | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of INR (prothrombin) tests orderedmean (sd) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Treating prescriber - Other; n (%) CHA2DS2 VASC score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Frasugrel; n (%) Use of Prasugrel; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 21 (0.3%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) | 707 (17.9%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) | -0.15 #DIV/01 -0.02 0.00 0.00 0.04 -0.02 0.01 0.01 0.04 -0.02 0.15 -0.04 0.15 -0.04 0.19 0.00 -0.02 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (34.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) | 0.11 #DIV/01 -0.04 0.03 0.03 0.03 -0.04 -0.02 0.03 -0.05 0.06 -0.09 -0.04 -0.01 0.04 -0.01 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 45 (0.3%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUEI 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) 2966 (5.5%) 470 (177) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #WALUEI | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (22.8%) 12128 (45.6%) 224375 (99.1%) 2243 (9.1%) 3.29 (1.79) #VALUEI | -0.15 -0.04 -0.01 #VALUE! #VALUE! #VALUE! 0.02 0.00 0.02 0.00 #VALUE! 0.00 0.00 -0.00 0.00 0.00 0.00 0.00 0. |
| Commercial; n (%) 2,640 (35.6%) 1277 (32.4%) 0.07 3,998 (28.6%) 835 (21.4%) 0.17 #VALUE! 6,638 (31.0%) 2112 (26.9%) 0.09Medicare Advantage; n (%) 4,773 (64.4%) 2663 (67.6%) -0.07 9,979 (71.4%) 3073 (78.6%) -0.17 #VALUE! 14,752 (69.0%) 573 (73.1%) -0.09Medicare Advantage Business Type Code | Prior cancer; n (%) Antibiotics, n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) OGP inhibitors; n (%) OGP inhibitors; n (%) OTHER gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of liNR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DSZ VASc score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diuretics+other diuretics+other hypertension drugs; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 21 (0.3%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) | 707 (17.9%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) | -0.15 #DIV/01 -0.02 0.00 0.00 0.04 -0.02 0.01 0.01 0.04 -0.02 0.15 -0.04 0.15 -0.04 0.19 0.00 -0.02 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (34.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) | 0.11 #DIV/01 -0.04 0.03 0.03 0.03 -0.04 -0.02 0.03 -0.05 0.06 -0.09 -0.04 -0.01 0.04 -0.01 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 45 (0.3%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUEI 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) 2966 (5.5%) 470 (177) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #WALUEI | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (22.8%) 12128 (45.6%) 224375 (99.1%) 2243 (9.1%) 3.29 (1.79) #VALUEI | -0.15 -0.04 -0.01 #VALUE! #VALUE! #VALUE! 0.02 0.00 0.02 0.00 #VALUE! 0.00 0.00 -0.00 0.00 0.00 0.00 0.00 0. |
| Medicare Advantage; n (%) 4,773 (64.4%) 2663 (67.6%) -0.07 9,979 (71.4%) 3073 (78.6%) -0.17 + #VALUE! 14,752 (69.0%) 5736 (73.1%) -0.09 Commercial vs Medicare Advantage Business Type CodeCOM = COMMERCIAL; n (%) 2,640 (35.6%) 1,277 (32.4%) 0.07 + #VALUE! 2,640 (35.6%) 1,277 (32.4%) 0.07 + #VALUE! 2,640 (35.6%) 1,277 (32.4%) 0.07 + #VALUE! 4,773 (64.4%) 2,663 (67.6%) 0.07 | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of link (prothrombin) tests orderedmean (sd) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DSZ VAGs core, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diuretics+other diuretics+other hypertension drugs; n (%) Commercial vs Medicare Advantage-Business Type | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 21 (0.3%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) | 707 (17.9%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) | -0.15 #DIV/01 -0.02 0.00 0.00 0.04 -0.02 0.01 0.01 0.04 -0.02 0.15 -0.04 0.15 -0.04 0.19 0.00 -0.02 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (34.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) | 0.11 #DIV/01 -0.04 0.03 0.03 0.03 -0.04 -0.02 0.03 -0.05 0.06 -0.09 -0.04 -0.01 0.04 -0.01 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 45 (0.3%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUEI 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) 2966 (5.5%) 470 (177) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #WALUEI | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (22.8%) 12128 (45.6%) 224375 (99.1%) 2243 (9.1%) 3.29 (1.79) #VALUEI | -0.15 -0.04 -0.01 #VALUE! #VALUE! #VALUE! 0.02 0.00 0.02 0.00 #VALUE! 0.00 0.00 -0.00 0.00 0.00 0.00 0.00 0. |
| Commercial vs Medicare Advantage- Business Type CodeCOM = COMMERCIAL; n (%) 2,640 (35.6%) 1,277 (32.4%) 0.07 #VALUE! 2,640 (35.6%) 1,277 (32.4%) 0.07MCR = MEDICARE; n (%) 4,773 (64.4%) 2,663 (67.6%) -0.07MCR = MEDICARE; n (%) #VALUE! 0,0.0% 2,663 (67.6%) -0.07MCR = MEDICARE; n (%) #VALUE! 0,0.0% 2,663 (67.6%) #DIV/O!NONE = NO BUSINESS LINE CODE (added in 2015); n (%) 0 (0.0%) #DIV/O!UNK = UNIKNOWN (added in 2015); n (%) 0 (0.0%) 0 (0.0%) #DIV/O!UNK = UNIKNOWN (added in 2015); n (%) 0 (0.0%) 0 (0.0%) #DIV/O!UNK = UNIKNOWN (added in 2015); n (%) 0 (0.0%) 0 (0.0%) #DIV/O!UNK = UNIKNOWN (added in 2015); n (%) 0 (0.0%) 0 (0.0%) #DIV/O! | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of liN( prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diurettics+other diuretics+other hypertension drugs; n (%) Commercial vs Medicare Advantage- Business Type Code - CORRECT ONE - OPTUM | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 21 (0.3%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) ** (0.1%) 0.73 (1.63) 2,275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) 1,136 (15.3%) | 707 (17.9%) 31 (0.9%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) 2.57 (1.68) ** (0.1%) | 0.15 #DIV/01 -0.02 0.00 0.00 0.04 -0.02 0.01 0.01 0.04 0.15 -0.04 0.19 0.00 -0.02 0.66 0.03 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0.46 (0.98) 1,377 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) | -0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.06 -0.06 -0.09 -0.01 -0.04 -0.01 -0.04 -0.02 -0.02 -0.03 -0.06 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 45 (0.3%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/0! 0.02 0.04 0.05 -0.07 -0.02 0.59 #DIV/0! | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUEI 269 (0.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) 2966 (5.5%) 2766 (5.5%) 2767 (32.9%) 25419 (47.1%) 53078 (38.3%) 4625 (8.6%) 4.22 (1.68) #WALUEI | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) 1359 (5.5%) 1474 (1.82) 8064 (22.8%) 1218 (45.6%) 22437 (99.1%) 2243 (9.1%) 3.29 (1.79) #VALUEI | -0.15 -0.04 -0.01 #VALUE! 0.02 0.00 0.00 0.02 0.00 #VALUE! 0.00 0.00 0.00 0.00 0.00 0.00 1.00 0.00 |
| Commercial vs Medicare Advantage- Business Type CodeCOM = COMMERCIAL; n (%) 2,640 (35.6%) 1,277 (32.4%) 0.07 #VALUE! 2,640 (35.6%) 1,277 (32.4%) 0.07MCR = MEDICARE; n (%) 4,773 (64.4%) 2,663 (67.6%) -0.07MCR = MEDICARE; n (%) #VALUE! 0,0.0% 2,663 (67.6%) -0.07MCR = MEDICARE; n (%) #VALUE! 0,0.0% 2,663 (67.6%) #DIV/O!NONE = NO BUSINESS LINE CODE (added in 2015); n (%) 0 (0.0%) #DIV/O!UNK = UNIKNOWN (added in 2015); n (%) 0 (0.0%) 0 (0.0%) #DIV/O!UNK = UNIKNOWN (added in 2015); n (%) 0 (0.0%) 0 (0.0%) #DIV/O!UNK = UNIKNOWN (added in 2015); n (%) 0 (0.0%) 0 (0.0%) #DIV/O!UNK = UNIKNOWN (added in 2015); n (%) 0 (0.0%) 0 (0.0%) #DIV/O! | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of liN( prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diurettics+other diuretics+other hypertension drugs; n (%) Commercial vs Medicare Advantage- Business Type Code - CORRECT ONE - OPTUM | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 21 (0.3%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) ** (0.1%) 0.73 (1.63) 2,275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) 1,136 (15.3%) | 707 (17.9%) 31 (0.9%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) 2.57 (1.68) ** (0.1%) | 0.15 #DIV/01 -0.02 0.00 0.00 0.04 -0.02 0.01 0.01 0.04 0.15 -0.04 0.19 0.00 -0.02 0.66 0.03 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 720 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0.46 (0.98) 1,377 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) | -0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.06 -0.06 -0.09 -0.01 -0.04 -0.01 -0.04 -0.02 -0.02 -0.03 -0.06 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 45 (0.3%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/0! 0.02 0.04 0.05 -0.07 -0.02 0.59 #DIV/0! | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUEI 269 (0.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) 2966 (5.5%) 2766 (5.5%) 2767 (32.9%) 25419 (47.1%) 53078 (38.3%) 4625 (8.6%) 4.22 (1.68) #WALUEI | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) 1359 (5.5%) 1474 (1.82) 8064 (22.8%) 1218 (45.6%) 22437 (99.1%) 2243 (9.1%) 3.29 (1.79) #VALUEI | -0.15 -0.04 -0.01 #VALUE! 0.02 0.00 0.00 0.02 0.00 #VALUE! 0.00 0.00 0.00 0.00 0.00 0.00 1.00 0.00 |
| CodeCode | Prior cancer; n (%) Antibiotics, n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of liNR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2D52 VASc score; 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diuretics-other diuretics+other hypertension drugs; n (%) Commercial vs Medicare Advantage-Business Type Code - CORRECT ONE - OPTUMCommercial; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 44 (0.6%) 42 (10.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 4 (0.1%) 0.73 (1.63) 2,275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) 1,136 (15.3%) | 707 (17.9%) 31 (0.8%) ** (0.1%) ** (0.1%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) 2.57 (1.68) ** (0.1%) 532 (13.5%) | 0.15 #DIV/01 -0.02 0.00 0.00 0.04 -0.02 0.01 0.01 -0.01 0.04 0.15 -0.04 0.19 0.00 -0.02 0.66 0.03 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) 1,808 (12.9%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 72 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) 427 (10.9%) | 0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.06 -0.09 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 45 (0.3%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 0.59 #DIV/01 0.09 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) 2966 (5.5%) 476LUE! 0.59 (1.17) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #VALUE! 10589 (19.6%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #NALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (32.8%) 11218 (45.6%) 24375 (99.1%) 2243 (9.1%) 3.29 (1.79) #VALUEI 4253 (17.3%) | -0.15 -0.04 -0.01 #VALUE! 0.02 0.00 0.00 0.02 0.00 #VALUE! 0.00 0.03 -0.07 -0.02 0.01 #VALUE! 0.06 |
| MCR = MEDICARE; n (%) 4,773 (64.4%) 2,663 (67.6%) -0.07 #VALUE! 4,773 (64.4%) 2,663 (67.6%) -0.07 | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other astroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin k therapy; n (%) Number of liNR (prothrombin) tests orderedmean (sd) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASC score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diuretics+other diuretics+other hypertension drugs; n (%) Commercial vs Medicare Advantage-Business Type Code - CORRECT ONE - OPTUMCommercial; n (%)Medicare Advantage; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 44 (0.6%) 42 (10.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 4 (0.1%) 0.73 (1.63) 2,275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) 1,136 (15.3%) | 707 (17.9%) 31 (0.8%) ** (0.1%) ** (0.1%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) 2.57 (1.68) ** (0.1%) 532 (13.5%) | 0.15 #DIV/01 -0.02 0.00 0.00 0.04 -0.02 0.01 0.01 -0.01 0.04 0.15 -0.04 0.19 0.00 -0.02 0.66 0.03 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) 1,808 (12.9%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 72 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) 427 (10.9%) | 0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.06 -0.09 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 45 (0.3%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 0.59 #DIV/01 0.09 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) 2966 (5.5%) 476LUE! 0.59 (1.17) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #VALUE! 10589 (19.6%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #NALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (32.8%) 11218 (45.6%) 24375 (99.1%) 2243 (9.1%) 3.29 (1.79) #VALUEI 4253 (17.3%) | -0.15 -0.04 -0.01 #VALUE! 0.02 0.00 0.00 0.02 0.00 #VALUE! 0.00 0.03 -0.07 -0.02 0.01 #VALUE! 0.06 |
| MCR = MEDICARE; n (%) 4,773 (64.4%) 2,663 (67.6%) -0.07 #VALUE! 4,773 (64.4%) 2,663 (67.6%) -0.07 | Prior cancer; n (%) Antibiotics, n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) Office inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of liNR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) Use of Loop Diuretics-other diuretics-tother hypertension drugs; n (%) Commercial vs Medicare Advantage- Business Type Code - CORRECT ONE - OPTUMCommercial; n (%)Medicare Advantage; n (%) Commercial vs Medicare Advantage- Business Type Commercial vs Medicare Advantage- Business Type | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 44 (0.6%) 42 (10.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 4 (0.1%) 0.73 (1.63) 2,275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) 1,136 (15.3%) | 707 (17.9%) 31 (0.8%) ** (0.1%) ** (0.1%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) 2.57 (1.68) ** (0.1%) 532 (13.5%) | 0.15 #DIV/01 -0.02 0.00 0.00 0.04 -0.02 0.01 0.01 -0.01 0.04 0.15 -0.04 0.19 0.00 -0.02 0.66 0.03 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) 1,808 (12.9%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 72 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) 427 (10.9%) | 0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.06 -0.09 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 45 (0.3%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 0.59 #DIV/01 0.09 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #VALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) 2966 (5.5%) 476LUE! 0.59 (1.17) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #VALUE! 10589 (19.6%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #NALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (32.8%) 11218 (45.6%) 24375 (99.1%) 2243 (9.1%) 3.29 (1.79) #VALUEI 4253 (17.3%) | -0.15 -0.04 -0.01 #VALUE! 0.02 0.00 0.00 0.02 0.00 #VALUE! 0.00 0.03 -0.07 -0.02 0.01 #VALUE! 0.06 |
| MCD = MEDICAID; n (%) 0 (0.0%) #DIV/0! #VALUE! 0 (0.0%) 0 (0.0%) #DIV/0!NNE = NO BUSINESS LINE CODE (added in 2015); n (%) 0 (0.0%) #DIV/0! #VALUE! 0 (0.0%) 0 (0.0%) #DIV/0!NNK = UNKNOWN (added in 2015); n (%) 0 (0.0%) #DIV/0! #VALUE! 0 (0.0%) 0 (0.0%) #DIV/0!NNK = UNKNOWN (added in 2015); n (%) 0 (0.0%) #DIV/0! #VALUE! 0 (0.0%) 0 (0.0%) #DIV/0! | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of link (prothrombin) tests orderedmean (sd) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Treating prescriber - Other; n (%) Treating prescriber - Bio days, Vmean (sd) Use of Prasugrel; n (%) Use of Prasugrel; n (%) Use of Prasugrel; n (%) Use of CLOOP Diuretics-other diuretics-other hypertension drugs; n (%) Commercial vs Medicare Advantage-Business Type Code - CORRECT ONE - OPTUMCommercial; n (%)Medicare Advantage; n (%) Commercial vs Medicare Advantage-Business Type Code | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 1,(1%) 12 (1 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 10.73 (1.63) 2,275 (0.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) 1,136 (15.3%) 2,640 (35.6%) 4,773 (64.4%) | 707 (17.9%) 330 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) 2.57 (1.68) ** (0.1%) 532 (13.5%) | 0.15 #DIV/01 -0.02 0.00 0.00 0.04 -0.02 0.01 0.01 0.01 0.04 0.15 -0.04 0.19 0.00 -0.02 0.66 0.03 0.05 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) 1,808 (12.9%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 72 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) 427 (10.9%) | 0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.06 -0.09 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 16,705 (99.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 0.59 #DIV/01 0.09 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUEI 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) #WALUEI 0.59 (1.17) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #WALUEI | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #/ALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #/ALUEI 0.54 (0.82) 8064 (27.8%) 2243 (9.1%) 2243 (9.1%) 3.29 (1.79) #/ALUEI 4253 (17.3%) | -0.15 -0.04 -0.01 #WALUE! #VALUE! #VALUE! 0.02 0.00 0.02 0.00 #VALUE! 0.00 0.03 -0.07 -0.02 0.01 #VALUE! |
| NONE = NO BUSINESS LINE CODE (added in 2015); n (%) 0 (0.0%) #DIV/0! #VALUE! 0 (0.0%) 0 (0.0%) #DIV/0!UNK = UNKNOWN (added in 2015); n (%) 0 (0.0%) #DIV/0! #VALUE! 0 (0.0%) 0 (0.0%) #DIV/0! | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGF inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin k therapy; n (%) Number of lNR (prothrombin) tests orderedmean (sd) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DSZ VASC score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diuretics+other diuretics+other hypertension drugs; n (%) Commercial s Medicare Advantage-Business Type Code - CORRECT ONE - OPTUMCommercial; n (%) Commercial; n (%) Commercial vs Medicare Advantage-Business Type CodeCOM = COMMERCIAL; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 21 (0.3%) 22 (1 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) 1,136 (15.3%) 2,640 (35.6%) | 707 (17.9%) 310 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) 2.57 (1.68) ** (0.1%) 532 (13.5%) | 0.15 #DIV/01 -0.02 0.00 0.00 0.04 -0.02 0.01 0.01 0.04 0.15 -0.04 0.15 -0.04 0.19 0.00 -0.02 0.66 0.03 0.05 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) 1,808 (12.9%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 72 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) 427 (10.9%) | 0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.06 -0.09 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 45 (0.3%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) 3,294 (19.7%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 0.59 #DIV/01 0.09 | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUEI 269 (0.5%) 869 (1.6%) 0.48 (0.78) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) 2966 (5.5%) 2966 (5.5%) 476 (1.7) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #WALUEI 10589 (19.6%) 6,638 (31.0%) 14,752 (69.0%) 2,640 (35.6%) | 4588 (18.7%) 2,046 (52.4%) 161 (0.7%) #VALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (22.8%) 12128 (45.6%) 2243 (9.1%) 2243 (9.1%) 2243 (9.1%) 3.29 (1.79) #VALUEI 4253 (17.3%) | -0.15 -0.04 -0.01 #VALUE! #VALUE! 0.02 0.00 0.02 0.00 #VALUE! 0.00 0.00 #VALUE! 0.00 0.01 #VALUE! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. |
| (%) 0 (0.0%) 0 (0.0%) #DIV/0! #VALUE! 0 (0.0%) 0 (0.0%) #DIV/0! + #VALUE! 0 (0.0%) 0 (0.0%) #DIV/0! + #VALUE! 0 (0.0%) 0 (0.0%) #DIV/0! | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of link (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Prasugrel; n (%) Use of Prasugrel; n (%) Commercial vs Medicare Advantage- Business Type Code - CORRECT ONE - OPTUMCommercial; n (%)McGleare AdVantage; n (%) Commercial vs Medicare Advantage- Business Type CodeCOM = COMMERCIAL; n (%)MCR = MEDICARE; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 44 (0.6%) 42 (1.03%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 47 (0.1%) 0.73 (1.63) 2,275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) 1,136 (15.3%) 4,773 (64.4%) | 707 (17.9%) 310 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (15.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,918 (99.9%) 295 (7.5%) 2.57 (1.68) ** (0.1%) 532 (13.5%) 1277 (32.4%) 2663 (67.6%) | 0.15 #DIV/01 -0.02 -0.00 -0.00 -0.04 -0.02 -0.01 -0.01 -0.04 -0.15 -0.04 -0.19 -0.02 -0.66 -0.03 -0.05 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) 1,808 (12.9%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 72 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) 427 (10.9%) | 0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.06 -0.09 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) **(0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 1,744 (10.4%) 3.61 (1.83) *** (0.0%) 3,294 (19.7%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 0.59 #DIV/01 0.09 | 7167 (33.3%) 7,040 (50.4%) 350 (0.6%) #VALUEI 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) #VALUEI 0.59 (1.17) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #VALUEI 10589 (19.6%) 6,638 (31.0%) 14,752 (69.0%) 2,640 (35.6%) 4,773 (64.4%) | 2,588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (32.8%) 12128 (45.6%) 24375 (99.1%) 2437 (99.1%) 3.29 (1.79) #VALUEI 4253 (17.3%) 2112 (26.9%) 5736 (73.1%) | -0.15 -0.04 -0.01 #WALUE! 0.02 0.00 0.00 0.00 0.00 #WALUE! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. |
| UNK = UNKNOWN (added in 2015); n (%) 0 (0.0%) 0 (0.0%) #DIV/0! + #VALUE! 0 (0.0%) 0 (0.0%) #DIV/0! | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) PGP inhibitors; n (%) PGP inhibitors; n (%) Other antiplatelet agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin k therapy; n (%) Number of link (prothrombin) tests orderedmean (sd) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diuretics+other diuretics+other hypertension drugs; n (%) Commercial vs Medicare Advantage- Business Type Code - CORRECT ONE - OPTUMCommercial vs Medicare Advantage- Business Type CodeCOM = COMMERCIAL; n (%)Medicare Advantage; n (%) Commercial vs Medicare Advantage- Business Type CodeCOM = COMMERCIAL; n (%)MCR = MEDICARE; n (%)MCR = MEDICARE; n (%) | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 1,1(-1%) 12 (1 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 100 (1.3%) 0.73 (1.63) 2,275 (80.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) 1,136 (15.3%) 4,773 (64.4%) 4,773 (64.4%) 4,773 (64.4%) 0 (0.05%) | 707 (17.9%) 310 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (15.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,918 (99.9%) 295 (7.5%) 2.57 (1.68) ** (0.1%) 532 (13.5%) 1277 (32.4%) 2663 (67.6%) | 0.15 #DIV/01 -0.02 -0.00 -0.00 -0.04 -0.02 -0.01 -0.01 -0.04 -0.15 -0.04 -0.19 -0.02 -0.66 -0.03 -0.05 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) 1,808 (12.9%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 72 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) 427 (10.9%) | 0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.06 -0.09 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) **(0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 1,744 (10.4%) 3.61 (1.83) *** (0.0%) 3,294 (19.7%) | -0.14 #DIV/01 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 0.59 #DIV/01 0.09 | 7167 (33.3%) 7,040 (50.4%) 350 (0.6%) #VALUEI 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) #VALUEI 0.59 (1.17) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #VALUEI 10589 (19.6%) 6,638 (31.0%) 14,752 (69.0%) 2,640 (35.6%) 4,773 (64.4%) | 2,588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #VALUEI 0.54 (0.82) 8064 (32.8%) 12128 (45.6%) 24375 (99.1%) 2437 (99.1%) 3.29 (1.79) #VALUEI 4253 (17.3%) 2112 (26.9%) 5736 (73.1%) | -0.15 -0.04 -0.01 #WALUE! 0.02 0.00 0.00 0.00 0.00 #WALUE! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. |
| *************************************** | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin K therapy; n (%) Number of liN( prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASC score, 180 days, Vmean (sd) Use of VASC score, 180 days, Vmean (sd) Use of Loop Diurettics+other diuretics+other hypertension drugs; n (%) Commercial vs Medicare Advantage- Business Type Code - CORRECT ONE - OPTUMCommercial ys Medicare Advantage- Business Type CodeMedicare Advantage; n (%) Commercial vs Medicare Advantage- Business Type CodeCOM = COMMERCIAL; n (%)MCR = MEDICARE; n (%)MCR = MEDICARE; n (%)MCR = MEDICARE; n (%)MCR = NO BUSINESS LINE CODE (added in 2015); rNONE = NO BUSINESS LINE CODE (added in 2015); rNONE = NO BUSINESS LINE CODE (added in 2015); r | 922 (12.4%) 3,535 (47.7%) 44 (0.6%) 21 (0.3%) 21 (0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 275 (30.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) 1,136 (15.3%) 4,773 (64.4%) 0 (0.0%) | 707 (17.9%) 330 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) 2.57 (1.68) ** (0.1%) 532 (13.5%) 1277 (32.4%) 2,663 (67.6%) 0 (0.0%) | 0.15 0.01 0.02 0.00 0.00 0.04 0.02 0.01 0.01 0.04 0.15 0.04 0.19 0.00 0.02 0.66 0.03 0.05 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) 1,808 (12.9%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 72 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) 427 (10.9%) | 0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.06 -0.09 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 16,705 (99.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) 3,294 (19.7%) | -0.14 #DIV/OI 0.00 0.00 0.00 0.00 0.02 0.02 -0.03 0.04 0.02 #DIV/OI 0.02 0.04 0.05 -0.07 -0.02 0.59 #DIV/OI 0.09 #VALUEI #VALUEI #VALUEI | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUEI 269 (0.5%) 869 (1.6%) 0.48 (0.78) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) 2966 (5.5%) 2966 (5.5%) 4762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #WALUEI 10589 (19.6%) 6,638 (31.0%) 14,752 (69.0%) 2,640 (35.6%) 4,773 (64.4%) 0 (0.0%) | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #VALUEI #VALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) 1359 (5.5%) 1359 (5.5%) 1212 (46.8%) 12128 (45.6%) 22437 (9.1%) 2243 (9.1%) 3.29 (1.79) #VALUEI 4253 (17.3%) 2112 (26.9%) 5736 (73.1%) 1,277 (32.4%) 2,663 (67.6%) 0 (0.0%) | -0.15 -0.04 -0.01 #WALUE! 0.02 0.00 0.00 0.00 0.00 #WALUE! 0.00 0.00 0.00 0.00 0.00 0.00 0.00 0. |
| cummerual vs meurcale Auvantager usua type | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGP inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) Proton pump inhibitor; n (%) Vitamin K therapy; n (%) Number of link (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Other; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASc score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Prasugrel; n (%) Use of Prasugrel; n (%) Commercial vs Medicare Advantage-Business Type Code - CORRECT ONE - OPTUMCommercial; n (%)MCD = MEDICANE; n (%)MCNE = NO BUSINESS LINE CODE (added in 2015); r (%) | 922 (12.4%) 3,535 (47.7%) 1,(4.0.6%) 14 (0.6%) 12 (1.0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 10.1%) 0.73 (1.63) 2,275 (0.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) 1,136 (15.3%) 2,640 (35.6%) 4,773 (64.4%) 0 (0.0%) | 707 (17.9%) 330 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) 2.57 (1.68) ** (0.1%) 532 (13.5%) 1277 (32.4%) 2663 (67.6%) 0 (0.0%) | 0.15 #DIV/01 -0.02 -0.00 -0.00 -0.04 -0.02 -0.01 -0.01 -0.01 -0.04 -0.15 -0.04 -0.15 -0.04 -0.15 -0.07 -0.07 #DIV/01 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) 1,808 (12.9%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 72 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) 427 (10.9%) | 0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.06 -0.09 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 16,705 (99.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) 3,294 (19.7%) | -0.14 #DIV/01 0.00 0.00 0.00 0.02 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 0.59 #DIV/01 0.09 #VALUEI #VALUEI #VALUEI | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) #WALUE! 0.59 (1.17) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #WALUE! 10589 (19.6%) 6,638 (31.0%) 14,752 (69.0%) 2,640 (35.6%) 4,773 (64.4%) 0 (0.0%) | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #WALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #WALUEI 0.54 (0.82) 8064 (22.8%) 24375 (99.1%) 2243 (9.1%) 3.29 (1.79) #WALUEI 4253 (17.3%) 2112 (26.9%) 5736 (73.1%) 1,277 (32.4%) 0 (0.0%) 0 (0.0%) | -0.15 -0.04 -0.01 #VALUE! #VALUE! #VALUE! 0.02 0.00 0.02 0.00 #VALUE! 0.00 0.03 -0.07 -0.02 0.06 0.09 -0.09 -0.09 -0.09 #DIV/0! |
| | Prior cancer; n (%) Antibiotics; n (%) Aspirin; n (%) Aspirin; n (%) Aspirin; n (%) Other antiplatelet agents; n (%) PGF inhibitors; n (%) Other gastroprotective agents; n (%) Number of lipid tests orderedmean (sd) Proton pump inhibitor; n (%) H2 receptor antagonist; n (%) Vitamin k therapy; n (%) Number of liNR (prothrombin) tests orderedmean (sd) Treating prescriber - Cardiologist; n (%) Treating prescriber - Primary Care Physician; n (%) Treating prescriber - Other; n (%) Alpha blockers; n (%) CHA2DS2 VASC score, 180 days, Vmean (sd) Use of Prasugrel; n (%) Use of Loop Diuretics-other diuretics-other hypertension drugs; n (%) Commercial vs Medicare Advantage-Business Type Code - CORRECT ONE - OPTUMCommercial; n (%)Medicare Advantage (%) Commercial vs Medicare Advantage-Business Type CodeCOM = COMMERCIAL; n (%)MCR = MEDICARE; n (%)MCR = MEDICARE; n (%)MCD = MEDICARD; n (%)MODE = NO BUSINESS LINE CODE (added in 2015); n (%)UNK = UNKNOWN (added in 2015); n (%) | 922 (12.4%) 3,535 (47.7%) 1,(4.0.6%) 14 (0.6%) 12 (1.0.3%) 1,375 (18.5%) 100 (1.3%) 0.49 (0.77) 1,695 (22.9%) 312 (4.2%) 10.1%) 0.73 (1.63) 2,275 (0.7%) 6,535 (88.2%) 7,407 (99.9%) 527 (7.1%) 3.72 (1.81) 13 (0.2%) 1,136 (15.3%) 2,640 (35.6%) 4,773 (64.4%) 0 (0.0%) | 707 (17.9%) 330 (49.0%) 31 (0.8%) ** (0.1%) ** (0.3%) 667 (16.9%) 58 (1.5%) 0.48 (0.78) 892 (22.6%) 174 (4.4%) ** (0.0%) 0.53 (0.88) 1,282 (32.5%) 3,215 (81.6%) 3,938 (99.9%) 295 (7.5%) 2.57 (1.68) ** (0.1%) 532 (13.5%) 1277 (32.4%) 2663 (67.6%) 0 (0.0%) | 0.15 #DIV/01 -0.02 -0.00 -0.00 -0.04 -0.02 -0.01 -0.01 -0.01 -0.04 -0.15 -0.04 -0.15 -0.04 -0.15 -0.07 -0.07 #DIV/01 | 1,383 (9.9%) 7,040 (50.4%) 160 (1.1%) 22 (0.2%) 67 (0.5%) 2,756 (19.7%) 215 (1.5%) 0.34 (0.75) 3,099 (22.2%) 497 (3.6%) 22 (0.2%) 0.53 (1.22) 4,338 (31.0%) 5,771 (41.3%) 13,310 (95.2%) 872 (6.2%) 3.50 (1.56) 27 (0.2%) 1,808 (12.9%) | 519 (13.3%) 2,046 (52.4%) 63 (1.6%) ** (0.1%) ** (0.1%) 72 (18.4%) 78 (2.0%) 0.36 (0.85) 825 (21.1%) 175 (4.5%) 0 (0.0%) 0.46 (0.98) 1,372 (35.1%) 1,695 (43.4%) 3,732 (95.5%) 204 (5.2%) 2.64 (1.73) ** (0.3%) 427 (10.9%) | 0.11 #DIV/01 -0.04 -0.03 -0.03 -0.04 -0.02 -0.03 -0.06 -0.09 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 -0.01 -0.04 | 4,862 (14.9%) 17,449 (53.5%) 146 (0.4%) 113 (0.3%) 181 (0.6%) 554 (1.7%) 0.54 (0.79) 10,056 (30.8%) 2,157 (6.5%) ** (0.0%) 0.58 (1.01) 11,149 (34.2%) 13,113 (40.2%) 3,226 (9.9%) 4.65 (1.70) ** (0.0%) | 3,362 (20.1%) 9,034 (53.9%) 67 (0.4%) 45 (0.3%) 100 (0.6%) 3,737 (22.3%) 258 (1.5%) 0.56 (0.80) 4,868 (29.1%) 1,010 (6.0%) ** (0.0%) 0.56 (0.77) 5,410 (32.3%) 6,308 (37.7%) 16,705 (99.7%) 1,744 (10.4%) 3.61 (1.83) ** (0.0%) 3,294 (19.7%) | -0.14 #DIV/01 0.00 0.00 0.00 0.02 0.02 0.02 -0.03 0.04 0.02 #DIV/01 0.02 0.04 0.05 -0.07 -0.02 0.59 #DIV/01 0.09 #VALUEI #VALUEI #VALUEI | 7167 (13.3%) 7,040 (50.4%) 350 (0.6%) #WALUE! 269 (0.5%) 11632 (21.5%) 869 (1.6%) 0.48 (0.78) 14850 (27.5%) 2966 (5.5%) #WALUE! 0.59 (1.17) 17762 (32.9%) 25419 (47.1%) 53078 (98.3%) 4625 (8.6%) 4.22 (1.68) #WALUE! 10589 (19.6%) 6,638 (31.0%) 14,752 (69.0%) 2,640 (35.6%) 4,773 (64.4%) 0 (0.0%) | 4588 (18.7%) 2,046 (52.4%) 2,046 (52.4%) 161 (0.7%) #WALUEI 5124 (20.8%) 394 (1.6%) 0.52 (0.81) 6585 (26.8%) 1359 (5.5%) #WALUEI 0.54 (0.82) 8064 (22.8%) 24375 (99.1%) 2243 (9.1%) 3.29 (1.79) #WALUEI 4253 (17.3%) 2112 (26.9%) 5736 (73.1%) 1,277 (32.4%) 0 (0.0%) 0 (0.0%) | -0.15 -0.04 -0.01 #VALUE! #VALUE! #VALUE! 0.02 0.00 0.02 0.00 #VALUE! 0.00 0.03 -0.07 -0.02 0.06 0.09 -0.09 -0.09 -0.09 #DIV/0! |

| 1 - Fee For Service; n (%) | - | - | 8,838 (63.2%) | 2,764 (70.7%) | -0.16 | - | - | 8,838 (63.2%) | 2,764 (70.7%) | -0.16 |
|---|---|---|---|---|---|---|---|---|---|---|
| 2 - Encounter; n (%) | - | | 1,141 (8.2%) | 309 (7.9%) | 0.01 | - | - | 1,141 (8.2%) | 309 (7.9%) | 0.01 |
| 3 - Medicare; n (%) | - | - | 3,608 (25.8%) | 750 (19.2%) | 0.16 | - | - | 3,608 (25.8%) | 750 (19.2%) | 0.16 |
| 4 - Medicare Encounter; n (%) | - | - | 390 (2.8%) | 85 (2.2%) | 0.04 | - | - | 390 (2.8%) | 85 (2.2%) | 0.04 |
| Metropolitan Statistical Area - Urban (any MSA) vs | | | | | | | | | | |
| Rural (non-MSA) | | | | | | | | 0 | 0 | 0.00 |
| Urban; n (%) | - | - | 11,109 (79.5%) | 2,903 (74.3%) | 0.12 | - | - | 11,109 (79.5%) | 2,903 (74.3%) | 0.12 |
| Rural; n (%) | - | - | 151 (1.1%) | 145 (3.7%) | -0.17 | - | - | 151 (1.1%) | 145 (3.7%) | -0.17 |
| Unknown/Missing; n (%) | - | | 2,717 (19.4%) | 860 (22.0%) | -0.06 | - | - | 2,717 (19.4%) | 860 (22.0%) | -0.06 |

Due to CMS cell suppression policy, all values less than 11 are denoted with \*\*

| | | | | | PS-matched | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Optum | | MarketScan | | | | Medicare | <u> </u> | | | POOLED | |
| Wasiahia. | Defenses mederic Comments | (1 F 20 ) C | CA DISE DAG | | (15 30) C | C+ D:# D | -f | - (15 20) C | C+ D:# D-4 | | Exposure - rivaroxaban | C+ D:4 |
| Variable<br>Number of patients | Reference-warfarin Copy oxaba<br>1,575 | an (15 or 20 mg) Copy<br>1,575 | St. Diff. Kete | erence- warfarin Copy 'oxaba<br>2,899 | | St. Diff. Ki | eference- warfarin Copy 'oxaba<br>8,511 | n (15 or 20 mg) Copy<br>8,511 | St. Diff. Ken | erence-warfarin Copy<br>12,985 | (15 or 20 mg) Copy<br>12,985 | St. Dif |
| Age | 1,5/5 | 1,575 | | 2,899 | 2,899 | | 8,511 | 8,511 | | 12,985 | 12,985 | |
| mean (sd) | 65.29 (15.26) | 65.87 (14.42) | -0.04 | 55.03 (16.16) | 55.22 (15.70) | -0.01 | 76.35 (7.86) | 76.58 (7.93) | -0.03 | 70.25 (11.27) | 70.51 (11.02) | -0.03 |
| Age categories without zero category | 03.29 (13.20) | 03.87 (14.42) | -0.04 | 33.03 (10.10) | 33.22 (13.70) | -0.01 | 70.33 (7.60) | 70.36 (7.33) | -0.03 | 70.23 (11.27) | 70.31 (11.02) | -0.0 |
| 18 - 54; n (%) | 373 (23.7%) | 319 (20.3%) | 0.08 | 1.394 (48.1%) | 1.388 (47.9%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1767 (13.6%) | 1707 (13.1%) | 0.0 |
| 55 - 64; n (%) | 269 (17.1%) | 268 (17.0%) | 0.00 | 821 (28.3%) | 827 (28.5%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1,090 (8.4%) | 1,095 (8.4%) | 0.0 |
| 65 - 74: n (%) | 424 (26.9%) | 512 (32.5%) | -0.12 | 313 (10.8%) | 338 (11.7%) | -0.03 | 4.015 (47.2%) | 3.893 (45.7%) | 0.03 | 4.752 (36.6%) | 4.743 (36.5%) | 0.0 |
| >=75; n (%) | 509 (32.3%) | 476 (30.2%) | 0.05 | 371 (12.8%) | 346 (11.9%) | 0.03 | 4,496 (52.8%) | 4,618 (54.3%) | -0.03 | 5,376 (41.4%) | 5,440 (41.9%) | -0.0 |
| Gender without zero category- United | 309 (32.3%) | 470 (30.2%) | 0.03 | 3/1 (12.0%) | 340 (11.5%) | 0.03 | 4,450 (32.6%) | 4,010 (34.3%) | -0.03 | 3,370 (41.4%) | 3,440 (41.5%) | -0.0 |
| Males; n (%) | 718 (45.6%) | 703 (44.6%) | 0.02 | 1,383 (47.7%) | 1.412 (48.7%) | -0.02 | 3.166 (37.2%) | 3.136 (36.8%) | 0.01 | 5,267 (40.6%) | 5.251 (40.4%) | 0.0 |
| Females: n (%) | 857 (54.4%) | 872 (55.4%) | -0.02 | 1,516 (52.3%) | 1,487 (51.3%) | 0.02 | 5,345 (62.8%) | 5,375 (63.2%) | -0.01 | 7,718 (59.4%) | 7,734 (59.6%) | 0.0 |
| Race | 637 (34.4%) | 672 (33.4%) | -0.02 | 1,310 (32.376) | 1,467 (31.370) | 0.02 | 3,343 (02.670) | 3,373 (03.2%) | -0.01 | 7,710 (35.470) | 7,734 (35.0%) | 0.0 |
| White; n (%) | | | | | | | 7,144 (83.9%) | 7,136 (83.8%) | | 7,144 (83.9%) | 7,136 (83.8%) | 0.0 |
| Black; n (%) | | | | | | | 932 (11.0%) | 947 (11.1%) | | 932 (11.0%) | 947 (11.1%) | 0.0 |
| Asian: n (%) | | | | | | | 81 (1.0%) | 77 (0.9%) | | 81 (1.0%) | 77 (0.9%) | 0.0 |
| Hispanic: n (%) | | | | | | | 188 (2.2%) | 192 (2.3%) | | 188 (2.2%) | 192 (2.3%) | 0.0 |
| North American Native: n (%) | | | | | | | 33 (0.4%) | 31 (0.4%) | | 33 (0.4%) | 31 (0.4%) | 0.0 |
| Other/Unknown; n (%) | | | | | | | 133 (1.6%) | 128 (1.5%) | | 133 (1.6%) | 128 (1.5%) | 0.0 |
| Region without zero category- United v3 (lumping | | | | | | | 133 (1.070) | 120 (1.3/0) | | 133 (1.0%) | 120 (1.3%) | 0.0 |
| missing&other category with West) | | | | | | | | | | | | |
| Northeast; n (%) | 182 (11.6%) | 189 (12.0%) | -0.01 | 490 (16.9%) | 522 (18.0%) | -0.03 | 1,623 (19.1%) | 1,606 (18.9%) | 0.01 | 2,295 (17.7%) | 2,317 (17.8%) | 0.0 |
| South; n (%) | 662 (42.0%) | 664 (42.2%) | 0.00 | 808 (27.9%) | 829 (28.6%) | -0.02 | 3,508 (41.2%) | 3,470 (40.8%) | 0.01 | 4,978 (38.3%) | 4,963 (38.2%) | 0.0 |
| Midwest; n (%) | 391 (24.8%) | 383 (24.3%) | 0.01 | 1,249 (43.1%) | 1,191 (41.1%) | 0.04 | 2,049 (24.1%) | 2,086 (24.5%) | -0.01 | 3,689 (28.4%) | 3,660 (28.2%) | 0.0 |
| West; n (%) | 340 (21.6%) | 339 (21.5%) | 0.00 | 309 (10.7%) | 320 (11.0%) | -0.01 | 1,331 (15.6%) | 1,349 (15.9%) | -0.01 | 1,980 (15.2%) | 2,008 (15.5%) | -0.0 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 43 (1.5%) | 37 (1.3%) | 0.02 | N/A | N/A | #VALUE! | 43 (1.5%) | 37 (1.3%) | 0.0 |
| CV Covariates | | | | | | | | | | | | |
| Ischemic heart disease; n (%) | 225 (14.3%) | 234 (14.9%) | -0.02 | 309 (10.7%) | 296 (10.2%) | 0.02 | 1,805 (21.2%) | 1,799 (21.1%) | 0.00 | 2,339 (18.0%) | 2,329 (17.9%) | 0.0 |
| Acute MI; n (%) | 15 (1.0%) | 19 (1.2%) | -0.02 | 51 (1.8%) | 41 (1.4%) | 0.03 | 129 (1.5%) | 123 (1.4%) | 0.01 | 195 (1.5%) | 183 (1.4%) | 0.0 |
| ACS/unstable angina; n (%) | ** (0.6%) | ** (0.6%) | 0.00 | ** (0.2%) | ** (0.3%) | -0.02 | 55 (0.6%) | 55 (0.6%) | 0.00 | #VALUE! | #VALUE! | #VALUE |
| Old MI; n (%) | 48 (3.0%) | 42 (2.7%) | 0.02 | 44 (1.5%) | 38 (1.3%) | 0.02 | 402 (4.7%) | 389 (4.6%) | 0.00 | 494 (3.8%) | 469 (3.6%) | 0.0 |
| Stable angina; n (%) | 28 (1.8%) | 34 (2.2%) | -0.03 | 46 (1.6%) | 39 (1.3%) | 0.03 | 155 (1.8%) | 162 (1.9%) | -0.01 | 229 (1.8%) | 235 (1.8%) | 0.0 |
| Coronary atherosclerosis and other forms of chronic | | 34 (E.E/o) | 0.03 | 40 (2.070) | 33 (1.370) | 0.05 | 155 (1.5%) | 102 (1.570) | 0.01 | 223 (2.070) | 255 (2.570) | 0.0 |
| ischemic heart disease; n (%) | 196 (12.4%) | 204 (13.0%) | -0.02 | 256 (8.8%) | 242 (8.3%) | 0.02 | 1.624 (19.1%) | 1.620 (19.0%) | 0.00 | 2.076 (16.0%) | 2.066 (15.9%) | 0.0 |
| Other atherosclerosis with ICD10 v2 Copy; n (%) | 16 (1.0%) | 17 (1.1%) | -0.01 | 31 (1.1%) | 15 (0.5%) | 0.07 | 124 (1.5%) | 84 (1.0%) | 0.05 | 171 (1.3%) | 116 (0.9%) | 0.04 |
| Previous cardiac procedure (CABG or PTCA or Stent) | == (=:=:=, | () | | () | () | | (, | - () | | | () | |
| v4: n (%) | ** (0.5%) | ** (0.3%) | 0.03 | 17 (0.6%) | 12 (0.4%) | 0.03 | 54 (0.6%) | 35 (0.4%) | 0.03 | #VALUE! | #VALUE! | #VALUE |
| History of CABG or PTCA; n (%) | 56 (3.6%) | 74 (4.7%) | -0.06 | 42 (1.4%) | 43 (1.5%) | -0.01 | 618 (7.3%) | 639 (7.5%) | -0.01 | 716 (5.5%) | 756 (5.8%) | -0.0 |
| Any stroke; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 000 (0.0%) | #DIV/0 |
| Ischemic stroke (w and w/o mention of cerebral | 2 (2.2.2) | - () | | - () | - () | | - (, | - () | | - () | () | |
| infarction); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 000 (0.0%) | #DIV/0 |
| Hemorrhagic stroke; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 0 (0.0%) | #DIV/0 |
| TIA: n (%) | 12 (0.8%) | 15 (1.0%) | -0.02 | 28 (1.0%) | 25 (0.9%) | 0.01 | 95 (1.1%) | 103 (1.2%) | -0.01 | 135 (1.0%) | 143 (1.1%) | -0.0 |
| Other cerebrovascular disease: n (%) | 22 (1.4%) | 29 (1.8%) | -0.03 | 23 (0.8%) | 29 (1.0%) | -0.02 | 178 (2.1%) | 183 (2.2%) | -0.01 | 223 (1.7%) | 241 (1.9%) | -0.0 |
| Cerebrovascular procedure; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 000 (0.0%) | 0 (0.0%) | #DIV/0 |
| Heart failure (CHF); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | ** (0.1%) | ** (0.0%) | 0.04 | <11 (0.0%) | <11 (0.0%) | #DIV/0! | #VALUE! | #VALUE! | #VALUE |
| Peripheral Vascular Disease (PVD) or PVD Surgery v2; | 2 (2.2.2) | - () | | (4-2) | (/ | | (0.01.) | () | | | | |
| n (%) | 183 (11.6%) | 189 (12.0%) | -0.01 | 329 (11.3%) | 325 (11.2%) | 0.00 | 1,107 (13.0%) | 1,097 (12.9%) | 0.00 | 1,619 (12.5%) | 1,611 (12.4%) | 0.00 |
| Atrial fibrillation; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 000 (0.0%) | #DIV/0 |
| Other cardiac dysrhythmia; n (%) | 174 (11.0%) | 182 (11.6%) | -0.02 | 305 (10.5%) | 296 (10.2%) | 0.01 | 1.118 (13.1%) | 1.099 (12.9%) | 0.01 | 1.597 (12.3%) | 1.577 (12.1%) | 0.0 |
| Cardiac conduction disorders: n (%) | 64 (4.1%) | 64 (4.1%) | 0.00 | 86 (3.0%) | 87 (3.0%) | 0.00 | 466 (5.5%) | 523 (6.1%) | -0.03 | 616 (4.7%) | 674 (5.2%) | -0.0 |
| Other CVD: n (%) | 272 (17.3%) | 261 (16.6%) | 0.02 | 430 (14.8%) | 454 (15.7%) | -0.03 | 1,402 (16.5%) | 1,367 (16.1%) | 0.01 | 2,104 (16.2%) | 2,082 (16.0%) | 0.0 |
| Diabetes-related complications | | (10.070) | 0.02 | .== (24.070) | (25., 70) | 0.03 | -, (20.5/0) | -, (10.1/0) | 3.01 | _,(10.2/0) | _,552 (25.570) | 0.0 |
| Occurrence of Diabetic Neuropathy v2 Copy; n (%) | 104 (6.6%) | 117 (7.4%) | -0.03 | 95 (3.3%) | 88 (3.0%) | 0.02 | 474 (5.6%) | 451 (5.3%) | 0.01 | 673 (5.2%) | 656 (5.1%) | 0.0 |
| Occurrence of diabetic nephropathy V2 copy, II (20) | 104 (0.0%) | 117 (7.470) | -0.03 | 33 (3.370) | 00 (3.0%) | 0.02 | 474 (5.6%) | 451 (5.570) | 0.01 | 073 (3.270) | 030 (3.170) | 0.0 |
| Copy; n (%) | 54 (3.4%) | 64 (4.1%) | -0.04 | 45 (1.6%) | 44 (1.5%) | 0.01 | 249 (2.9%) | 217 (2.5%) | 0.02 | 348 (2.7%) | 325 (2.5%) | 0.0 |
| Hypoglycemia v2; n (%) | 20 (1.3%) | 26 (1.7%) | -0.03 | 33 (1.1%) | 31 (1.1%) | 0.00 | 241 (2.8%) | 216 (2.5%) | 0.02 | 294 (2.3%) | 273 (2.1%) | 0.0 |
| Hyperglycemia: n (%) | 103 (6.5%) | 101 (6.4%) | 0.00 | 137 (4.7%) | 134 (4.6%) | 0.00 | 644 (7.6%) | 648 (7.6%) | 0.02 | 884 (6.8%) | 883 (6.8%) | 0.0 |
| Diabetic ketoacidosis: n (%) | 13 (0.8%) | ** (0.4%) | 0.05 | ** (0.4%) | 15 (0.5%) | -0.01 | 28 (0.3%) | 29 (0.3%) | 0.00 | #VALUE! | #VALUE! | #VALUE |
| Hypertension: 1 inpatient or 2 outpatient claims | 13 (0.8%) | ·· (U.476) | 0.05 | · (U.476) | ±3 (U.3%) | -0.01 | 28 (U.3%) | 29 (U.5%) | 0.00 | #VALUE! | #VALUE! | #VALUE |
| within 365 days; n (%) | 1,009 (64.1%) | 1.044 (66.3%) | -0.05 | 1.471 (50.7%) | 1.490 (51.4%) | -0.01 | 6.804 (79.9%) | 6.845 (80.4%) | -0.01 | 9.284 (71.5%) | 9.379 (72.2%) | -0.0 |
| Hyperlipidemia v2; n (%) | 725 (46.0%) | 766 (48.6%) | -0.05 | 952 (32.8%) | 964 (33.3%) | -0.01 | 4,628 (54.4%) | 4,625 (54.3%) | 0.00 | 6,305 (48.6%) | 6,355 (48.9%) | -0.0 |
| Edema; n (%) | 491 (31.2%) | 509 (32.3%) | -0.03 | 701 (24.2%) | 707 (24.4%) | 0.00 | 2,208 (25.9%) | 2,213 (26.0%) | 0.00 | 3400 (26.2%) | 3429 (26.4%) | 0.0 |
| Renal Dysfunction (non-diabetic) v2; n (%) | 491 (31.2%)<br>363 (23.0%) | 378 (24.0%) | -0.02<br>-0.02 | 701 (24.2%)<br>452 (15.6%) | 707 (24.4%)<br>470 (16.2%) | -0.02 | 2,208 (25.9%) 2,153 (25.3%) | 2,213 (26.0%) | -0.02 | 2968 (22.9%) | 3429 (26.4%) | -0.0 |
| | 363 (23.0%)<br>176 (11.2%) | 378 (24.0%)<br>185 (11.7%) | -0.02<br>-0.02 | 452 (15.6%)<br>229 (7.9%) | 470 (16.2%)<br>254 (8.8%) | -0.02 | 2,153 (25.3%)<br>1.009 (11.9%) | | -0.02<br>-0.01 | 2968 (22.9%)<br>1414 (10.9%) | 3078 (23.7%)<br>1467 (11.3%) | -0.0 |
| Occurrence of acute renal disease v2; n (%) | | | | | | | | 1,028 (12.1%) | | | | |
| Occurrence of chronic renal insufficiency; n (%) | 200 (12.7%) | 209 (13.3%) | -0.02 | 160 (5.5%) | 167 (5.8%) | -0.01 | 1,274 (15.0%) | 1,293 (15.2%) | -0.01 | 1634 (12.6%) | 1669 (12.9%) | -0.0 |
| Chronic kidney disease v2; n (%) | 193 (12.3%) | 199 (12.6%) | -0.01 | 150 (5.2%) | 148 (5.1%) | 0.00 | 1,205 (14.2%) | 1,224 (14.4%) | -0.01 | 1548 (11.9%) | 1571 (12.1%) | -0.0 |
| CKD Stage 3-4; n (%) | 117 (7.4%) | 132 (8.4%) | -0.04 | 73 (2.5%) | 79 (2.7%) | -0.01 | 724 (8.5%) | 715 (8.4%) | 0.00 | 914 (7.0%) | 926 (7.1%) | 0.0 |
| Occurrence of hypertensive nephropathy; n (%) | 117 (7.4%) | 129 (8.2%) | -0.03 | 67 (2.3%) | 73 (2.5%) | -0.01 | 922 (10.8%) | 937 (11.0%) | -0.01 | 1106 (8.5%) | 1139 (8.8%) | -0.0 |
| Occurrence of miscellaneous renal insufficiency v2; | | | | | | | | | | | | |
| (%) | 123 (7.8%) | 133 (8.4%) | -0.02 | 195 (6.7%) | 199 (6.9%) | -0.01 | 765 (9.0%) | 733 (8.6%) | 0.01 | 1083 (8.3%) | 1065 (8.2%) | 0.0 |
| Other Covariates | | | | | | | | | | | | |
| Liver disease; n (%) Osteoarthritis; n (%) | 0 (0.0%)<br>506 (32.1%) | 0 (0.0%)<br>515 (32.7%) | #DIV/0!<br>-0.01 | 0 (0.0%)<br>656 (22.6%) | 0 (0.0%)<br>651 (22.5%) | #DIV/0!<br>0.00 | 0 (0.0%)<br>3.140 (36.9%) | 0 (0.0%)<br>3,181 (37.4%) | #DIV/0!<br>-0.01 | 0 (0.0%)<br>4302 (33.1%) | 0 (0.0%)<br>4347 (33.5%) | #DIV/0<br>-0.01 |

| Other arthritis, arthropathies and musculoskeletal | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| pain: n (%) | 1,330 (84.4%) | 1,329 (84.4%) | 0.00 | 2,280 (78.6%) | 2,265 (78.1%) | 0.01 | 6,544 (76.9%) | 6,553 (77.0%) | 0.00 | 10154 (78.2%) | 10147 (78.1%) | 0.00 |
| Dorsopathies; n (%) | 563 (35.7%) | 552 (35.0%) | 0.01 | 948 (32.7%) | 909 (31.4%) | 0.03 | 2,792 (32.8%) | 2,816 (33.1%) | -0.01 | 4303 (33.1%) | 4277 (32.9%) | 0.00 |
| Fractures; n (%) | 200 (12.7%) | 197 (12.5%) | 0.01 | 321 (11.1%) | 299 (10.3%) | 0.03 | 1,177 (13.8%) | 1,110 (13.0%) | 0.02 | 1698 (13.1%) | 1606 (12.4%) | 0.02 |
| | | | -0.01 | | | | | | | | | 0.02 |
| Falls v2; n (%) | 178 (11.3%) | 184 (11.7%) | | 106 (3.7%) | 104 (3.6%) | 0.01 | 427 (5.0%) | 439 (5.2%) | -0.01 | 711 (5.5%) | 727 (5.6%) | |
| Osteoporosis; n (%) | 148 (9.4%) | 154 (9.8%) | -0.01 | 120 (4.1%) | 119 (4.1%) | 0.00 | 1,301 (15.3%) | 1,287 (15.1%) | 0.01 | 1569 (12.1%) | 1560 (12.0%) | 0.00 |
| Depression; n (%) | 296 (18.8%) | 315 (20.0%) | -0.03 | 417 (14.4%) | 407 (14.0%) | 0.01 | 1,407 (16.5%) | 1,395 (16.4%) | 0.00 | 2120 (16.3%) | 2117 (16.3%) | 0.00 |
| Anxiety; n (%) | 278 (17.7%) | 285 (18.1%) | -0.01 | 412 (14.2%) | 398 (13.7%) | 0.01 | 1,230 (14.5%) | 1,230 (14.5%) | 0.00 | 1920 (14.8%) | 1913 (14.7%) | 0.00 |
| Sleep_Disorder; n (%) | 137 (8.7%) | 152 (9.7%) | -0.03 | 301 (10.4%) | 293 (10.1%) | 0.01 | 602 (7.1%) | 616 (7.2%) | 0.00 | 1040 (8.0%) | 1061 (8.2%) | -0.01 |
| Dementia; n (%) | 175 (11.1%) | 173 (11.0%) | 0.00 | 142 (4.9%) | 131 (4.5%) | 0.02 | 1,430 (16.8%) | 1,386 (16.3%) | 0.01 | 1747 (13.5%) | 1690 (13.0%) | 0.01 |
| Delirium; n (%) | 70 (4.4%) | 71 (4.5%) | 0.00 | 86 (3.0%) | 86 (3.0%) | 0.00 | 492 (5.8%) | 464 (5.5%) | 0.01 | 648 (5.0%) | 621 (4.8%) | 0.01 |
| Psychosis; n (%) | 51 (3.2%) | 44 (2.8%) | 0.02 | 51 (1.8%) | 50 (1.7%) | 0.01 | 346 (4.1%) | 311 (3.7%) | 0.02 | 448 (3.5%) | 405 (3.1%) | 0.02 |
| Obesity; n (%) | 372 (23.6%) | 383 (24.3%) | -0.02 | 665 (22.9%) | 664 (22.9%) | 0.00 | 1,485 (17.4%) | 1,452 (17.1%) | 0.01 | 2522 (19.4%) | 2499 (19.2%) | 0.01 |
| Overweight; n (%) | 82 (5.2%) | 78 (5.0%) | 0.01 | 84 (2.9%) | 76 (2.6%) | 0.02 | 368 (4.3%) | 383 (4.5%) | -0.01 | 534 (4.1%) | 537 (4.1%) | 0.00 |
| Smoking: n (%) | 464 (29.5%) | 469 (29.8%) | -0.01 | 512 (17.7%) | 522 (18.0%) | -0.01 | 2.580 (30.3%) | 2,587 (30.4%) | 0.00 | 3556 (27.4%) | 3578 (27.6%) | 0.00 |
| Alcohol abuse or dependence; n (%) | 52 (3.3%) | 53 (3.4%) | -0.01 | 61 (2.1%) | 59 (2.0%) | 0.01 | 100 (1.2%) | 86 (1.0%) | 0.02 | 213 (1.6%) | 198 (1.5%) | 0.01 |
| Drug abuse or dependence; n (%) | 68 (4.3%) | 58 (3.7%) | 0.03 | 77 (2.7%) | 78 (2.7%) | 0.00 | 96 (1.1%) | 103 (1.2%) | -0.01 | 241 (1.9%) | 239 (1.8%) | 0.01 |
| COPD; n (%) | 215 (13.7%) | 228 (14.5%) | -0.02 | 237 (8.2%) | 234 (8.1%) | 0.00 | 1,454 (17.1%) | 1,433 (16.8%) | 0.01 | 1906 (14.7%) | 1895 (14.6%) | 0.00 |
| Asthma; n (%) | 156 (9.9%) | 154 (9.8%) | 0.00 | 258 (8.9%) | 262 (9.0%) | 0.00 | 765 (9.0%) | 746 (8.8%) | 0.01 | 1179 (9.1%) | 1162 (8.9%) | 0.01 |
| | | | -0.02 | 274 (9.5%) | | 0.00 | | | 0.01 | | | 0.01 |
| Obstructive sleep apnea; n (%) | 137 (8.7%) | 145 (9.2%) | | | 268 (9.2%) | | 485 (5.7%) | 464 (5.5%) | | 896 (6.9%) | 877 (6.8%) | |
| Pneumonia; n (%) | 133 (8.4%) | 136 (8.6%) | -0.01 | 242 (8.3%) | 232 (8.0%) | 0.01 | 843 (9.9%) | 805 (9.5%) | 0.01 | 1218 (9.4%) | 1173 (9.0%) | 0.01 |
| Other Medications | | | | | | | | | | | | |
| Use of ACE inhibitors; n (%) | 385 (24.4%) | 394 (25.0%) | -0.01 | 559 (19.3%) | 548 (18.9%) | 0.01 | 2,410 (28.3%) | 2,442 (28.7%) | -0.01 | 3354 (25.8%) | 3384 (26.1%) | -0.01 |
| Use of ARBs; n (%) | 215 (13.7%) | 218 (13.8%) | 0.00 | 353 (12.2%) | 369 (12.7%) | -0.02 | 1,572 (18.5%) | 1,589 (18.7%) | -0.01 | 2140 (16.5%) | 2176 (16.8%) | -0.01 |
| Use of Loop Diuretics - United; n (%) | 177 (11.2%) | 174 (11.0%) | 0.01 | 230 (7.9%) | 241 (8.3%) | -0.01 | 1,423 (16.7%) | 1,427 (16.8%) | 0.00 | 1830 (14.1%) | 1842 (14.2%) | 0.00 |
| Use of other diuretics- United; n (%) | 19 (1.2%) | 26 (1.7%) | -0.04 | 47 (1.6%) | 45 (1.6%) | 0.00 | 176 (2.1%) | 170 (2.0%) | 0.01 | 242 (1.9%) | 241 (1.9%) | 0.00 |
| Use of nitrates-United; n (%) | 35 (2.2%) | 38 (2.4%) | -0.01 | 57 (2.0%) | 47 (1.6%) | 0.03 | 382 (4.5%) | 367 (4.3%) | 0.01 | 474 (3.7%) | 452 (3.5%) | 0.01 |
| Use of other hypertension drugs; n (%) | 66 (4.2%) | 70 (4.4%) | -0.01 | 117 (4.0%) | 91 (3.1%) | 0.05 | 522 (6.1%) | 528 (6.2%) | 0.00 | 705 (5.4%) | 689 (5.3%) | 0.00 |
| Use of Anti-arrhythmics; n (%) | ** (0.3%) | ** (0.3%) | 0.00 | ** (0.4%) | ** (0.3%) | 0.02 | 37 (0.4%) | 40 (0.5%) | -0.01 | #VALUE! | #VALUE! | #VALUE! |
| Use of COPD/asthma meds- United: n (%) | 259 (16.4%) | 230 (14.6%) | 0.05 | 414 (14.3%) | 484 (16.7%) | -0.07 | 1.627 (19.1%) | 1.601 (18.8%) | 0.01 | 2300 (17.7%) | 2315 (17.8%) | 0.00 |
| Use of statins: n (%) | 498 (31.6%) | 529 (33.6%) | -0.04 | 680 (23.5%) | 699 (24.1%) | -0.01 | 3,519 (41.3%) | 3,513 (41.3%) | 0.00 | 4697 (36.2%) | 4741 (36.5%) | -0.01 |
| Use of other lipid-lowering drugs; n (%) | 86 (5.5%) | 80 (5.1%) | 0.02 | 130 (4.5%) | 146 (5.0%) | -0.02 | 563 (6.6%) | 571 (6.7%) | 0.00 | 779 (6.0%) | 797 (6.1%) | 0.00 |
| Use of antiplatelet agents; n (%) | 87 (5.5%) | 86 (5.5%) | 0.00 | 167 (5.8%) | 172 (5.9%) | 0.00 | 766 (9.0%) | 749 (8.8%) | 0.01 | 1020 (7.9%) | 1007 (7.8%) | 0.00 |
| Use of heparin and other low-molecular weight | 07 (3.370) | 00 (3.370) | 0.00 | 107 (3.070) | 172 (3.370) | 0.00 | 700 (3.0%) | 743 (0.070) | 0.01 | 1020 (7.570) | 1007 (7.070) | 0.00 |
| heparins; n (%) | 245 (15.6%) | 210 (13.3%) | 0.07 | ** (0.2%) | ** (0.1%) | 0.03 | 986 (11.6%) | 906 (10.6%) | 0.03 | #VALUE! | #VALUE! | #VALUE! |
| Use of NSAIDs: n (%) | 338 (21.5%) | 335 (21.3%) | 0.00 | 686 (23.7%) | 669 (23.1%) | 0.03 | 1,714 (20.1%) | 1.677 (19.7%) | 0.03 | 2738 (21.1%) | 2681 (20.6%) | 0.01 |
| ,, | () | () | | | | | | -, (, | | | | |
| Use of oral corticosteroids; n (%) | 416 (26.4%) | 420 (26.7%) | -0.01 | 748 (25.8%) | 872 (30.1%) | -0.10 | 2,555 (30.0%) | 2,516 (29.6%) | 0.01 | 3719 (28.6%) | 3808 (29.3%) | -0.02 |
| Use of bisphosphonate (United); n (%) | 54 (3.4%) | 54 (3.4%) | 0.00 | 44 (1.5%) | 49 (1.7%) | -0.02 | 424 (5.0%) | 429 (5.0%) | 0.00 | 522 (4.0%) | 532 (4.1%) | -0.01 |
| Use of opioids- United; n (%) | 830 (52.7%) | 829 (52.6%) | 0.00 | 1,743 (60.1%) | 1,733 (59.8%) | 0.01 | 4,168 (49.0%) | 4,215 (49.5%) | -0.01 | 6741 (51.9%) | 6777 (52.2%) | -0.01 |
| Use of antidepressants; n (%) | 460 (29.2%) | 448 (28.4%) | 0.02 | 717 (24.7%) | 709 (24.5%) | 0.00 | 2,420 (28.4%) | 2,431 (28.6%) | 0.00 | 3597 (27.7%) | 3588 (27.6%) | 0.00 |
| Use of antipsychotics; n (%) | 85 (5.4%) | 81 (5.1%) | 0.01 | 115 (4.0%) | 115 (4.0%) | 0.00 | 579 (6.8%) | 570 (6.7%) | 0.00 | 779 (6.0%) | 766 (5.9%) | 0.00 |
| Labs | | | | | | | | | | 4,474 | 4,474 | |
| Lab values- HbA1c (%) v3; n (%) | 190 (12.1%) | 169 (10.7%) | 0.04 | 29 (1.0%) | 29 (1.0%) | 0.00 | N/A | N/A | #VALUE! | 219 (4.9%) | 198 (4.4%) | 0.02 |
| Lab values- HbA1c (%) (within 3 months) v3; n (%) | 110 (7.0%) | 103 (6.5%) | 0.02 | 17 (0.6%) | 19 (0.7%) | -0.01 | N/A | N/A | #VALUE! | 127 (2.8%) | 122 (2.7%) | 0.01 |
| Lab values- HbA1c (%) (within 6 months) v3; n (%) | 190 (12.1%) | 169 (10.7%) | 0.04 | 29 (1.0%) | 29 (1.0%) | 0.00 | N/A | N/A | #VALUE! | 219 (4.9%) | 198 (4.4%) | 0.02 |
| Lab values- BNP; n (%) | ** (0.4%) | ** (0.5%) | -0.01 | 0 (0.0%) | ** (0.1%) | -0.04 | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values- BNP (within 3 months); n (%) | ** (0.4%) | ** (0.4%) | 0.00 | 0 (0.0%) | ** (0.1%) | -0.04 | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values- BNP (within 6 months); n (%) | ** (0.4%) | ** (0.5%) | -0.01 | 0 (0.0%) | ** (0.1%) | -0.04 | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values- BUN (mg/dl); n (%) | 437 (27.7%) | 449 (28.5%) | -0.02 | 35 (1.2%) | 55 (1.9%) | -0.06 | N/A | N/A | #VALUE! | 472 (10.5%) | 504 (11.3%) | -0.03 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 290 (18.4%) | 322 (20.4%) | -0.05 | 23 (0.8%) | 39 (1.3%) | -0.05 | N/A | N/A | #VALUE! | 313 (7.0%) | 361 (8.1%) | -0.04 |
| Lab values- BUN (mg/dl) (within 6 months); n (%) | 437 (27.7%) | 449 (28.5%) | -0.02 | 35 (1.2%) | 55 (1.9%) | -0.06 | N/A | N/A | #VALUE! | 472 (10.5%) | 504 (11.3%) | -0.03 |
| Lab values- Creatinine (mg/dl) v2; n (%) | 452 (28.7%) | 466 (29.6%) | -0.02 | 38 (1.3%) | 59 (2.0%) | -0.05 | N/A | N/A | #VALUE! | 490 (11.0%) | 525 (11.7%) | -0.02 |
| | 432 (20.770) | 400 (25.0%) | -0.02 | 30 (1.370) | 35 (2.0%) | -0.03 | N/A | IN/A | #VALUE: | 450 (11.0%) | 323 (11.7%) | -0.02 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2;<br>n (%) | 301 (19.1%) | 337 (21.4%) | -0.06 | 25 (0.9%) | 42 (1.4%) | -0.05 | N/A | N/A | #VALUE! | 326 (7.3%) | 379 (8.5%) | -0.04 |
| Lab values- Creatinine (mg/dl) (within 6 months) v2; | 301 (19.1%) | 337 (21.470) | -0.00 | 23 (0.5%) | 42 (1.470) | -0.03 | N/A | IV/A | #VALUE: | 320 (7.3%) | 373 (0.370) | -0.04 |
| | 453 (30 70/) | 466 (29.6%) | -0.02 | 20 (4 20/) | EQ (2.00/) | 0.05 | N/A | NI/A | #A/ALLIEL | 400 (11 00/) | EDE (11 70/) | -0.02 |
| n (%) | 452 (28.7%) | , | | 38 (1.3%) | 59 (2.0%) | -0.05 | N/A | N/A | #VALUE! | 490 (11.0%) | 525 (11.7%) | |
| Lab values- HDL level (mg/dl); n (%) | 242 (15.4%) | 263 (16.7%) | -0.04 | 21 (0.7%) | 32 (1.1%) | -0.04 | N/A | N/A | #VALUE! | 263 (5.9%) | 295 (6.6%) | -0.03 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 123 (7.8%) | 146 (9.3%) | -0.05 | ** (0.2%) | 19 (0.7%) | -0.07 | N/A | N/A | #VALUE! | #VALUE! | 165 (3.7%) | #VALUE! |
| cas values ripe rever (ing/or) (within 5 months), ff (%) | 123 (7.0/0) | 140 (3.3/0) | -0.05 | (0.270) | 13 (0.770) | -0.07 | N/A | N/A | #VALUE! | #VALUE: | 103 (3.770) | #VALUE! |
| Lab values- HDL level (mg/dl) (within 6 months); n (%) | 242 (15.4%) | 263 (16.7%) | -0.04 | 21 (0.7%) | 32 (1.1%) | -0.04 | N/A | N/A | #VALUE! | 263 (5.9%) | 295 (6.6%) | -0.03 |
| Lab values-LDL level (mg/dl) v2; n (%) | 244 (15.5%) | 264 (16.8%) | -0.04 | 24 (0.8%) | 32 (1.1%) | -0.03 | N/A | N/A | #VALUE! | 268 (6.0%) | 296 (6.6%) | -0.02 |
| | 244 (13.3%) | 204 (10.6%) | -0.04 | 24 (0.676) | 32 (1.170) | -0.03 | N/A | IV/A | #VALUE: | 208 (0.0%) | 250 (0.0%) | -0.02 |
| Lab values- LDL level (mg/dl) (within 3 months) v2; n | 430 (0.40() | 4.45 (0.20() | | ** (0.20/) | 40 (0.50() | | **** | **/* | | | 452 (2.50() | 10.441.1151 |
| (%) | 128 (8.1%) | 145 (9.2%) | -0.04 | ** (0.3%) | 18 (0.6%) | -0.04 | N/A | N/A | #VALUE! | #VALUE! | 163 (3.6%) | #VALUE! |
| Lab values-LDL level (mg/dl) (within 6 months) v2; n | 244/12 | 204 (1) | | 2.4 | a- / | | | | | 200 (0.00) | 20-1 | |
| (%) | 244 (15.5%) | 264 (16.8%) | -0.04 | 24 (0.8%) | 32 (1.1%) | -0.03 | N/A | N/A | #VALUE! | 268 (6.0%) | 296 (6.6%) | -0.02 |
| Lab values- NT-proBNP; n (%) | ** (0.1%) | ** (0.1%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values- NT-proBNP (within 3 months); n (%) | ** (0.1%) | ** (0.1%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values- NT-proBNP (within 6 months); n (%) | ** (0.1%) | ** (0.1%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | N/A | N/A | #VALUE! | #VALUE! | #VALUE! | #VALUE! |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 245 (15.6%) | 263 (16.7%) | -0.03 | 20 (0.7%) | 32 (1.1%) | -0.04 | N/A | N/A | #VALUE! | 265 (5.9%) | 295 (6.6%) | -0.03 |
| Lab values-Total cholesterol (mg/dl) (within 3 | | | | | | | | | | | | |
| months) v2; n (%) | 125 (7.9%) | 145 (9.2%) | -0.05 | ** (0.2%) | 19 (0.7%) | -0.07 | N/A | N/A | #VALUE! | #VALUE! | 164 (3.7%) | #VALUE! |
| Lab values-Total cholesterol (mg/dl) (within 6 | | | | | | | | | | | | |
| months) v2; n (%) | 245 (15.6%) | 263 (16.7%) | -0.03 | 20 (0.7%) | 32 (1.1%) | -0.04 | N/A | N/A | #VALUE! | 265 (5.9%) | 295 (6.6%) | -0.03 |
| Lab values-Triglyceride level (mg/dl); n (%) | 244 (15.5%) | 265 (16.8%) | -0.04 | 21 (0.7%) | 32 (1.1%) | -0.04 | N/A | N/A | #VALUE! | 265 (5.9%) | 297 (6.6%) | -0.03 |
| Lab values-Triglyceride level (mg/dl) (within 3 | | | | | | | | | | • | | |
| months); n (%) | 126 (8.0%) | 146 (9.3%) | -0.05 | ** (0.2%) | 18 (0.6%) | -0.06 | N/A | N/A | #VALUE! | #VALUE! | 164 (3.7%) | #VALUE! |
| | 7 | | | ** | | | • • | *** | | | | |

| Lab values-Triglyceride level (mg/dl) (within 6 | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| months): n (%) | 244 (15.5%) | 265 (16.8%) | -0.04 | 21 (0.7%) | 32 (1.1%) | -0.04 | N/A | N/A | #VALUE! | 265 (5.9%) | 297 (6.6%) | -0.03 |
| Lab result number- HbA1c (%) mean (only 2 to 20 | , | , | | | , | | | | | , | , | |
| included) v4 | 189 | 169 | | 27 | 28 | | N/A | N/A | | 216 | 197 | |
| mean (sd) | 6.88 (1.71) | 6.69 (1.48) | 0.12 | 7.17 (1.18) | 7.17 (1.32) | 0.00 | N/A | N/A | #VALUE! | 6.92 (1.66) | 6.76 (1.46) | 0.10 |
| Missing; n (%) | 1,386 (88.0%) | 1,406 (89.3%) | -0.04 | 2,872 (99.1%) | 2,871 (99.0%) | 0.01 | N/A | N/A | #VALUE! | 4,258 (95.2%) | 4,277 (95.6%) | -0.02 |
| Lab result number- BNP mean v2 | 7 | 8 | | - | 2 | | N/A | N/A | | 7 | 10 | |
| mean (sd) | 94.99 (97.03) | 197.30 (393.25) | -0.36 | - (-) | 32.00 (28.28) | #VALUE! | N/A | N/A | #VALUE! | #VALUE! | 164.24 (393.40) | #VALUE! |
| Missing; n (%) | 1,568 (99.6%) | 1,567 (99.5%) | 0.01 | 2,899 (100.0%) | 2,897 (99.9%) | 0.04 | N/A | N/A | #VALUE! | 4,467 (99.8%) | 4,464 (99.8%) | 0.00 |
| Lab result number- BUN (mg/dI) mean v2 | 437 | 449 | | 35 | 55 | | N/A | N/A | | 472 | 504 | |
| mean (sd) | 18.11 (8.11) | 17.57 (7.17) | 0.07 | 17.18 (8.16) | 16.40 (6.60) | 0.11 | N/A | N/A | #VALUE! | 18.04 (8.12) | 17.44 (7.12) | 0.08 |
| Missing; n (%) | 1,138 (72.3%) | 1,126 (71.5%) | 0.02 | 2,864 (98.8%) | 2,844 (98.1%) | 0.06 | N/A | N/A | #VALUE! | 4,002 (89.5%) | 3,970 (88.7%) | 0.03 |
| Lab result number- Creatinine (mg/dl) mean (only 0.1 | | | | | | | | | | | | |
| to 15 included) v3 | 447 | 460 | | 37 | 57 | | N/A | N/A | | 484 | 517 | |
| mean (sd) | 0.99 (0.36) | 0.97 (0.28) | 0.06 | 0.95 (0.32) | 0.95 (0.28) | 0.00 | N/A | N/A | #VALUE! | 0.99 (0.36) | 0.97 (0.28) | 0.06 |
| Missing; n (%) | 1,128 (71.6%) | 1,115 (70.8%) | 0.02 | 2,862 (98.7%) | 2,842 (98.0%) | 0.05 | N/A | N/A | #VALUE! | 3,990 (89.2%) | 3,957 (88.4%) | 0.03 |
| Lab result number- HDL level (mg/dl) mean (only | | | | | | | | | | | | |
| =<5000 included) v2 | 242 | 263 | | 21 | 32 | | N/A | N/A | | 263 | 295 | |
| mean (sd) | 52.41 (17.47) | 53.27 (16.64) | -0.05 | 48.62 (13.24) | 44.83 (11.26) | 0.31 | N/A | N/A | #VALUE! | 52.11 (17.22) | 52.35 (16.18) | -0.01 |
| Missing; n (%) | 1,333 (84.6%) | 1,312 (83.3%) | 0.04 | 2,878 (99.3%) | 2,867 (98.9%) | 0.04 | N/A | N/A | #VALUE! | 4,211 (94.1%) | 4,179 (93.4%) | 0.03 |
| Lab result number-LDL level (mg/dl) mean (only | | | | | | | | | | | | |
| =<5000 included) v2 | 239 | 262 | | 21 | 30 | | N/A | N/A | | 260 | 292 | |
| mean (sd) | 101.44 (33.15) | 100.96 (36.42) | 0.01 | 103.33 (25.48) | 94.27 (29.11) | 0.33 | N/A | N/A | #VALUE! | 101.59 (32.68) | 100.27 (35.82) | 0.04 |
| Missing; n (%) | 1,336 (84.8%) | 1,313 (83.4%) | 0.04 | 2,878 (99.3%) | 2,869 (99.0%) | 0.03 | N/A | N/A | #VALUE! | 4,214 (94.2%) | 4,182 (93.5%) | 0.03 |
| Lab result number-Total cholesterol (mg/dl) mean | | | | | | | | | | | | |
| (only =<5000 included) v2 | 245 | 263 | | 20 | 32 | | N/A | N/A | | 265 | 295 | |
| mean (sd) | 180.67 (41.98) | 181.58 (40.29) | -0.02 | 180.45 (27.83) | 180.69 (46.88) | -0.01 | N/A | N/A | #VALUE! | 180.65 (41.20) | 181.48 (41.11) | -0.02 |
| Missing; n (%) | 1,330 (84.4%) | 1,312 (83.3%) | 0.03 | 2,879 (99.3%) | 2,867 (98.9%) | 0.04 | N/A | N/A | #VALUE! | 4,209 (94.1%) | 4,179 (93.4%) | 0.03 |
| Lab result number-Triglyceride level (mg/dl) mean | | | | | | | | | | | | |
| (only =<5000 included) v2 | 244 | 265 | | 21 | 32 | | N/A | N/A | | 265 | 297 | |
| mean (sd) | 134.91 (69.13) | 136.25 (69.41) | -0.02 | 143.67 (74.18) | 177.70 (98.70) | -0.39 | N/A | N/A | #VALUE! | 135.60 (69.66) | 140.72 (73.17) | -0.07 |
| Missing; n (%) | 1,331 (84.5%) | 1,310 (83.2%) | 0.04 | 2,878 (99.3%) | 2,867 (98.9%) | 0.04 | N/A | N/A | #VALUE! | 4,209 (94.1%) | 4,177 (93.4%) | 0.03 |
| Lab result number- Hemoglobin mean (only >0 | | | | | | | | | | | | |
| included) | 368 | 376 | | 25 | 49 | | N/A | N/A | | 393 | 425 | |
| mean (sd) | 13.18 (1.94) | 13.23 (1.89) | -0.03 | 12.30 (3.19) | 12.67 (3.06) | -0.12 | N/A | N/A | #VALUE! | 13.12 (2.04) | 13.17 (2.06) | -0.02 |
| Missing; n (%) | 1,207 (76.6%) | 1,199 (76.1%) | 0.01 | 2,874 (99.1%) | 2,850 (98.3%) | 0.07 | N/A | N/A | #VALUE! | 4,081 (91.2%) | 4,049 (90.5%) | 0.02 |
| Lab result number- Serum sodium mean (only > 90 | | | | | | | | | | | | |
| and < 190 included) | 431 | 438 | | 35 | 53 | | N/A | N/A | | 466 | 491 | |
| mean (sd) | 140.16 (2.94) | 140.09 (2.65) | 0.03 | 139.41 (2.22) | 138.69 (3.08) | 0.27 | N/A | N/A | #VALUE! | 140.10 (2.90) | 139.94 (2.70) | 0.06 |
| Missing; n (%) | 1,144 (72.6%) | 1,137 (72.2%) | 0.01 | 2,864 (98.8%) | 2,846 (98.2%) | 0.05 | N/A | N/A | #VALUE! | 4,008 (89.6%) | 3,983 (89.0%) | 0.02 |
| Lab result number- Albumin mean (only >0 and <=10 | | | | | | | | | | | | |
| included) | 393 | 384 | | 27 | 45 | | N/A | N/A | | 420 | 429 | |
| mean (sd) | 4.07 (0.42) | 4.06 (0.44) | 0.02 | 3.88 (0.89) | 3.96 (0.75) | -0.10 | N/A | N/A | #VALUE! | 4.06 (0.46) | 4.05 (0.48) | 0.02 |
| Missing; n (%) | 1,182 (75.0%) | 1,191 (75.6%) | -0.01 | 2,872 (99.1%) | 2,854 (98.4%) | 0.06 | N/A | N/A | #VALUE! | 4,054 (90.6%) | 4,045 (90.4%) | 0.01 |
| Lab result number- Glucose (fasting or random) mean | | | | | | | | | | | | |
| (only 10-1000 included) | 430 | 438 | | 33 | 54 | | N/A | N/A | | 463 | 492 | |
| mean (sd) | 114.69 (54.46) | 113.20 (40.43) | 0.03 | 141.69 (58.99) | 149.10 (79.94) | -0.11 | N/A | N/A | #VALUE! | 116.61 (54.85) | 117.14 (46.40) | -0.01 |
| Missing; n (%) | 1,145 (72.7%) | 1,137 (72.2%) | 0.01 | 2,866 (98.9%) | 2,845 (98.1%) | 0.07 | N/A | N/A | #VALUE! | 4,011 (89.7%) | 3,982 (89.0%) | 0.02 |
| Lab result number- Potassium mean (only 1-7 | | | | | | | | | | | | |
| included) | 439 | 451 | | 34 | 52 | | N/A | N/A | | 473 | 503 | |
| mean (sd) | 4.36 (0.43) | 4.32 (0.43) | 0.09 | 4.11 (0.33) | 4.32 (0.38) | -0.59 | N/A | N/A | #VALUE! | 4.34 (0.42) | 4.32 (0.43) | 0.05 |
| Missing; n (%) | 1,136 (72.1%) | 1,124 (71.4%) | 0.02 | 2,865 (98.8%) | 2,847 (98.2%) | 0.05 | N/A | N/A | #VALUE! | 4,001 (89.4%) | 3,971 (88.8%) | 0.02 |
| Comorbidity Scores | | | | | | | | | | | | |
| CCI (180 days)- ICD9 and ICD10 v2 | | | | | | | | | | | | |
| mean (sd) | 2.24 (2.49) | 2.23 (2.44) | 0.00 | 1.54 (2.15) | 1.51 (2.17) | 0.01 | 2.33 (2.65) | 2.27 (2.61) | 0.02 | 2.14 (2.53) | 2.10 (2.50) | 0.02 |
| Non-Frailty; n (%) | 758 (48.1%) | 742 (47.1%) | 0.02 | 1,188 (41.0%) | 1,206 (41.6%) | -0.01 | 227 (2.7%) | 162 (1.9%) | 0.05 | 2,173 (16.7%) | 2,110 (16.2%) | 0.01 |
| Frailty Score (mean): Empirical Version 365 days, v2 | | | | | | | | | | | | |
| mean (sd) | 0.20 (0.07) | 0.20 (0.07) | 0.00 | 0.17 (0.06) | 0.17 (0.06) | 0.00 | 0.11 (0.08) | 0.11 (0.08) | 0.00 | 0.13 (0.07) | 0.13 (0.07) | 0.00 |
| Healthcare Utilization | | | | | | | | | | | | |
| Any hospitalization; n (%) | 1,171 (74.3%) | 1,168 (74.2%) | 0.00 | 2,898 (100.0%) | 2,899 (100.0%) | #DIV/0! | 6,540 (76.8%) | 6,597 (77.5%) | -0.02 | 10,609 (81.7%) | 10,664 (82.1%) | -0.01 |
| Any hospitalization within prior 30 days; n (%) | 1,051 (66.7%) | 1,076 (68.3%) | -0.03 | 2,867 (98.9%) | 2,861 (98.7%) | 0.02 | 6,186 (72.7%) | 6,226 (73.2%) | -0.01 | 10104 (77.8%) | 10163 (78.3%) | -0.01 |
| Any hospitalization during prior 31-180 days; n (%) | 285 (18.1%) | 260 (16.5%) | 0.04 | 345 (11.9%) | 385 (13.3%) | -0.04 | 1,609 (18.9%) | 1,500 (17.6%) | 0.03 | 2239 (17.2%) | 2145 (16.5%) | 0.02 |
| Internal medicine/family medicine visits; n (%) | 1,414 (89.8%) | 1,433 (91.0%) | -0.04 | 2,306 (79.5%) | 2,292 (79.1%) | 0.01 | 7,909 (92.9%) | 8,030 (94.3%) | -0.06 | 11629 (89.6%) | 11755 (90.5%) | -0.03 |
| Internal medicine/family medicine visits (30 days | | | | | | | | | | | | |
| prior) v2; n (%) | 1,257 (79.8%) | 1,288 (81.8%) | -0.05 | 1,654 (57.1%) | 1,591 (54.9%) | 0.04 | 7,300 (85.8%) | 7,400 (86.9%) | -0.03 | 10211 (78.6%) | 10279 (79.2%) | -0.01 |
| Internal medicine/family medicine visits (31 to 180 | | | | | | | | | | | | |
| days prior) v2; n (%) | 1,105 (70.2%) | 1,103 (70.0%) | 0.00 | 1,893 (65.3%) | 1,870 (64.5%) | 0.02 | 6,307 (74.1%) | 6,289 (73.9%) | 0.00 | 9305 (71.7%) | 9262 (71.3%) | 0.01 |
| Cardiologist visit; n (%) | 681 (43.2%) | 702 (44.6%) | -0.03 | 626 (21.6%) | 642 (22.1%) | -0.01 | 4,247 (49.9%) | 4,211 (49.5%) | 0.01 | 5554 (42.8%) | 5555 (42.8%) | 0.00 |
| Number of Cardiologist visits (30 days prior); n (%) | 496 (31.5%) | 500 (31.7%) | 0.00 | 377 (13.0%) | 359 (12.4%) | 0.02 | 3,097 (36.4%) | 3,041 (35.7%) | 0.01 | 3970 (30.6%) | 3900 (30.0%) | 0.01 |
| Number of Cardiologist visits (31 to 180 days prior); | | | | | | | | | | | | |
| n (%) | 315 (20.0%) | 327 (20.8%) | -0.02 | 351 (12.1%) | 355 (12.2%) | 0.00 | 2,225 (26.1%) | 2,169 (25.5%) | 0.01 | 2891 (22.3%) | 2851 (22.0%) | 0.01 |
| Electrocardiogram v2; n (%) | 897 (57.0%) | 888 (56.4%) | 0.01 | 1,056 (36.4%) | 1,062 (36.6%) | 0.00 | 5,347 (62.8%) | 5,402 (63.5%) | -0.01 | 7300 (56.2%) | 7352 (56.6%) | -0.01 |
| Use of glucose test strips; n (%) | 27 (1.7%) | 21 (1.3%) | 0.03 | 31 (1.1%) | 30 (1.0%) | 0.01 | 131 (1.5%) | 130 (1.5%) | 0.00 | 189 (1.5%) | 181 (1.4%) | 0.01 |
| Dialysis; n (%) | ** (0.1%) | 0 (0.0%) | 0.04 | ** (0.2%) | ** (0.2%) | 0.00 | <11 (0.1%) | <11 (0.1%) | 0.00 | #VALUE! | #VALUE! | #VALUE! |
| number of different/distinct medication | | | | | | | | | | | | |
| prescriptions | | | | | | | | | | | | |
| mean (sd) | 9.11 (5.28) | 9.12 (5.40) | 0.00 | 9.08 (5.24) | 9.08 (5.82) | 0.00 | 9.99 (5.30) | 9.94 (5.25) | 0.01 | 9.68 (5.28) | 9.65 (5.40) | 0.01 |
| Number of Hospitalizations | | | | | | | | | | | | |
| mean (sd) | 0.97 (0.80) | 0.99 (0.84) | -0.02 | 1.29 (0.70) | 1.29 (0.64) | 0.00 | 1.11 (0.92) | 1.10 (0.89) | 0.01 | 1.13 (0.86) | 1.13 (0.83) | 0.00 |

| Number of hospital days | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 5.10 (5.19) | 5.11 (7.06) | 0.00 | 7.00 (6.55) | 6.98 (8.63) | 0.00 | 6.22 (6.56) | 6.04 (8.07) | 0.02 | 6.26 (6.41) | 6.14 (8.08) | 0.02 |
| Number of Emergency Department (ED) visits v3 | | , | | | , | | , | , | | , | | |
| mean (sd) | 2.07 (2.62) | 2.04 (1.86) | 0.01 | 2.58 (5.38) | 2.66 (7.21) | -0.01 | 2.15 (2.27) | 2.12 (1.90) | 0.01 | 2.24 (3.27) | 2.23 (3.79) | 0.00 |
| Number of Office visits | | | | | | | | | | | | |
| mean (sd) | 5.47 (4.54) | 5.63 (4.70) | -0.03 | 5.58 (5.27) | 5.57 (5.04) | 0.00 | 13.86 (15.96) | 13.58 (15.05) | 0.02 | 10.99 (13.25) | 10.83 (12.52) | 0.01 |
| Number of internal medicine/family medicine visits | | | | | | | | | | | | |
| mean (sd) | 11.72 (18.22) | 9.93 (12.31) | 0.12 | 6.37 (11.98) | 6.10 (10.85) | 0.02 | 12.38 (12.28) | 11.56 (12.82) | 0.07 | 10.96 (13.08) | 10.14 (12.34) | 0.06 |
| Number of Cardiologist visits<br>mean (sd) | 1.41 (3.19) | 1.57 (3.56) | -0.05 | 0.60 (1.92) | 0.57 (1.90) | 0.02 | 1.91 (4.01) | 1.88 (3.85) | 0.01 | 1.56 (3.55) | 1.55 (3.47) | 0.00 |
| Number electrocardiograms received v2 | 1.41 (3.13) | 1.37 (3.30) | -0.03 | 0.00 (1.52) | 0.37 (1.30) | 0.02 | 1.51 (4.01) | 1.00 (3.03) | 0.01 | 1.30 (3.33) | 1.55 (5.47) | 0.00 |
| mean (sd) | 1.26 (1.97) | 1.25 (1.69) | 0.01 | 0.65 (1.20) | 0.66 (1.17) | -0.01 | 1.42 (1.74) | 1.40 (1.64) | 0.01 | 1.23 (1.67) | 1.22 (1.55) | 0.01 |
| Number of HbA1c tests ordered | , | , | | , | , | | , , | | | , , | ,, | |
| mean (sd) | 0.36 (0.67) | 0.34 (0.65) | 0.03 | 0.21 (0.57) | 0.22 (0.55) | -0.02 | 0.38 (0.71) | 0.37 (0.70) | 0.01 | 0.34 (0.68) | 0.33 (0.66) | 0.01 |
| Number of glucose tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.41 (5.52) | 0.41 (5.16) | 0.00 | 0.14 (0.62) | 0.15 (0.64) | -0.02 | 0.19 (0.89) | 0.18 (0.69) | 0.01 | 0.21 (2.07) | 0.20 (1.91) | 0.01 |
| Number of lipid tests ordered<br>mean (sd) | 0.49 (0.78) | 0.47 (0.74) | 0.03 | 0.35 (0.80) | 0.34 (0.78) | 0.01 | 0.53 (0.77) | 0.53 (0.75) | 0.00 | 0.48 (0.78) | 0.48 (0.76) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd | 0.45 (0.76) | 0.47 (0.74) | 0.03 | 0.33 (0.80) | 0.34 (0.78) | 0.01 | 0.33 (0.77) | 0.33 (0.73) | 0.00 | 0.46 (0.76) | 0.48 (0.70) | 0.00 |
| digit level Copy | | | | | | | | | | | | |
| mean (sd) | 9.94 (12.57) | 10.03 (12.80) | -0.01 | 7.61 (11.53) | 7.46 (11.79) | 0.01 | 12.03 (13.75) | 11.42 (13.25) | 0.05 | 10.79 (13.14) | 10.37 (12.88) | 0.03 |
| For PS | | | | | | | | | | | | |
| Hemorrhagic stroke+Other cerebrovascular | | | | | | | | | | | | |
| disease+Cerebrovascular procedure (for PS); n (%) | 22 (1.4%) | 29 (1.8%) | -0.03 | 23 (0.8%) | 29 (1.0%) | -0.02 | 178 (2.1%) | 183 (2.2%) | -0.01 | 223 (1.7%) | 241 (1.9%) | -0.02 |
| Major trauma potentially causing prolonged immobili | 189 (12.0%) | 189 (12.0%) | #DIV/0! | 313 (10.8%) | 301 (10.4%) | #DIV/0! | 836 (9.8%) | 771 (9.1%) | #DIV/0! | 313 (10.8%) | 301 (10.4%) | 0.01 |
| Occurrence of creatinine tests ordered (for PS): n (%) | 112 (7.1%) | 133 (8.4%) | -0.05 | 183 (6.3%) | 194 (6.7%) | -0.02 | 898 (10.6%) | 898 (10.6%) | 0.00 | 1193 (9.2%) | 1225 (9.4%) | -0.01 |
| Occurrence of BUN tests ordered (for PS); n (%) | 63 (4.0%) | 58 (3.7%) | 0.02 | 109 (3.8%) | 115 (4.0%) | -0.01 | 514 (6.0%) | 500 (5.9%) | 0.00 | 686 (5.3%) | 673 (5.2%) | 0.00 |
| Occurrence of chronic renal insufficiency w/o CKD | (, | | | () | ( , | | () | 222 (2.2) | | ( | 2.2 (2.2) | |
| (for PS) v2; n (%) | 106 (6.7%) | 105 (6.7%) | 0.00 | 96 (3.3%) | 97 (3.3%) | 0.00 | 656 (7.7%) | 687 (8.1%) | -0.01 | 858 (6.6%) | 889 (6.8%) | -0.01 |
| Chronic kidney disease Stage 1-2 (for PS); n (%) | 27 (1.7%) | 30 (1.9%) | -0.02 | 21 (0.7%) | 22 (0.8%) | -0.01 | 153 (1.8%) | 155 (1.8%) | 0.00 | 201 (1.5%) | 207 (1.6%) | -0.01 |
| Chronic kidney disease Stage 3-6 (for PS); n (%) | 117 (7.4%) | 132 (8.4%) | -0.04 | 73 (2.5%) | 79 (2.7%) | -0.01 | 724 (8.5%) | 715 (8.4%) | 0.00 | 914 (7.0%) | 926 (7.1%) | 0.00 |
| Acute kidney injury; n (%) | 180 (11.4%) | 191 (12.1%) | #DIV/0! | 239 (8.2%) | 264 (9.1%) | #DIV/0!<br>-0.01 | 1,052 (12.4%) | 1,062 (12.5%) | #DIV/0! | 239 (8.2%) | 264 (9.1%) | -0.03<br>0.02 |
| Bladder stones+Kidney stones (for PS); n (%)<br>Alcohol abuse or dependence+Drug abuse or | 52 (3.3%) | 49 (3.1%) | 0.01 | 83 (2.9%) | 89 (3.1%) | -0.01 | 302 (3.5%) | 260 (3.1%) | 0.02 | 437 (3.4%) | 398 (3.1%) | 0.02 |
| dependence (for PS); n (%) | 114 (7.2%) | 105 (6.7%) | 0.02 | 132 (4.6%) | 129 (4.4%) | 0.01 | 186 (2.2%) | 179 (2.1%) | 0.01 | 432 (3.3%) | 413 (3.2%) | 0.01 |
| Other atherosclerosis+Cardiac conduction | | . , | | , , | | | | | | , , | | |
| disorders+Other CVD (for PS) v2 Copy; n (%) | 327 (20.8%) | 310 (19.7%) | 0.03 | 506 (17.5%) | 526 (18.1%) | -0.02 | 1,794 (21.1%) | 1,779 (20.9%) | 0.00 | 2627 (20.2%) | 2615 (20.1%) | 0.00 |
| Previous cardiac procedure (CABG or PTCA or Stent) + | | | | | | | | | | | | |
| History of CABG or PTCA (for PS) v3; n (%) | 59 (3.7%) | 74 (4.7%) | -0.05 | 54 (1.9%)<br>230 (7.9%) | 51 (1.8%) | 0.01 | 631 (7.4%)<br>1.003 (11.8%) | 648 (7.6%)<br>973 (11.4%) | -0.01<br>#DIV/0! | 744 (5.7%)<br>230 (7.9%) | 773 (6.0%)<br>233 (8.0%) | -0.01<br>0.00 |
| Diabetes with complication; n (%) | 192 (12.2%) | 203 (12.9%) | #DIV/0! | , | 233 (8.0%) | #DIV/0! | , , | | , | , | | |
| Delirium + Psychosis (for PS); n (%) | 107 (6.8%) | 100 (6.3%) | 0.02 | 123 (4.2%) | 121 (4.2%) | 0.00 | 729 (8.6%) | 682 (8.0%) | 0.02 | 959 (7.4%) | 903 (7.0%) | 0.02 |
| Delirium + Psychosis (for PS); n (%)<br>Any use of Meglitinides (for PS); n (%) | 107 (6.8%)<br>** (0.1%) | 100 (6.3%)<br>** (0.3%) | , | 123 (4.2%)<br>** (0.1%) | 121 (4.2%)<br>** (0.1%) | , | , , | | , | , | 903 (7.0%)<br>#VALUE! | 0.02<br>#VALUE! |
| Delirium + Psychosis (for PS); n (%) | 107 (6.8%) | 100 (6.3%) | 0.02<br>-0.04 | 123 (4.2%) | 121 (4.2%) | 0.00<br>0.00 | 729 (8.6%)<br>22 (0.3%) | 682 (8.0%)<br>33 (0.4%) | 0.02<br>-0.02 | 959 (7.4%)<br>#VALUE! | 903 (7.0%) | 0.02 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) | 107 (6.8%)<br>** (0.1%)<br>0 (0.0%)<br>120 (7.6%)<br>149 (9.5%) | 100 (6.3%)<br>** (0.3%)<br>** (0.2%)<br>133 (8.4%)<br>147 (9.3%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>0.01 | 123 (4.2%)<br>** (0.1%)<br>0 (0.0%)<br>78 (2.7%)<br>211 (7.3%) | 121 (4.2%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) | 0.00<br>0.00<br>-0.04<br>-0.01<br>0.02 | 729 (8.6%)<br>22 (0.3%)<br><11 (0.1%)<br>730 (8.6%)<br>907 (10.7%) | 682 (8.0%)<br>33 (0.4%)<br><11 (0.1%)<br>721 (8.5%)<br>938 (11.0%) | 0.02<br>-0.02<br>0.00<br>0.00<br>-0.01 | 959 (7.4%)<br>#VALUE!<br>#VALUE!<br>928 (7.1%)<br>1267 (9.8%) | 903 (7.0%)<br>#VALUE!<br>#VALUE!<br>939 (7.2%)<br>1280 (9.9%) | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>0.00 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of beta blockers; n (%) | 107 (6.8%)<br>** (0.1%)<br>0 (0.0%)<br>120 (7.6%)<br>149 (9.5%)<br>366 (23.2%) | 100 (6.3%)<br>** (0.3%)<br>** (0.2%)<br>133 (8.4%)<br>147 (9.3%)<br>379 (24.1%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>0.01<br>-0.02 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) | 121 (4.2%) ** (0.1%) ** (0.1%) *5 (2.9%) 195 (6.7%) 546 (18.8%) | 0.00<br>0.00<br>-0.04<br>-0.01<br>0.02<br>0.02 | 729 (8.6%)<br>22 (0.3%)<br><11 (0.1%)<br>730 (8.6%)<br>907 (10.7%)<br>2,831 (33.3%) | 682 (8.0%)<br>33 (0.4%)<br><11 (0.1%)<br>721 (8.5%)<br>938 (11.0%)<br>2,870 (33.7%) | 0.02<br>-0.02<br>0.00<br>0.00<br>-0.01<br>-0.01 | 959 (7.4%)<br>#VALUE!<br>#VALUE!<br>928 (7.1%)<br>1267 (9.8%)<br>3759 (28.9%) | 903 (7.0%)<br>#VALUE!<br>#VALUE!<br>939 (7.2%)<br>1280 (9.9%)<br>3795 (29.2%) | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>0.00<br>-0.01 |
| Delirium + Psychosis (for PS); n (%) An y use of Meglitinides (for PS); n (%) Any use of AGIs (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of bet a blockers; n (%) Use of calcium channel blockers; n (%) | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) | 100 (6.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>0.01<br>-0.02<br>-0.03 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) | 0.00<br>0.00<br>-0.04<br>-0.01<br>0.02<br>0.02<br>0.00 | 729 (8.6%)<br>22 (0.3%)<br><11 (0.1%)<br>730 (8.6%)<br>907 (10.7%)<br>2,831 (33.3%)<br>2,270 (26.7%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) | 0.02<br>-0.02<br>0.00<br>0.00<br>-0.01<br>-0.01 | 959 (7.4%)<br>#VALUE!<br>#VALUE!<br>928 (7.1%)<br>1267 (9.8%)<br>3759 (28.9%)<br>3004 (23.1%) | 903 (7.0%)<br>#VALUE!<br>#VALUE!<br>939 (7.2%)<br>1280 (9.9%)<br>3795 (29.2%)<br>2994 (23.1%) | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>0.00<br>-0.01<br>0.00 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of AGIs (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of beta blockers; n (%) Use of otalicum channel blockers; n (%) All antidiabetic medications except Insulin; n (%) | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) | 100 (6.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>0.01<br>-0.02<br>-0.03<br>0.00 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) | 121 (4.2%) ** (0.1%) ** (0.1%) *5 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) | 0.00<br>0.00<br>-0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) | 0.02<br>-0.02<br>0.00<br>0.00<br>-0.01<br>-0.01<br>-0.01 | 959 (7.4%) #VALUE! #VALUE! 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) | 903 (7.0%)<br>#VALUE!<br>#VALUE!<br>939 (7.2%)<br>1280 (9.9%)<br>3795 (29.2%)<br>2994 (23.1%)<br>2052 (15.8%) | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>0.00<br>-0.01<br>0.00<br>-0.01 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of theta blockers; n (%) Use of of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - Insulin Copy; n (%) | 107 (6.8%)<br>** (0.1%)<br>0 (0.0%)<br>120 (7.6%)<br>149 (9.5%)<br>366 (23.2%)<br>297 (18.9%)<br>241 (15.3%)<br>96 (6.1%) | 100 (6.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>0.01<br>-0.02<br>-0.03<br>0.00 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) | 121 (4.2%) ** (0.1%) ** (0.1%) *5 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) | 0.00<br>0.00<br>-0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) | 0.02<br>-0.02<br>0.00<br>0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.01 | 959 (7.4%)<br>#VALUE!<br>#VALUE!<br>928 (7.1%)<br>1267 (9.8%)<br>3759 (28.9%)<br>3004 (23.1%)<br>2011 (15.5%)<br>617 (4.8%) | 903 (7.0%)<br>#VALUE!<br>#VALUE!<br>939 (7.2%)<br>1280 (9.9%)<br>3795 (29.2%)<br>2994 (23.1%)<br>2052 (15.8%)<br>670 (5.2%) | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>0.00<br>-0.01<br>0.00<br>-0.01<br>-0.02 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of Alois (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of bet a blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except insulin; n (%) DM Medications - Insulin Copy; n (%) Use of Low Intensity Statins; n (%) | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) | 100 (6.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>0.01<br>-0.02<br>-0.03<br>0.00<br>0.00 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) | 0.00<br>0.00<br>-0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.02 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,355 (27.6%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) | 0.02<br>-0.02<br>0.00<br>0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.01<br>-0.02 | 959 (7.4%) #WALUE! #WALUE! 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 617 (4.8%) 3056 (23.5%) | 903 (7.0%) #VALUE! #VALUE! 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 3147 (24.2%) | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>0.00<br>-0.01<br>0.00<br>-0.01<br>-0.02 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of theta blockers; n (%) Use of of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - Insulin Copy; n (%) | 107 (6.8%)<br>** (0.1%)<br>0 (0.0%)<br>120 (7.6%)<br>149 (9.5%)<br>366 (23.2%)<br>297 (18.9%)<br>241 (15.3%)<br>96 (6.1%) | 100 (6.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>0.01<br>-0.02<br>-0.03<br>0.00 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) | 121 (4.2%) ** (0.1%) ** (0.1%) *5 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) | 0.00<br>0.00<br>-0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) | 0.02<br>-0.02<br>0.00<br>0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.01 | 959 (7.4%)<br>#VALUE!<br>#VALUE!<br>928 (7.1%)<br>1267 (9.8%)<br>3759 (28.9%)<br>3004 (23.1%)<br>2011 (15.5%)<br>617 (4.8%) | 903 (7.0%)<br>#VALUE!<br>#VALUE!<br>939 (7.2%)<br>1280 (9.9%)<br>3795 (29.2%)<br>2994 (23.1%)<br>2052 (15.8%)<br>670 (5.2%) | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>0.00<br>-0.01<br>0.00<br>-0.01<br>-0.02 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thisaide; n (%) Use of beta blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except insulin; n (%) DM Medications - Insulin Copy; n (%) Use of Low intensity Statins; n (%) Use of High Intensity Statins; n (%) | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) | 100 (6.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>0.01<br>-0.02<br>-0.03<br>0.00<br>0.00 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) | 0.00<br>0.00<br>-0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.04<br>0.02 | 729 (8.6%) 22 (0.3%) 41 (0.1%) 730 (8.6%) 907 (10.7%) 2.831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) | 0.02<br>-0.02<br>0.00<br>0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01 | 959 (7.4%) #VALUE! #VALUE! 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 617 (4.8%) 3056 (23.5%) | 903 (7.0%) #VALUE! #VALUE! 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 3147 (24.2%) 1661 (12.8%) | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>0.00<br>-0.01<br>0.00<br>-0.01<br>-0.02<br>-0.02 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of theta blockers; n (%) Use of teat a blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except insulin; n (%) DM Medications - Insulin Copy; n (%) Use of High Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) | 100 (6.3%) ** (0.3%) ** (0.2%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>0.01<br>-0.02<br>-0.03<br>0.00<br>0.00<br>-0.05<br>0.00<br>-0.11 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) | 0.00<br>0.00<br>-0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.04<br>0.02<br>-0.05 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 2,872 (33.7%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) | 0.02<br>-0.02<br>0.00<br>0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>0.00<br>-0.06 | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 417 (4.8%) 3056 (23.5%) 1676 (12.9%) 3345 (30.4%) | 903 (7.0%) #VALUEI #VALUEI 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 3147 (24.2%) 1661 (12.8%) 4307 (33.2%) | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>0.00<br>-0.01<br>0.00<br>-0.01<br>-0.02<br>-0.02<br>0.00<br>-0.06 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of Adis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of the blockers; n (%) Use of beta blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - Insulin Copy; n (%) Use of Low Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP tests | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) ** (0.4%) 278 (17.7%) | 100 (6.3%) ** (0.3%) ** (0.2%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.11<br>-0.06<br>-0.07 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.02<br>-0.04<br>-0.05<br>-0.05 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2.831 (33.3%) 2.270 (26.7%) 1.433 (16.8%) 380 (4.5%) 2.353 (27.6%) 1.202 (14.1%) 2.872 (33.7%) 58 (0.7%) 1,743 (20.5%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.00<br>-0.02<br>-0.04<br>-0.02 | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 617 (4.8%) 3056 (23.5%) 1676 (12.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) | 903 (7.0%) #VALUEI 939 (7.2%) 1280 (9.9%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 1407 (24.2%) 1611 (12.8%) #VALUEI 2709 (20.9%) | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.06<br>#VALUE!<br>-0.03 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of theta blockers; n (%) Use of teat a blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except insulin; n (%) DM Medications - Insulin Copy; n (%) Use of High Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) ** (0.4%) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.11<br>-0.06 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 552 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) | 0.00<br>0.00<br>-0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.04 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2.831 (33.3%) 2.270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 2,872 (33.7%) 58 (0.7%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) | 0.02<br>-0.02<br>0.00<br>0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>0.00<br>-0.06<br>0.06 | 959 (7.4%) #WALUE! 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 617 (4.8%) 3056 (23.5%) 1676 (12.9%) 3945 (30.4%) | 903 (7.0%) #WALUEI 939 (7.2%) 1280 (9.9%) 1295 (9.2%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 3147 (24.2%) 1661 (12.8%) 4307 (33.2%) #WALUEI | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>0.00<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.06 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of theta blockers; n (%) Use of theta blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - insulin Copy; n (%) Use of tigh Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) | 107 (6.8%) **(0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) **(0.4%) 278 (17.7%) 0.08 (0.35) | 100 (6.3%) ** (0.3%) ** (0.2%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.11<br>-0.06<br>-0.07 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.02<br>-0.04<br>-0.05<br>-0.05 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2.831 (33.3%) 2.270 (26.7%) 1.433 (16.8%) 380 (4.5%) 2.353 (27.6%) 1.202 (14.1%) 2.872 (33.7%) 58 (0.7%) 1,743 (20.5%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.00<br>-0.02<br>-0.04<br>-0.02 | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 617 (4.8%) 3056 (23.5%) 1676 (12.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) | 903 (7.0%) #VALUEI 939 (7.2%) 1280 (9.9%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 1407 (24.2%) 1611 (12.8%) #VALUEI 2709 (20.9%) | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.06<br>#VALUE!<br>-0.03 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of the blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except insulin; n (%) DM Medications - Insulin Copy; n (%) Use of Low Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Cardiac biomarkers tests (tropnin, CK-MBs, N | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) ** (0.4%) 278 (17.7%) 0.08 (0.35) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.11<br>-0.06<br>-0.07 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 574 (19.8%) 0.05 (0.25) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.02<br>-0.04<br>-0.05<br>-0.05 | 729 (8.6%) 22 (0.3%) 41 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 2,872 (33.7%) 58 (0.7%) 1,743 (20.5%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.00<br>-0.02<br>-0.04<br>-0.02 | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 3015 (23.5%) 1676 (12.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) 0.08 (0.32) | 903 (7.0%) #VALUEI 939 (7.2%) 1280 (9.9%) 1280 (9.9%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 3147 (24.2%) 1661 (12.8%) 4307 (33.2%) #VALUEI 2709 (20.9%) | 0.02<br>#VALUE!<br>#VALUE!<br>0.00<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.06<br>#VALUE!<br>-0.03 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of theta blockers; n (%) Use of theta blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - insulin Copy; n (%) Use of tigh Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) | 107 (6.8%) **(0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) **(0.4%) 278 (17.7%) 0.08 (0.35) | 100 (6.3%) ** (0.3%) ** (0.2%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.11<br>-0.06<br>-0.07 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.02<br>-0.04<br>-0.05<br>-0.05<br>-0.04 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2.831 (33.3%) 2.270 (26.7%) 1.433 (16.8%) 380 (4.5%) 2.353 (27.6%) 1.202 (14.1%) 2.872 (33.7%) 58 (0.7%) 1,743 (20.5%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.02<br>-0.04<br>-0.06<br>-0.04 | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 617 (4.8%) 3056 (23.5%) 1676 (12.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) | 903 (7.0%) #VALUEI 939 (7.2%) 1280 (9.9%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 1407 (24.2%) 1611 (12.8%) #VALUEI 2709 (20.9%) | 0.02 #VALUE! 0.00 0.00 -0.01 0.00 -0.01 -0.02 -0.02 -0.02 -0.00 -0.06 #VALUE! -0.03 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of AGIs (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thailardie; n (%) Use of beta blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - Insulin Copy; n (%) Use of Low Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Cardiac biomarkers tests (tropnin, CK-MBs, Nmean (sd) Number of Ambulatory Blood pressure monitoring tests | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) ** (0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.11<br>-0.06<br>-0.07 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) 0.05 (0.25) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.04<br>-0.05<br>-0.04<br>-0.03 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 2,872 (33.7%) 58 (0.7%) 1,743 (20.5%) 0.09 (0.34) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.01<br>-0.06<br>-0.06<br>-0.04<br>-0.02 | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3050 (23.1%) 2011 (15.5%) 3016 (23.1%) 3056 (23.5%) 1676 (12.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) 0.08 (0.32) | 903 (7.0%) #WALUEI #WALUEI 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 670 (5.2%) 3147 (24.2%) 3161 (12.8%) 4307 (33.2%) #WALUEI 2709 (20.9%) 0.08 (0.32) | 0.02<br>#VALUE!<br>0.00<br>0.00<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.02<br>-0.06<br>#VALUE!<br>-0.03 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of AGIs (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of theta blockers; n (%) Use of theta blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - Insulin Copy; n (%) Use of I will intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Cardiac biomarkers tests (tropnin, CK-MBs, Nmean (sd) | 107 (6.8%) **(0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) **(0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.11<br>-0.06<br>-0.07 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 574 (19.8%) 0.05 (0.25) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.02<br>-0.04<br>-0.05<br>-0.05<br>-0.04 | 729 (8.6%) 22 (0.3%) 41 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 2,872 (33.7%) 58 (0.7%) 1,743 (20.5%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.02<br>-0.04<br>-0.06<br>-0.04 | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 3015 (23.5%) 1676 (12.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) 0.08 (0.32) | 903 (7.0%) #VALUEI 939 (7.2%) 1280 (9.9%) 1280 (9.9%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 3147 (24.2%) 1661 (12.8%) 4307 (33.2%) #VALUEI 2709 (20.9%) | 0.02 #VALUE! 0.00 0.00 -0.01 0.00 -0.01 -0.02 -0.02 -0.02 -0.00 -0.06 #VALUE! -0.03 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of Adis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of the blockers; n (%) Use of beta blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - Insulin Copy; n (%) Use of Low Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Cardiac biomarkers tests (tropnin, CK-MBs, Nmean (sd) Number of Ambulatory Blood pressure monitoring testsmean (sd) | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) ** (0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.11<br>-0.06<br>-0.07 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) 0.05 (0.25) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.04<br>-0.05<br>-0.04<br>-0.03 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 2,872 (33.7%) 58 (0.7%) 1,743 (20.5%) 0.09 (0.34) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.01<br>-0.06<br>-0.06<br>-0.04<br>-0.02 | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3050 (23.1%) 2011 (15.5%) 3016 (23.1%) 3056 (23.5%) 1676 (12.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) 0.08 (0.32) | 903 (7.0%) #WALUEI #WALUEI 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 670 (5.2%) 3147 (24.2%) 3161 (12.8%) 4307 (33.2%) #WALUEI 2709 (20.9%) 0.08 (0.32) | 0.02<br>#VALUE!<br>0.00<br>0.00<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.02<br>-0.06<br>#VALUE!<br>-0.03 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of beta blockers; n (%) Use of beta blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - Insulin Copy; n (%) Use of Low intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Ambulatory Blood pressure monitoring testsmean (sd) Nof days on antihypertensive medications during baseli | 107 (6.8%) **(0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) **(0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) | 100 (6.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) 0.37 (1.19) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.05<br>-0.07<br>-0.00 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) 0.24 (0.91) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) 0.05 (0.25) 0.26 (0.93) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.02<br>-0.02<br>-0.04<br>-0.05<br>-0.04<br>-0.03<br>-0.04 | 729 (8.6%) 22 (0.3%) 41 (0.1%) 730 (8.6%) 907 (10.7%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 2,872 (33.7%) 58 (0.7%) 1,743 (20.5%) 0.09 (0.34) 0.23 (0.59) | 682 (8.0%) 33 (0.4%) 411 (0.1%) 721 (8.5%) 938 (11.0%) 9.870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) 0.23 (0.58) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.02<br>-0.01<br>-0.00<br>-0.06<br>-0.04<br>-0.02 | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 617 (4.8%) 3056 (23.5%) 1676 (21.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) 0.08 (0.32) | 903 (7.0%) #VALUEI #VALUEI 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 3147 (24.2%) 4307 (33.2%) #VALUEI 2709 (20.9%) 0.08 (0.32) 0.25 (0.77) | 0.02 #VALUE! #VALUE! #VAUE! 0.00 0.00 -0.01 0.00 -0.01 -0.02 -0.02 -0.00 -0.06 #VALUE! -0.03 0.00 0.00 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of Adis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of the blockers; n (%) Use of beta blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - Insulin Copy; n (%) Use of Low Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Cardiac biomarkers tests (tropnin, CK-MBs, Nmean (sd) Number of Ambulatory Blood pressure monitoring testsmean (sd) | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) ** (0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.11<br>-0.06<br>-0.07 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) 0.05 (0.25) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.04<br>-0.05<br>-0.04<br>-0.03 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 2,872 (33.7%) 58 (0.7%) 1,743 (20.5%) 0.09 (0.34) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.01<br>-0.06<br>-0.06<br>-0.04<br>-0.02 | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3050 (23.1%) 2011 (15.5%) 3016 (23.1%) 3056 (23.5%) 1676 (12.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) 0.08 (0.32) | 903 (7.0%) #WALUEI #WALUEI 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 670 (5.2%) 3147 (24.2%) 3161 (12.8%) 4307 (33.2%) #WALUEI 2709 (20.9%) 0.08 (0.32) | 0.02<br>#VALUE!<br>0.00<br>0.00<br>-0.01<br>-0.01<br>-0.02<br>-0.02<br>-0.02<br>-0.06<br>#VALUE!<br>-0.03 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglittinides (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of thiazide; n (%) Use of theat blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - Insulin Copy; n (%) Use of High Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Ambulatory Blood pressure monitoring testsmean (sd) N of days on antihypertensive medications during baselimean (sd) | 107 (6.8%) **(0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) **(0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) | 100 (6.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) 0.37 (1.19) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.05<br>-0.07<br>-0.00 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) 0.24 (0.91) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) 0.05 (0.25) 0.26 (0.93) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.02<br>-0.02<br>-0.04<br>-0.05<br>-0.04<br>-0.03<br>-0.04 | 729 (8.6%) 22 (0.3%) 41 (0.1%) 730 (8.6%) 907 (10.7%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 2,872 (33.7%) 58 (0.7%) 1,743 (20.5%) 0.09 (0.34) 0.23 (0.59) | 682 (8.0%) 33 (0.4%) 411 (0.1%) 721 (8.5%) 938 (11.0%) 9.870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) 0.23 (0.58) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.02<br>-0.01<br>-0.00<br>-0.06<br>-0.04<br>-0.02 | 959 (7.4%) #VALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 617 (4.8%) 3056 (23.5%) 1676 (21.9%) 3945 (30.4%) #VALUEI 2565 (19.8%) 0.08 (0.32) | 903 (7.0%) #VALUEI #VALUEI 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 3147 (24.2%) 4307 (33.2%) #VALUEI 2709 (20.9%) 0.08 (0.32) 0.25 (0.77) | 0.02 #VALUE! #VALUE! #VAUE! 0.00 0.00 -0.01 0.00 -0.01 -0.02 -0.02 -0.00 -0.06 #VALUE! -0.03 0.00 0.00 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGIs (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of theta blockers; n (%) Use of theta blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - insulin Copy; n (%) Use of High Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Cardiac biomarkers tests (tropnin, CK-MBs, Nmean (sd) Number of Ambulatory Blood pressure monitoring testsmean (sd) N of days on antihypertensive medications during baselimean (sd) N of days in database anytime priormean (sd) | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) ** (0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) ine 80.03 (79.04) 1,668.43 (1,266.59) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) 0.37 (1.19) 0.00 (0.00) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.05<br>-0.07<br>-0.00 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) 0.24 (0.91) 0.00 (0.02) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) 0.05 (0.25) 0.26 (0.93) 0.00 (0.03) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>-0.02<br>-0.02<br>-0.05<br>-0.04<br>-0.03<br>-0.04 | 729 (8.6%) 22 (0.3%) <11 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 5,8 (0.7%) 1,743 (20.5%) 0.09 (0.34) 0.23 (0.59) 0.00 (0.03) | 682 (8.0%) 33 (0.4%) 411 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) 0.23 (0.58) 0.00 (0.06) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.00<br>-0.06<br>-0.04<br>-0.02<br>-0.00 | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 617 (4.8%) 3056 (23.5%) 167 (21.9%) 3946 (30.4%) #WALUEI 2565 (19.8%) 0.08 (0.32) 0.24 (0.74) 92.83 (77.61) | 903 (7.0%) #VALUEI 939 (7.2%) 1280 (9.9%) 1290 (9.9%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 3147 (24.2%) 1661 (12.8%) 4307 (33.2%) #VALUEI 2709 (20.9%) 0.08 (0.32) 0.25 (0.77) | 0.02<br>#VALUE!<br>0.00<br>0.00<br>-0.01<br>-0.02<br>-0.02<br>-0.02<br>-0.06<br>#VALUE!<br>-0.03<br>0.00 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of AGIs (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of beta blockers; n (%) Use of beta blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications - Insulin Copy; n (%) Use of Low intensity Statins; n (%) Use of High Intensity Statins; n (%) Gardiovascular stress test; n (%) Echocardiogram; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Ambulatory Blood pressure monitoring testsmean (sd) N of days on antihypertensive medications during baselimean (sd) N of days on database anytime priormean (sd) Mean Copay for per prescription cost (charges in U.S. \$) | 107 (6.8%) **(0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) **(0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) 5: 0.00 (0.05) ine 80.03 (79.04) 1,668.43 (1,266.59) (180-1 day prior) | 100 (6.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) 0.37 (1.19) 0.00 (0.00) 83.44 (80.30) 1,713.11 (1,303.00) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.07<br>-0.06<br>-0.07<br>-0.00<br>-0.05<br>-0.00<br>-0.00 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) 0.24 (0.91) 0.00 (0.02) 62.02 (76.84) 1,982.39 (1,383.61) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) 0.05 (0.25) 0.26 (0.93) 0.00 (0.03) 61.63 (76.67) 2,031.47 (1,419.09) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.02<br>-0.02<br>-0.04<br>-0.03<br>-0.04<br>-0.03<br>-0.04<br>-0.04 | 729 (8.6%) 22 (0.3%) 41 (0.1%) 730 (8.6%) 907 (10.7%) 907 (10.7%) 2.831 (33.3%) 2.270 (26.7%) 1.433 (16.8%) 380 (4.5%) 2.353 (27.6%) 1.202 (14.1%) 2.872 (33.7%) 58 (0.7%) 1.743 (20.5%) 0.09 (0.34) 0.23 (0.59) 0.00 (0.03) | 682 (8.0%) 33 (0.4%) 411 (0.1%) 721 (8.5%) 938 (11.0%) 938 (11.0%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.5%) 37 (0.4%) 0.09 (0.34) 0.23 (0.58) 0.00 (0.06) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.02<br>-0.01<br>-0.00<br>-0.06<br>-0.04<br>-0.02<br>-0.00<br>-0.00 | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 617 (4.8%) 3056 (23.5%) 1676 (22.5%) 3945 (30.4%) #WALUEI 2565 (19.8%) 0.08 (0.32) 0.24 (0.74) 0.00 (0.03) 92.83 (77.61) | 903 (7.0%) #WALUEI #WALUEI 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 670 (5.2%) 3447 (24.2%) 1460 (12.8%) 4307 (33.2%) 9.08 (0.32) 0.08 (0.32) 0.25 (0.77) 0.00 (0.05) | 0.02 #VALUE! #VALUE! 0.00 0.00 -0.01 0.00 -0.01 -0.02 -0.02 -0.06 #VALUE! -0.03 0.00 0.00 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of thiazide; n (%) Use of theat blockers; n (%) Use of teat blockers; n (%) All antidiabetic medications except insulin; n (%) DM Medications - Insulin Copy; n (%) Use of tight intensity Statins; n (%) Use of tight intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Ambulatory Blood pressure monitoring testsmean (sd) N of days on antihypertensive medications during baselimean (sd) N of days in database anytime priormean (sd) Mean Copay for per prescription cost (charges in U.S. S)mean (sd) | 107 (6.8%) ** (0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) ** (0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) ; 0.00 (0.05) ine 80.03 (79.04) 1,668.43 (1,266.59) (180-1 day prior) 23.17 (31.74) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) 0.37 (1.19) 0.00 (0.00) 83.44 (80.30) 1,713.11 (1,303.00) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.07<br>-0.05<br>-0.00<br>-0.05<br>-0.00<br>-0.05 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 331 (11.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) 0.24 (0.91) 0.00 (0.02) 62.02 (76.84) 1,982.39 (1,383.61) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) 0.05 (0.25) 0.26 (0.93) 0.00 (0.03) 61.63 (76.67) 2,031.47 (1,419.09) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.00<br>-0.02<br>-0.02<br>-0.04<br>-0.02<br>-0.05<br>-0.04<br>-0.03<br>-0.04<br>-0.02<br>-0.04 | 729 (8.6%) 22 (0.3%) 41 (0.1%) 730 (8.6%) 907 (10.7%) 907 (10.7%) 1.433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 2,872 (33.7%) 58 (0.7%) 1,743 (20.5%) 0.09 (0.34) 0.23 (0.59) 0.00 (0.03) 105.69 (77.60) 628.51 (384.70) | 682 (8.0%) 33 (0.4%) 411 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) 0.23 (0.58) 0.00 (0.06) 106.89 (77.05) 605.19 (348.57) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.06<br>-0.06<br>-0.00<br>-0.01<br>-0.00<br>- | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 617 (4.8%) 3056 (23.5%) 1676 (12.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) 0.08 (0.32) 0.24 (0.74) 0.00 (0.03) 92.83 (77.61) 1056.91 (847.86) | 903 (7.0%) #WALUEI #WALUEI 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 3147 (24.2%) #WALUEI 2709 (20.9%) 0.08 (0.32) 0.25 (0.77) 0.00 (0.05) 93.94 (77.37) 1058.00 (857.35) | 0.02 #VALUE! #VALUE! 0.00 0.00 -0.01 0.00 -0.02 -0.02 -0.02 -0.06 #VALUE! -0.03 0.00 0.00 0.00 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGIs (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of theat blockers; n (%) Use of theat blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications-insulin Copy; n (%) Use of High Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Cardiac biomarkers tests (tropnin, CK-MBs, Nmean (sd) Number of Ambulatory Blood pressure monitoring testsmean (sd) N of days on antihypertensive medications during baselimean (sd) N of days in database anytime priormean (sd) Mean Copay for per prescription cost (charges in U.S. S)mean (sd)Missing: n (%) | 107 (6.8%) **(0.1%) 0 (0.0%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) **(0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) 5: 0.00 (0.05) ine 80.03 (79.04) 1,668.43 (1,266.59) (180-1 day prior) 23.17 (31.74) 94 (6.0%) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.9%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) 0.37 (1.19) 0.00 (0.00) 83.44 (80.30) 1,713.11 (1,303.00) 23.95 (33.91) 90 (5.7%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.07<br>-0.05<br>-0.00<br>-0.05<br>-0.00<br>-0.05<br>-0.07 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 552 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) ** (0.2%) 544 (18.8%) 0.04 (0.21) 0.24 (0.91) 0.00 (0.02) 62.02 (76.84) 1,982.39 (1,383.61) 14.78 (20.67) 210 (7.2%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) 0.05 (0.25) 0.26 (0.93) 0.00 (0.03) 61.63 (76.67) 2,031.47 (1,419.09) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>-0.02<br>-0.02<br>-0.04<br>-0.03<br>-0.04<br>-0.03<br>-0.04 | 729 (8.6%) 22 (0.3%) 411 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 58 (0.7%) 1,743 (20.5%) 0.09 (0.34) 0.23 (0.59) 0.00 (0.03) 105.69 (77.60) 628.51 (384.70) 108.61 (103.27) 286 (3.4%) | 682 (8.0%) 33 (0.4%) 411 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) 0.23 (0.58) 0.00 (0.06) 106.89 (77.05) 605.19 (348.57) 109.54 (113.72) 297 (3.5%) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.02<br>-0.00<br>- | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 417 (4.8%) 3056 (23.5%) 1676 (12.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) 0.08 (0.32) 0.24 (0.74) 1056.91 (847.86) | 903 (7.0%) #VALUEI 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 2052 (15.8%) 4307 (33.2%) #VALUEI 2709 (20.9%) 0.08 (0.32) 0.25 (0.77) 0.00 (0.05) 93.94 (77.37) 1058.00 (857.35) 78.03 (98.05) 608 (4.7%) | 0.02 #VALUE! #VALUE! 0.00 0.00 -0.01 -0.02 -0.02 -0.02 -0.06 #VALUE! -0.03 0.00 0.00 0.00 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGIs (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of thiagh thiazide; n (%) DM Medications - Insulin Copy; n (%) Use of High Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Cardiac biomarkers tests (tropnin, CK-MBs, Nmean (sd) Number of Ambulatory Blood pressure monitoring testsmean (sd) N of days on antihypertensive medications during baselimean (sd) Mean Copay for per prescription cost (charges in U.S. S)mean (sd) Mean Copay for per prescription cost (charges in U.S. S)mean (sd)Missing: n (%) Colonoscopy; n (%) | 107 (6.8%) **(0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) **(0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) i 0.00 (0.05) ine 80.03 (79.04) 1,668.43 (1,266.59) (180-1 day prior) 23.17 (31.74) 94 (6.0%) 61 (3.9%) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) 0.37 (1.19) 0.00 (0.00) 83.44 (80.30) 1,713.11 (1,303.00) 23.95 (33.91) 90 (5.7%) 61 (3.9%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.05<br>-0.00<br>-0.05<br>-0.07<br>-0.00<br>-0.05<br>-0.00<br>-0.05<br>-0.00<br>-0.05<br>-0.00<br>-0.05<br>-0.00<br>-0.05<br>-0.00<br>- | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 552 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) 0.24 (0.91) 0.00 (0.02) 62.02 (76.84) 1,982.39 (1,383.61) 14.78 (20.67) 210 (7.2%) 127 (4.4%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 0.05 (0.25) 0.26 (0.93) 0.00 (0.03) 61.63 (76.67) 2,031.47 (1,419.09) 14.89 (66.84) 221 (7.6%) 121 (4.2%) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>0.02<br>-0.02<br>-0.04<br>-0.03<br>-0.04<br>-0.02<br>-0.04<br>-0.03 | 729 (8.6%) 22 (0.3%) 21 (0.1%) 730 (8.6%) 907 (10.7%) 907 (10.7%) 2.831 (33.3%) 2.270 (26.7%) 1.433 (16.8%) 380 (4.5%) 2.353 (27.6%) 1.202 (14.1%) 2.872 (33.7%) 58 (0.7%) 1.743 (20.5%) 0.09 (0.34) 0.23 (0.59) 0.00 (0.03) 105.69 (77.60) 628.51 (384.70) 108.61 (103.27) 286 (3.4%) 353 (4.1%) | 682 (8.0%) 33 (0.4%) 411 (0.1%) 721 (8.5%) 938 (11.0%) 938 (11.0%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) 0.23 (0.58) 0.00 (0.06) 106.89 (77.05) 605.19 (348.57) 109.54 (113.72) 297 (3.5%) 333 (3.9%) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.06<br>-0.04<br>-0.02<br>-0.00<br>- | 959 (7.4%) #WALUE! 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 617 (4.8%) 3056 (23.5%) 1767 (12.9%) 3945 (30.4%) #WALUE! 2565 (19.8%) 0.08 (0.32) 0.24 (0.74) 0.00 (0.03) 92.83 (77.61) 1056.91 (847.86) 77.30 (84.90) 590 (4.5%) 541 (4.2%) | 903 (7.0%) #VALUE! #VALUE! 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 3147 (24.2%) 4307 (33.2%) #VALUE! 2709 (20.9%) 0.08 (0.32) 0.25 (0.77) 0.00 (0.05) 93.94 (77.37) 1058.00 (857.35) 78.03 (98.05) 608 (4.7%) 515 (4.0%) | 0.02 #VALUE! #VAUE! 0.00 0.00 -0.01 0.00 -0.02 -0.02 -0.02 -0.00 -0.06 #VALUE! -0.03 0.00 0.00 0.00 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGIs (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of theat blockers; n (%) Use of theat blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except Insulin; n (%) DM Medications-insulin Copy; n (%) Use of High Intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Cardiac biomarkers tests (tropnin, CK-MBs, Nmean (sd) Number of Ambulatory Blood pressure monitoring testsmean (sd) N of days on antihypertensive medications during baselimean (sd) N of days in database anytime priormean (sd) Mean Copay for per prescription cost (charges in U.S. S)mean (sd)Missing: n (%) | 107 (6.8%) **(0.1%) 0 (0.0%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) **(0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) 5: 0.00 (0.05) ine 80.03 (79.04) 1,668.43 (1,266.59) (180-1 day prior) 23.17 (31.74) 94 (6.0%) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.9%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) 0.37 (1.19) 0.00 (0.00) 83.44 (80.30) 1,713.11 (1,303.00) 23.95 (33.91) 90 (5.7%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.07<br>-0.05<br>-0.00<br>-0.05<br>-0.07 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 552 (19.4%) 437 (15.1%) 337 (11.6%) 141 (4.9%) 391 (13.5%) 284 (9.8%) ** (0.2%) 544 (18.8%) 0.04 (0.21) 0.24 (0.91) 0.00 (0.02) 62.02 (76.84) 1,982.39 (1,383.61) 14.78 (20.67) 210 (7.2%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) 0.05 (0.25) 0.26 (0.93) 0.00 (0.03) 61.63 (76.67) 2,031.47 (1,419.09) | 0.00<br>0.00<br>0.04<br>-0.01<br>0.02<br>0.02<br>-0.02<br>-0.02<br>-0.04<br>-0.03<br>-0.04<br>-0.03<br>-0.04 | 729 (8.6%) 22 (0.3%) 411 (0.1%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 58 (0.7%) 1,743 (20.5%) 0.09 (0.34) 0.23 (0.59) 0.00 (0.03) 105.69 (77.60) 628.51 (384.70) 108.61 (103.27) 286 (3.4%) | 682 (8.0%) 33 (0.4%) 411 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) 0.23 (0.58) 0.00 (0.06) 106.89 (77.05) 605.19 (348.57) 109.54 (113.72) 297 (3.5%) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.02<br>-0.00<br>-0.02<br>-0.00<br>- | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 417 (4.8%) 3056 (23.5%) 1676 (12.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) 0.08 (0.32) 0.24 (0.74) 1056.91 (847.86) | 903 (7.0%) #VALUEI 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 2052 (15.8%) 4307 (33.2%) #VALUEI 2709 (20.9%) 0.08 (0.32) 0.25 (0.77) 0.00 (0.05) 93.94 (77.37) 1058.00 (857.35) 78.03 (98.05) 608 (4.7%) | 0.02 #VALUE! #VALUE! 0.00 0.00 -0.01 -0.02 -0.02 -0.02 -0.06 #VALUE! -0.03 0.00 0.00 0.00 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglithindes (for PS); n (%) Any use of AGis (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of thiazide; n (%) Use of theat blockers; n (%) Use of teat a blockers; n (%) Use of tableatic medications except insulin; n (%) DM Medications - Insulin Copy; n (%) Use of tow Intensity Statins; n (%) Use of High Intensity Statins; n (%) Use of High Intensity Statins; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Ambulatory Blood pressure monitoring testsmean (sd) N of days on antihypertensive medications during baselimean (sd) N of days in database anytime priormean (sd) Mean Copay for per prescription cost (charges in U.S. \$)mean (sd)Missing; n (%) Colonoscopy; n (%) Fecal occult blood (FOB) test; n (%) | 107 (6.8%) ** (0.1%) 0 (0.0%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 96 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) ** (0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) ** 0.00 (0.05) ine 80.03 (79.04) 1,668.43 (1,266.59) (180-1 day prior) 23.17 (31.74) 94 (6.0%) 61 (3.9%) 52 (3.3%) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 313 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 320 (20.3%) 0.08 (0.30) 0.37 (1.19) 0.00 (0.00) 83.44 (80.30) 1,713.11 (1,303.00) 23.95 (33.91) 90 (5.7%) 61 (3.9%) 54 (3.4%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>-0.05<br>-0.07<br>-0.05<br>-0.00<br>-0.05<br>-0.00<br>-0.05<br>-0.00<br>-0.05 | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 562 (19.4%) 437 (15.1%) 337 (11.6%) 331 (11.6%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) 0.24 (0.91) 0.00 (0.02) 62.02 (76.84) 1,982.39 (1,383.61) 14.78 (20.67) 210 (7.2%) 127 (4.4%) 76 (2.6%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) 0.05 (0.25) 0.26 (0.93) 0.00 (0.03) 61.63 (76.67) 2,031.47 (1,419.09) 14.89 (66.84) 221 (7.6%) 121 (4.2%) 76 (2.6%) | 0.00 0.00 0.00 0.00 0.04 0.01 0.02 0.00 0.02 0.02 0.02 0.04 0.02 0.05 -0.04 0.02 0.05 -0.04 -0.03 -0.04 -0.04 -0.02 0.00 0.00 0.01 -0.04 | 729 (8.6%) 22 (0.3%) 21 (0.13%) 21 (0.15%) 730 (8.6%) 907 (10.7%) 2,831 (33.3%) 2,270 (26.7%) 1,433 (16.8%) 380 (4.5%) 2,353 (27.6%) 1,202 (14.1%) 2,872 (33.7%) 58 (0.7%) 1,743 (20.5%) 0.09 (0.34) 0.23 (0.59) 0.00 (0.03) 105.69 (77.60) 628.51 (384.70) 108.61 (103.27) 286 (3.4%) 353 (4.1%) 244 (2.9%) | 682 (8.0%) 33 (0.4%) <11 (0.1%) 721 (8.5%) 938 (11.0%) 2,870 (33.7%) 2,240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) 0.23 (0.58) 0.00 (0.06) 106.89 (77.05) 605.19 (348.57) 109.54 (113.72) 297 (3.5%) 333 (3.9%) 224 (2.6%) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.01<br>-0.02<br>-0.00<br>- | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3759 (28.9%) 3004 (23.1%) 2011 (15.5%) 617 (4.8%) 3056 (23.5%) 476 (12.9%) 3945 (30.4%) #WALUEI 2565 (19.8%) 0.08 (0.32) 0.24 (0.74) 0.00 (0.03) 92.83 (77.61) 1056.91 (847.86) 77.30 (84.90) 590 (4.5%) 541 (4.2%) 372 (2.9%) | 903 (7.0%) #WALUEI #WALUEI 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 2052 (15.8%) 670 (5.2%) 3147 (24.2%) 4307 (33.2%) #WALUEI 2709 (20.9%) 0.08 (0.32) 0.25 (0.77) 0.00 (0.05) 93.94 (77.37) 1058.00 (857.35) 78.03 (98.05) 608 (4.7%) 515 (4.0%) 354 (2.7%) | 0.02 #VALUE! #VALUE! 0.00 0.00 -0.01 -0.02 -0.02 -0.02 -0.06 #VALUE! -0.03 0.00 0.00 0.00 0.00 |
| Delirium + Psychosis (for PS); n (%) Any use of Meglitinides (for PS); n (%) Any use of AGIs (for PS); n (%) CKD stage 3-6 + dialysis (for PS); n (%) Use of beta blockers; n (%) Use of beta blockers; n (%) Use of calcium channel blockers; n (%) All antidiabetic medications except insulin; n (%) DM Medications - Insulin Copy; n (%) Use of Low intensity Statins; n (%) Use of High Intensity Statins; n (%) Malignant hypertension; n (%) Cardiovascular stress test; n (%) Echocardiogram; n (%) Number of BNP testsmean (sd) Number of Cardiac biomarkers tests (tropnin, CK-MBs, Nmean (sd) Number of Ambulatory Blood pressure monitoring testsmean (sd) N of days on antihypertensive medications during baselimean (sd) Mean Copay for per prescription cost (charges in U.S. \$)mean (sd) Mean Copay for per prescription cost (charges in U.S. \$)mean (sd) Mean Copay for per prescription cost (charges in U.S. \$)mean (sd) | 107 (6.8%) **(0.1%) 0 (0.0%) 120 (7.6%) 149 (9.5%) 366 (23.2%) 297 (18.9%) 241 (15.3%) 95 (6.1%) 312 (19.8%) 190 (12.1%) 107 (6.8%) **(0.4%) 278 (17.7%) 0.08 (0.35) Ayoglobin, CPK) 0.31 (1.04) 6 80.03 (79.04) 1,668.43 (1,266.59) (180-1 day prior) 23.17 (31.74) 94 (6.0%) 61 (3.9%) 52 (3.3%) 253 (16.1%) | 100 (6.3%) ** (0.3%) ** (0.3%) ** (0.2%) 133 (8.4%) 147 (9.3%) 379 (24.1%) 331 (19.9%) 239 (15.2%) 96 (6.1%) 344 (21.8%) 190 (12.1%) 152 (9.7%) ** (0.1%) 320 (20.3%) 0.08 (0.30) 0.37 (1.19) 0.00 (0.00) 83.44 (80.30) 1,713.11 (1,303.00) 23.95 (33.91) 90 (5.7%) 61 (3.9%) 54 (3.4%) 238 (15.1%) | 0.02<br>-0.04<br>-0.06<br>-0.03<br>-0.01<br>-0.02<br>-0.03<br>-0.00<br>-0.05<br>-0.00<br>- | 123 (4.2%) ** (0.1%) 0 (0.0%) 78 (2.7%) 211 (7.3%) 211 (7.3%) 437 (15.1%) 337 (11.6%) 347 (15.1%) 349 (14.6%) 391 (13.5%) 284 (9.8%) 966 (33.3%) ** (0.2%) 544 (18.8%) 0.04 (0.21) 0.24 (0.91) 0.00 (0.02) 62.02 (76.84) 1,982.39 (1,383.61) 14.78 (20.67) 210 (7.2%) 127 (4.4%) 76 (2.6%) 270 (9.3%) | 121 (4.2%) ** (0.1%) ** (0.1%) ** (0.1%) ** (0.1%) 85 (2.9%) 195 (6.7%) 546 (18.8%) 441 (15.2%) 359 (12.4%) 153 (5.3%) 430 (14.8%) 271 (9.3%) 1,037 (35.8%) 12 (0.4%) 574 (19.8%) 0.05 (0.25) 0.26 (0.93) 0.00 (0.03) 61.63 (76.67) 2,031.47 (1,419.09) 14.89 (66.84) 221 (7.6%) 121 (4.2%) 76 (2.6%) 279 (9.6%) | 0.00 0.00 0.00 0.04 -0.01 0.02 0.02 0.02 -0.02 -0.02 -0.04 -0.03 -0.04 -0.03 -0.04 -0.03 -0.04 -0.03 -0.04 -0.00 0.01 | 729 (8.6%) 22 (0.3%) 21 (0.1%) 730 (8.6%) 907 (10.7%) 907 (10.7%) 2.831 (33.3%) 2.270 (26.7%) 1.433 (16.8%) 380 (4.5%) 2.353 (27.6%) 1,202 (14.1%) 2.872 (33.7%) 58 (0.7%) 1,743 (20.5%) 0.09 (0.34) 0.23 (0.59) 0.00 (0.03) 105.69 (77.60) 628.51 (384.70) 108.61 (103.27) 286 (3.4%) 353 (4.1%) 244 (2.9%) 2,434 (28.6%) | 682 (8.0%) 33 (0.4%) 411 (0.1%) 721 (8.5%) 938 (11.0%) 9.240 (26.3%) 1,454 (17.1%) 421 (4.9%) 2,373 (27.9%) 1,200 (14.1%) 3,118 (36.6%) 37 (0.4%) 1,815 (21.3%) 0.09 (0.34) 0.23 (0.58) 0.00 (0.06) 106.89 (77.05) 605.19 (348.57) 109.54 (113.72) 297 (3.5%) 333 (3.9%) 224 (2.6%) 2,417 (28.4%) | 0.02<br>-0.02<br>-0.02<br>-0.00<br>-0.01<br>-0.01<br>-0.01<br>-0.02<br>-0.06<br>-0.04<br>-0.02<br>-0.00<br>- | 959 (7.4%) #WALUEI 928 (7.1%) 1267 (9.8%) 3004 (23.1%) 3004 (23.1%) 3014 (23.1%) 617 (4.8%) 3056 (23.5%) 1676 (12.9%) 3945 (30.4%) 47VALUEI 2565 (19.8%) 0.08 (0.32) 0.24 (0.74) 0.00 (0.03) 92.83 (77.61) 1056.91 (847.86) 77.30 (84.90) 590 (4.5%) 541 (4.2%) 372 (2.9%) 3257 (22.8%) | 903 (7.0%) #VALUEI #VALUEI 939 (7.2%) 1280 (9.9%) 3795 (29.2%) 2994 (23.1%) 670 (5.2%) 3147 (24.2%) 3160 (12.8%) 4307 (33.2%) 0.08 (0.32) 0.25 (0.77) 0.00 (0.05) 93.94 (77.37) 1058.00 (857.35) 78.03 (98.05) 608 (4.7%) 515 (4.0%) 354 (2.7%) 2934 (22.5%) | 0.02 #VALUE! #VOLUE! #VOLUE! #VOLUE! 0.00 0.00 -0.01 -0.02 -0.02 -0.06 #VALUE! -0.03 0.00 0.00 0.00 0.00 |

| PSA test or Prostate exam for DRE; n (%) | 157 (10.0%) | 154 (9.8%) | 0.01 | 234 (8.1%) | 237 (8.2%) | 0.00 | 886 (10.4%) | 872 (10.2%) | 0.01 | 1277 (9.8%) | 1263 (9.7%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Bone mineral density; n (%) | 67 (4.3%) | 60 (3.8%) | 0.03 | 51 (1.8%) | 49 (1.7%) | 0.01 | 382 (4.5%) | 381 (4.5%) | 0.00 | 500 (3.9%) | 490 (3.8%) | 0.01 |
| Use of CNS stimulants; n (%) | 15 (1.0%) | ** (0.6%) | 0.04 | 47 (1.6%) | 59 (2.0%) | -0.03 | 35 (0.4%) | 34 (0.4%) | 0.00 | 97 (0.7%) | #VALUE! | #VALUE! |
| Use of estrogens, progestins, androgens; n (%) | 86 (5.5%) | 78 (5.0%) | 0.02 | 355 (12.2%) | 323 (11.1%) | 0.03 | 311 (3.7%) | 299 (3.5%) | 0.01 | 752 (5.8%) | 700 (5.4%) | 0.02 |
| Use of Angiogenesis inhibitors; n (%) | 0 (0.0%) | ** (0.1%) | -0.04 | ** (0.1%) | ** (0.2%) | -0.03 | 10 (0.1%) | 8 (0.1%) | 0.00 | #VALUE! | #VALUE! | #VALUE! |
| | | | | | | | | - 1 | | | | |
| Use of Oral Immunosuppressants; n (%) | ** (0.6%) | ** (0.3%) | 0.04 | 27 (0.9%) | 13 (0.4%) | 0.06 | 6 (0.1%) | 12 (0.1%) | 0.00 | #VALUE! | #VALUE! | #VALUE! |
| Use of fondaparinux or Bivalirudin; n (%) | ** (0.5%) | ** (0.4%) | 0.01 | 20 (0.7%) | 16 (0.6%) | 0.01 | 19 (0.2%) | 24 (0.3%) | -0.02 | #VALUE! | #VALUE! | #VALUE! |
| Use of other direct thrombin inhibitors (lepirudin, des | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Use of Ticagrelor ON CED; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | ** (0.1%) | ** (0.1%) | 0.00 | 1 (0.0%) | 1 (0.0%) | #DIV/0! | #VALUE! | #VALUE! | #VALUE! |
| Use of Ticagrelor; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | ** (0.1%) | ** (0.1%) | 0.00 | 14 (0.2%) | 12 (0.1%) | 0.03 | #VALUE! | #VALUE! | #VALUE! |
| Number of D-dimer tests | | | | | | | | | | | | |
| mean (sd) | 0.08 (0.29) | 0.07 (0.31) | 0.03 | 0.07 (0.29) | 0.06 (0.29) | 0.03 | 0.08 (0.30) | 0.09 (0.30) | -0.03 | 0.08 (0.30) | 0.08 (0.30) | 0.00 |
| Numbe of CRP, high-sensitivity CRP tests | | | | | | | | | | | | |
| mean (sd) | 0.17 (0.67) | 0.16 (0.70) | 0.01 | 0.14 (0.61) | 0.14 (0.58) | 0.00 | 0.16 (0.86) | 0.16 (0.69) | 0.00 | 0.16 (0.79) | 0.16 (0.67) | 0.00 |
| Number of PT or aPTTt tests | | | | | | | | | | | | |
| mean (sd) | 1.03 (2.00) | 1.02 (1.76) | 0.01 | 0.71 (1.58) | 0.72 (1.57) | -0.01 | 0.56 (0.92) | 0.55 (1.01) | 0.01 | 0.65 (1.26) | 0.64 (1.26) | 0.00 |
| Number of Bleeding time tests | | , , | | , , | , , | | | | | | , , | |
| mean (sd) | 0.00 (0.00) | 0.00 (0.00) | #DIV/0! | 0.00 (0.03) | 0.00 (0.03) | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 |
| HAS-BLED Score (ICD-9 and ICD-10), 180 days | 0.00 (0.00) | 0.00 (0.00) | #514/0: | 0.00 (0.03) | 0.00 (0.03) | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 | 0.00 (0.02) | 0.00 (0.02) | 0.00 |
| mean (sd) | 2.89 (1.02) | 2.93 (1.07) | -0.04 | 2.37 (1.00) | 2.37 (0.99) | 0.00 | 3.49 (0.82) | 3.48 (0.81) | 0.01 | 3.17 (0.89) | 3.17 (0.89) | 0.00 |
| N of Generic name drugs | 2.89 (1.02) | 2.93 (1.07) | -0.04 | 2.37 (1.00) | 2.37 (0.99) | 0.00 | 3.49 (0.82) | 3.46 (0.81) | 0.01 | 3.17 (0.89) | 3.17 (0.89) | 0.00 |
| mean (sd) | 18.54 (17.31) | 18.70 (19.99) | -0.01 | 13.69 (11.34) | 13.71 (12.94) | 0.00 | 18.66 (14.45) | 18.74 (16.05) | -0.01 | 17.54 (14.21) | 17.61 (15.96) | 0.00 |
| N of Brand name drugs | | | | | | | | | | | | |
| mean (sd) | 3.61 (6.03) | 3.61 (4.03) | 0.00 | 3.54 (5.26) | 3.63 (3.55) | -0.02 | 3.99 (6.55) | 3.97 (4.25) | 0.00 | 3.84 (6.22) | 3.85 (4.08) | 0.00 |
| Use of clopidogrel ; n (%) | 60 (3.8%) | 63 (4.0%) | -0.01 | 91 (3.1%) | 100 (3.4%) | -0.02 | 539 (6.3%) | 543 (6.4%) | 0.00 | 690 (5.3%) | 706 (5.4%) | 0.00 |
| Systemic embolism; n (%) | 62 (3.9%) | 53 (3.4%) | 0.03 | 145 (5.0%) | 156 (5.4%) | -0.02 | 216 (2.5%) | 210 (2.5%) | 0.00 | 423 (3.3%) | 419 (3.2%) | 0.01 |
| DVT; n (%) | 1,575 (100.0%) | 1,575 (100.0%) | #DIV/0! | 2,897 (99.9%) | 2,898 (100.0%) | -0.04 | 8,504 (99.9%) | 8,503 (99.9%) | 0.00 | 12976 (99.9%) | 12976 (99.9%) | 0.00 |
| Post-thrombotic syndrome; n (%) | ** (0.3%) | ** (0.3%) | #DIV/0! | ** (0.2%) | ** (0.2%) | #DIV/0! | 23 (0.3%) | 20 (0.2%) | #DIV/0! | ** (0.2%) | ** (0.2%) | 0.00 |
| PE: n (%) | 163 (10.3%) | 158 (10.0%) | 0.01 | 141 (4.9%) | 132 (4.6%) | 0.01 | 599 (7.0%) | 612 (7.2%) | -0.01 | 903 (7.0%) | 902 (6.9%) | 0.00 |
| Coagulation defects: n (%) | 43 (2.7%) | 46 (2.9%) | #DIV/0! | 110 (3.8%) | 110 (3.8%) | #DIV/0! | 159 (1.9%) | 141 (1.7%) | #DIV/0! | 110 (3.8%) | 110 (3.8%) | 0.00 |
| Coagulation delects, it (70) | 45 (2.770) | 40 (2.570) | #514/0: | 110 (5.670) | 110 (5.670) | #514/0: | 155 (1.570) | 141 (1.770) | #DIV/0: | 110 (3.0%) | 110 (3.670) | 0.00 |
| Diabetes: 1 inpatient or 2 outpatient claims within 18 | 391 (24.8%) | 393 (25.0%) | 0.00 | 516 (17.8%) | 543 (18.7%) | -0.02 | 2,342 (27.5%) | 2,351 (27.6%) | 0.00 | 3249 (25.0%) | 3287 (25.3%) | -0.01 |
| Diabetes: 1 inpution of 2 output on counts within 20 | 331 (24.070) | 333 (23.0%) | 0.00 | 310 (17.070) | 343 (20.770) | 0.02 | 2,542 (27.570) | 2,551 (27.676) | 0.00 | 3243 (23.0%) | 5257 (25.570) | 0.01 |
| | ** (0.1%) | ** (0.1%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 12 (0.1%) | 10 (0.1%) | 0.00 | #VALUE! | #VALUE! | #VALUE! |
| Intracranial or retroperitoneal hemorrhage: 1 inpatier | | | | | , | | , | | | | | |
| Peptic Ulcer Disease; n (%) | 399 (25.3%) | 407 (25.8%) | -0.01 | 574 (19.8%) | 571 (19.7%) | 0.00 | 2,559 (30.1%) | 2,560 (30.1%) | 0.00 | 3532 (27.2%) | 3538 (27.2%) | 0.00 |
| Major Surgery ; n (%) | 154 (9.8%) | 147 (9.3%) | #DIV/0! | 262 (9.0%) | 261 (9.0%) | #DIV/0! | 854 (10.0%) | 835 (9.8%) | #DIV/0! | 262 (9.0%) | 261 (9.0%) | 0.00 |
| Upper GI bleed; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Lower/ unspecified GI bleed; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Urogenital bleed; n (%) | ** (0.3%) | ** (0.3%) | 0.00 | 27 (0.9%) | 30 (1.0%) | -0.01 | 1 (0.0%) | 0 (0.0%) | #DIV/0! | #VALUE! | #VALUE! | #VALUE! |
| Other bleeds; n (%) | 106 (6.7%) | 110 (7.0%) | -0.01 | 170 (5.9%) | 170 (5.9%) | 0.00 | 512 (6.0%) | 490 (5.8%) | 0.01 | 788 (6.1%) | 770 (5.9%) | 0.01 |
| Prior cancer: n (%) | 237 (15.0%) | 228 (14.5%) | 0.01 | 351 (12.1%) | 331 (11.4%) | 0.02 | 1.577 (18.5%) | 1.523 (17.9%) | 0.02 | 2165 (16.7%) | 2082 (16.0%) | 0.02 |
| Antibiotics: n (%) | 751 (47.7%) | 774 (49.1%) | #DIV/0! | 1,526 (52.6%) | 1,514 (52.2%) | #DIV/0! | 4.722 (55.5%) | 4,673 (54.9%) | #DIV/0! | 1,526 (52.6%) | 1,514 (52.2%) | 0.01 |
| Aspirin: n (%) | ** (0.6%) | ** (0.6%) | 0.00 | 51 (1.8%) | 48 (1.7%) | 0.01 | 37 (0.4%) | 42 (0.5%) | -0.01 | #VALUE! | #VALUE! | #VALUE! |
| Aspirin/dipyridamole; n (%) | ** (0.2%) | ** (0.2%) | 0.00 | ** (0.1%) | ** (0.1%) | 0.00 | 26 (0.3%) | 30 (0.4%) | -0.02 | #VALUE! | #VALUE! | #VALUE! |
| | ** (0.3%) | ** (0.3%) | 0.00 | ** (0.1%) | ** (0.3%) | -0.04 | | | 0.00 | #VALUE! | #VALUE! | #VALUE! |
| Other antiplatelet agents; n (%) | | | 0.00 | | | 0.04 | 53 (0.6%) | 50 (0.6%) | 0.00 | | | |
| PGP inhibitors; n (%) | 280 (17.8%) | 281 (17.8%) | | 546 (18.8%) | 548 (18.9%) | | 1,954 (23.0%) | 1,957 (23.0%) | | 2780 (21.4%) | 2786 (21.5%) | 0.00 |
| Other gastroprotective agents; n (%) | 24 (1.5%) | 26 (1.7%) | -0.02 | 56 (1.9%) | 49 (1.7%) | 0.02 | 141 (1.7%) | 143 (1.7%) | 0.00 | 221 (1.7%) | 218 (1.7%) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.49 (0.78) | 0.47 (0.74) | 0.03 | 0.35 (0.80) | 0.34 (0.78) | 0.01 | 0.55 (0.84) | 0.56 (0.83) | -0.01 | 0.50 (0.82) | 0.50 (0.81) | 0.00 |
| Proton pump inhibitor; n (%) | 380 (24.1%) | 379 (24.1%) | 0.00 | 618 (21.3%) | 633 (21.8%) | -0.01 | 2,625 (30.8%) | 2,667 (31.3%) | -0.01 | 3623 (27.9%) | 3679 (28.3%) | -0.01 |
| H2 receptor antagonist; n (%) | 73 (4.6%) | 66 (4.2%) | 0.02 | 117 (4.0%) | 119 (4.1%) | -0.01 | 578 (6.8%) | 546 (6.4%) | 0.02 | 768 (5.9%) | 731 (5.6%) | 0.01 |
| Vitamin K therapy; n (%) | ** (0.1%) | ** (0.1%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 2 (0.0%) | 1 (0.0%) | #DIV/0! | #VALUE! | #VALUE! | #VALUE! |
| Number of INR (prothrombin) tests ordered | | | | | | | | | | | | |
| mean (sd) | 0.73 (1.55) | 0.58 (1.00) | 0.12 | 0.52 (1.11) | 0.47 (1.03) | 0.05 | 0.53 (0.86) | 0.50 (0.85) | 0.04 | 0.55 (1.03) | 0.50 (0.91) | 0.00 |
| Treating prescriber - Cardiologist; n (%) | 508 (32.3%) | 509 (32.3%) | 0.00 | 1,002 (34.6%) | 994 (34.3%) | 0.01 | 3,097 (36.4%) | 3,041 (35.7%) | 0.01 | 4607 (35.5%) | 4544 (35.0%) | 0.01 |
| Treating prescriber - Primary Care Physician; n (%) | 1.368 (86.9%) | 1.399 (88.8%) | -0.06 | 1.243 (42.9%) | 1.247 (43.0%) | 0.00 | 3,431 (40.3%) | 3,422 (40.2%) | 0.00 | 6042 (46.5%) | 6068 (46.7%) | 0.00 |
| Treating prescriber - Other; n (%) | 1,574 (99.9%) | 1,574 (99.9%) | 0.00 | 2,754 (95.0%) | 2,761 (95.2%) | -0.01 | 8,475 (99.6%) | 8,483 (99.7%) | -0.02 | 12803 (98.6%) | 12818 (98.7%) | -0.01 |
| Alpha blockers: n (%) | 121 (7.7%) | 124 (7.9%) | -0.01 | 162 (5.6%) | 159 (5.5%) | 0.00 | 868 (10.2%) | 862 (10.1%) | 0.00 | 1151 (8.9%) | 1145 (8.8%) | 0.00 |
| CHA2DS2 VASc score, 180 days, V | 121 (7.770) | 127 (1.370) | -0.01 | 102 (3.070) | 133 (3.3/0) | 0.00 | 000 (10.270) | 002 (10.1/0) | 0.00 | 1131 (0.570) | 1145 (0.070) | 0.00 |
| | 2.42 (4.04) | 2 22 (4 70) | 0.05 | 2.00 (4.70) | 2.00 (4.50) | 0.05 | 4.00 (4.03) | 4.7 (4.02) | -0.05 | 2.70 (4.00) | 2 70 (4 70) | 0.00 |
| mean (sd) | 3.13 (1.81) | 3.22 (1.79) | -0.05<br>0.04 | 2.90 (1.70) | 2.98 (1.68) | -0.05<br>0.00 | 4.08 (1.83) | 4.17 (1.82) | | 3.70 (1.80)<br>#VALUE! | 3.79 (1.79)<br>#VALUE! | #VALUFI |
| Use of Prasugrel; n (%) | ** (0.1%) | 0 (0.0%) | 0.04 | ** (0.1%) | ** (0.1%) | 0.00 | 1 (0.0%) | 1 (0.0%) | #DIV/0! | #VALUE! | #VALUE! | #VALUE! |
| 11 - 12 - 15 - 15 - 15 - 15 - 15 - 15 - | 227 (45 00/) | 247 (45 70/) | 0.00 | 254 (42 40() | 240 (42 00() | 0.00 | 4.054(24.00() | 4 004 (22 20) | 0.04 | 2452 (40.00() | 2407 (40 20() | 0.04 |
| Use of Loop Diuretics+other diuretics+other hyperten: | 237 (15.0%) | 247 (15.7%) | -0.02 | 351 (12.1%) | 349 (12.0%) | 0.00 | 1,864 (21.9%) | 1,901 (22.3%) | -0.01 | 2452 (18.9%) | 2497 (19.2%) | -0.01 |
| and the second s | NADECT ONE | | | | | | _ | _ | | | | |
| Commercial vs Medicare Advantage- Business Type Code - CC | | | | | | | 0 | 0 | | | | |
| Commercial; n (%) | 495 (31.4%) | 471 (29.9%) | 0.03 | 688 (23.7%) | 708 (24.4%) | -0.02 | - | - | #VALUE! | 1,183 (26.4%) | 1,179 (26.4%) | 0.00 |
| Medicare Advantage; n (%) | 1,080 (68.6%) | 1104 (70.1%) | -0.03 | 2211 (76.3%) | 2191 (75.6%) | 0.02 | - | - | #VALUE! | 3,291 (73.6%) | 3,295 (73.6%) | 0.00 |
| Commercial vs Medicare Advantage- Business Type Code | | | | | | | | | | | | |
| COM = COMMERCIAL; n (%) | 495 (31.4%) | 471 (29.9%) | 0.03 | - | - | #VALUE! | - | - | #VALUE! | 495 (31.4%) | 471 (29.9%) | 0.03 |
| MCR = MEDICARE; n (%) | 1,080 (68.6%) | 1,104 (70.1%) | -0.03 | | - | #VALUE! | - | | #VALUE! | 1,080 (68.6%) | 1,104 (70.1%) | -0.03 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| | | | | | | | | | | | . , | |
| NONE = NO BUSINESS LINE CODE (added in 2015); n ( | | - / | #DIV/0! | | | #VALUE! | _ | _ | #VALUE! | 0 (0.0%) | 0 (0 00/) | #DIV/0! |
| | 0 (0.0%) | 0 (0.0%) | #DIV/U: | | - | | | | | 0 (0.070) | 0 (0.0%) | |
| UNK = UNKNOWN (added in 2015); n (%) | | | #DIV/0! | | | #VALUE! | _ | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| UNK = UNKNOWN (added in 2015); n (%) Commercial vs Medicare Advantage- Data Type | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | , | -<br>-<br>0 | - 0 | | | - | | | | , |

| 1 - Fee For Service; n (%)2 - Encounter; n (%)3 - Medicare; n (%)4 - Medicare Encounter; n (%) | -<br>-<br>- | -<br>-<br>- | 1,985 (68.5%)<br>226 (7.8%)<br>625 (21.6%)<br>63 (2.2%) | 1,967 (67.9%)<br>224 (7.7%)<br>643 (22.2%)<br>65 (2.2%) | -<br>-<br>- | -<br>-<br>- | 1,985 (68.5%)<br>226 (7.8%)<br>625 (21.6%)<br>63 (2.2%) | 1,967 (67.9%)<br>224 (7.7%)<br>643 (22.2%)<br>65 (2.2%) | 0.00<br>0.00<br>0.00<br>0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Metropolitan Statistical Area - Urban (any MSA) vs Rural (non-MSA) | | | | | | | 0 | 0 | 0.00 |
| Urban; n (%) | - | - | 2,156 (74.4%) | 2,161 (74.5%) | - | | 2,156 (74.4%) | 2,161 (74.5%) | |
| Rural; n (%) | - | - | 100 (3.4%) | 95 (3.3%) | - | | 100 (3.4%) | 95 (3.3%) | |
| Unknown/Missing; n (%) | - | | 643 (22.2%) | 643 (22.2%) | - | - | 643 (22.2%) | 643 (22.2%) | |